

## **PROTOCOL**

# **HVTN 703/HPTN 081**

A phase 2b study to evaluate the safety and efficacy of VRC01 broadly neutralizing monoclonal antibody in reducing acquisition of HIV-1 infection in women in sub-Saharan Africa

**DAIDS DOCUMENT ID 12045** 

#### **CLINICAL TRIAL SPONSORED BY**

Division of AIDS (DAIDS)

National Institute of Allergy and Infectious Diseases (NIAID)

National Institutes of Health (NIH)

Department of Health and Human Services (DHHS)

Bethesda, Maryland, USA

## STUDY PRODUCT(S) PROVIDED BY

Dale and Betty Bumpers Vaccine Research Center (VRC), NIAID, NIH, DHHS Bethesda, Maryland, USA

**December 14, 2017** HVTN 703/HPTN 081 Version 4.0

## **Contents**

| 1 | Overviev | N | 5 |
|---|---|---|---|
| | 1.1 | Protocol Team | 8 |
| 2 | Backgro | und | 11 |
| | 2.1 | Rationale for trial concept | |
| | 2.2 | bnAbs to HIV-1 | |
| | 2.3 | VRC01: VRC-HIVMAB060-00-AB | 15 |
| | 2.4 | Trial design rationale | 16 |
| | 2.5 | Combination prevention for HIV acquisition | 22 |
| | 2.6 | Plans for future product development and testing | 25 |
| | 2.7 | Preclinical safety studies | |
| | 2.8 | Nonhuman primate (NHP) studies of VRC01 | 29 |
| | 2.9 | Clinical trial experience | 32 |
| | 2.10 | Potential risks of study products and administration | 40 |
| 3 | Objectiv | es and endpoints | 42 |
| | 3.1 | Primary objectives and endpoints | |
| | 3.2 | Secondary objectives and endpoints | |
| | 3.3 | Exploratory objectives | |
| 4 | Statistica | al considerations | 44 |
| | 4.1 | Outline of the statistical considerations section | |
| | 4.2 | PE parameters for measuring mAb efficacy and associated primary and | |
| | | secondary hypothesis tests | |
| | 4.3 | Statistical rationale for the 3-arm design compared to a 2-arm design | 45 |
| | 4.4 | Sample size calculations for testing for overall PE (Primary objective 2). | 46 |
| | 4.5 | Power for the secondary analysis comparing HIV-1 incidence between the | he |
| | | 10 mg/kg mAb group versus the 30 mg/kg mAb group | 54 |
| | 4.6 | Sample size calculations for safety | 55 |
| | 4.7 | Monitoring of the trial | 56 |
| | 4.8 | Assessment of PrEP use | 61 |
| | 4.9 | Randomization | 61 |
| | 4.10 | Blinding | 62 |
| | 4.11 | Statistical analyses. | 62 |
| 5 | Selection | n and withdrawal of participants | 77 |
| | 5.1 | Inclusion criteria | 77 |
| | 5.2 | Exclusion criteria | 79 |
| | 5.3 | Participant departure from infusion schedule or withdrawal | 80 |
| 6 | Study pr | oduct preparation and administration | 83 |
| | 6.1 | Study product regimen | |
| | 6.2 | Study product formulation | |
| | 6.3 | Preparation of study products | |
| | 6.4 | Administration | |
| | 6.5 | Acquisition of study products | |
| | 6.6 | Pharmacy records | |
| | 6.7 | Final disposition of study products | 88 |

## HVTN 703/HPTN 081 Version 4.0 / December 14, 2017

| 7 | Clinical 1 | procedures | 89 |
|---|---|---|---|
| | 7.1 | Informed consent | 89 |
| | 7.2 | Pre-enrollment procedures | 91 |
| | 7.3 | Enrollment and infusion visits | 92 |
| | 7.4 | Post-infusion visits for HIV-uninfected study participants | 94 |
| | 7.5 | HIV counseling and testing | 95 |
| | 7.6 | Follow-up visits for HIV-infected participants | 96 |
| | 7.7 | Follow-up visits for participants who discontinue infusions for reason | |
| | | than HIV infection. | |
| | 7.8 | Contraception status | |
| | 7.9 | Urine testing | 98 |
| | 7.10 | Assessments of reactogenicity | |
| | | Visit windows and missed visits | |
| | 7.12 | Early termination visit | 100 |
| | | Pregnancy | |
| 0 | | | |
| 8 | | ction assessment and clinical response | |
| | 8.1<br>8.2 | HIV symptom assessment | |
| | | HIV screening test (prior to randomization) | |
| | 8.3 | HIV testing postinfusion | |
| | 8.4 | Endpoint adjudication | |
| | 8.5 | HIV infection during the study | |
| | 8.6 | Medical care for participants who become HIV infected | 103 |
| 9 | Laborato | ry | |
| | 9.1 | CRS laboratory procedures | |
| | 9.2 | Total blood volume | 104 |
| | 9.3 | Assay timepoints | 104 |
| | 9.4 | VRC01 mAb levels | 104 |
| | 9.5 | Endpoint assays: humoral | 105 |
| | 9.6 | ARV detection | 105 |
| | 9.7 | Host (human) genotyping | 106 |
| | 9.8 | Lab assay algorithm | 106 |
| | 9.9 | Possible additional studies | 106 |
| | | Other use of stored specimens | |
| | 9.11 | Biohazard containment | 107 |
| 10 | Safety m | onitoring and safety review | 108 |
| 10 | 10.1 | | |
| | | Safety reporting | |
| | | Safety pause and prompt PSRT AE review | |
| | | Review of cumulative safety data | |
| | | Study termination | |
| | | Social impact reporting | |
| 1.1 | | | |
| 11 | | conduct | |
| | | Emergency communication with study participants | |
| 12 | Ethical c | onsiderations | 118 |
| 12 | ID D/EC/ | RE review considerations | 120 |

## HVTN 703/HPTN 081 Version 4.0 / December 14, 2017

| 13.1 | Minimized risks to participants | 120 |
|---|---|---|
| 13.2 | Reasonable risk/benefit balance | 121 |
| 13.3 | Equitable subject selection | 121 |
| | Appropriate informed consent. | |
| | Adequate safety monitoring | |
| 13.6 | Protect privacy/confidentiality | 122 |
| 14 Version l | nistory | 123 |
| 15 Documen | nt references (other than literature citations) | 129 |
| 16 Acronym | ns and abbreviations | 131 |
| 17 Literature | e cited | 134 |
| Appendix A | Sample informed consent form | 148 |
| Appendix B | Approved birth control methods (for sample informed consent form) | 168 |
| Appendix C | Sample consent form for use of samples and information in other studies | 169 |
| Appendix D | Tables of procedures (for sample informed consent form) | 174 |
| Appendix E | Sample consent form for participants with HIV infection at enrollment or during the study | |
| Appendix F | Schedule 1—Laboratory procedures for HIV-uninfected participants | 181 |
| Appendix G | Schedule 2—Laboratory procedures for HIV-1-infected participants | 183 |
| Appendix H | Schedule 3—Laboratory procedures for participants discovered to have been HIV-1–infected at enrollment or who become HIV-2–infected | 185 |
| Appendix I | Schedule 4—Laboratory procedures for participants who discontinue infusions for reasons other than HIV infection | 187 |
| Appendix J | Schedule 1—Procedures at CRS for HIV-uninfected participants | 188 |
| Appendix K | Schedule 2—Procedures at CRS for HIV-1-infected participants | 190 |
| Appendix L | Schedule 3—Procedures at CRS for participants discovered to have been HIV-1–infected at enrollment or who become HIV-2–infected | |
| Appendix M | Schedule 4—Procedures at CRS for participants who discontinue infusion for reasons other than HIV infection | |
| Appendix N | Protocol Signature Page | 193 |

## 1 Overview

#### **Title**

A phase 2b study to evaluate the safety and efficacy of VRC01 broadly neutralizing monoclonal antibody in reducing acquisition of HIV-1 infection in women in sub-Saharan Africa

#### **Primary objectives**

- To evaluate the safety and tolerability of VRC01 mAb administered through IV infusion in sub-Saharan African women
- To determine if the VRC01 mAb prevents HIV-1 infection and to estimate the level of efficacy in sub-Saharan African women

#### Study products and routes of administration

- VRC01: human monoclonal antibody (mAb) VRC-HIVMAB060-00-AB in formulation buffer at pH 5.8 in sufficient normal saline (Sodium Chloride for Injection 0.9%, USP) to be administered at a final volume of 150 mL intravenously (IV)
- Control for VRC01: Sodium Chloride for Injection 0.9%, USP administered at a volume of 150 mL IV

Table 1-1 Schema

| | | | | Infusion schedule (Weeks) [A = VRC01 infusion; C = Control infusion] | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Treatment | N* | W0 | W8 | W16 | W24 | W32 | W40 | W48 | W56 | W64 | W72 | W80* | W104† |
| Group | VRC01 | 634* | | ۸ | _ | | Α | Α | ^ | ^ | ^ | ^ | | |
| 1 | 10 mg/kg | 634 | Α | Α | Α | Α | А | А | Α | Α | Α | Α | | |
| Group | VRC01 | 634* | Α | Α | Α | Α | Α | Α | Α | Α | Α | Α | | |
| 2 | 30 mg/kg | 034 | А | 4 | А | А | А | A | A | A | 4 | 4 | | |
| Group | Control | 634* | _ | ( | С | С | С | С | С | С | _ | С | | |
| 3 | Control | 034 | C | ر | C | C | C | J | J | J | J | J | | |
| | Total: 1900 (63300 VRC01 30 mg/kg; 633 VRC01 10 mg/kg; 634 control) | | | | | | | | | | | | | |

<sup>\*</sup> Due to the randomization scheme, the numbers of vaccine and control recipients may differ slightly.

## **Participants**

1900 women in sub-Saharan Africa aged 18-40 who are at risk of HIV-1 infection; 2:1 active:control allocation; total approximately 1268 VRC01 mAb, 634 control

<sup>\*</sup> Week 80 is the last study visit for the primary endpoint analysis of prevention efficacy.

<sup>+</sup> Week 104 is the last study visit for the co-primary endpoint analysis of safety and tolerability.

#### Design

Multicenter, randomized, controlled, double-blind trial

## **Duration per participant**

24 months of scheduled clinic visits

## **Estimated total study duration**

60 months (includes enrollment and follow-up, including follow-up for HIV-infected participants)

## Study product providers

Dale and Betty Bumpers Vaccine Research Center (VRC), NIAID, NIH, DHHS (Bethesda, Maryland, USA)

#### Core operations

HIV Vaccine Trials Network (HVTN) Leadership Group/Core Operations Center, Fred Hutchinson Cancer Research Center (FHCRC) (Seattle, Washington, USA)

HIV Prevention Trials Network (HPTN) Leadership and Operations Center (LOC), FHI360 (Durham, North Carolina, USA)

## Statistical and data management center (SDMC)

Statistical Center for HIV/AIDS Research and Prevention (SCHARP), FHCRC (Seattle, Washington, USA)

DF/Net Research (Seattle, Washington, USA)

#### **Endpoint assay laboratories**

- University of Washington Virology Specialty Laboratory (UW-VSL) (Seattle, Washington, USA);
- Duke University Medical Center (Durham, North Carolina, USA)
- FHCRC/University of Washington (Seattle, Washington, USA)
- South Africa Immunology Laboratory, National Institute for Communicable Diseases (SAIL-NICD) (Johannesburg, South Africa)
- HIV Sero-Molecular Laboratory, National Institute for Communicable Diseases (HSML-NICD) (Johannesburg, South Africa)

- NIAID Vaccine Immune T-Cell Antibody Laboratory (NVITAL) (Gaithersburg, Maryland, USA)
- (NIAID) Vaccine Research Center (VRC) (Bethesda, Maryland, USA)
- HPTN Laboratory Center, Johns Hopkins University (JHU) (Baltimore, Maryland, USA)
- University of Cape Town (UCT) (Cape Town, South Africa)
- University of Colorado, Denver (UC Denver) (Denver, Colorado, USA)

## Study sites

Clinical Research Sites (CRSs) to be specified in the Site Announcement Memo

#### Safety monitoring

HVTN 703/HPTN 081 Protocol Safety Review Team (PSRT); NIAID Data and Safety Monitoring Board (DSMB)

#### 1.1 Protocol Team

#### Protocol leadership

Chair

leader

ChairLawrence Corey<br/>HVTN, FHCRCStatisticians<br/>SCHARP, FHCRCAllan DeCamp<br/>SCHARP, FHCRC206-667-6770206-667-7892

lcorey@fhcrc.org adecamp@scharp.org

Myron Cohen Peter Gilbert

HPTN, University of SCHARP, FHCRC North Carolina 206-667-7299 pgilbert@scharp.org

mscohen@med.unc.edu

Cochairs Srilatha Edupuganti Michal Juraska
Emory University SCHARP, FHCRC
404-712-1434 206-667-5568

sedupug@emory.edu mjuraska@scharp.org

Nyaradzo Mgodi Deborah Donnell

UZ-UCSF Collaborative SCHARP, FHCRC

Research Programme, 206-667-5661

Harare, Zimbabwe deborah@scharp.org 263-4-704890

Protocol Team Shelly Karuna Medical officers Margarita Gomez Lorenzo

HVTN Core, FHCRC Vaccine Research Program 206-667-4355 (VRP), DAIDS, NIAID

skaruna@hvtn.org 240-627-3510 gomezmm@niaid.nih.gov

HVTN John Hural David Burns

Laboratory lead HVTN Laboratory Prevention Sciences Program

 Program
 (PSP), DAIDS, NIAID

 206-667-1683
 301-435-8896

 jhural@hvtn.org
 burnsda@niaid.nih.gov

#### Other contributors to the original protocol

nmmgodi@uz-ucsf.co.zw

HVTN Core<br/>medical monitorShelly KarunaDAIDS Protocol<br/>pharmacistKatherine ShinMedical monitorHVTN Core, FHCRCpharmacistDAIDS, NIAID<br/>240-627-3047

BioethicsMark BarnesHVTN RegionalSimba TakuvaconsultantHPTN Ethics Workingmedical liaison,HVTN Core, FHCRCGroupSouthern Africa

HVTN/HPTNKen MayerHVTN RegionalKeitumetse DiphokoConsultativeFenway Health, Boston,clinical safetyHCRISA

investigators USA liaison for Africa
LaRon Nelson HVTN Regional Robert De La Grecca

Univ. of Rochester, Rochester, NY, USA South America Rochester Roc

Manuel VillaránHVTN ClinicalMaija AndersonIMPACTA, Lima, Perusafety specialistHVTN Core, FHCRC

Sinead DelanyMoretlwe

HVTN Statistical
research associates

Nidhi Kochar
SCHARP, FHCRC

Wits Reproductive Health and HIV Institute, Johannesburg,

South Africa

## HVTN 703/HPTN 081 Version 4.0 / December 14, 2017

| Product<br>developer<br>representatives | John Mascola<br>VRC | | Abby Isaacs<br>SCHARP, FHCRC |
|---|---|---|---|
| | Barney Graham<br>VRC | | Jing Wang<br>SCHARP, FHCRC |
| | Julie Ledgerwood<br>VRC | HVTN Social<br>behavioral<br>scientist | Michele Andrasik<br>HVTN Core,<br>FHCRC |
| HVTN<br>Laboratory<br>Program<br>representatives | On Ho<br>HVTN Laboratory<br>Program, FHCRC | HPTN LOC<br>director | Nirupama Sista<br>HPTN LOC, FHI360 |
| | David Montefiori<br>HVTN Laboratory<br>Program, Duke Univ.,<br>Durham, NC, USA. | HPTN Clinical<br>research<br>managers | Philip Andrew<br>HPTN LOC, FHI360 |
| | Robert Coombs<br>University of Washington<br>Virology Specialty<br>Laboratory, Seattle, WA,<br>USA | | Elizabeth Greene<br>HPTN LOC, FHI360 |
| HPTN<br>Laboratory<br>Center<br>representatives | Susan Eshleman<br>HPTN Laboratory Center<br>(LC), Johns Hopkins<br>Univ., Baltimore, MD,<br>USA | HVTN Clinical<br>trials manager | Carissa Karg<br>HVTN Core,<br>FHCRC |
| | Vanessa Cummings<br>HPTN LC, Johns Hopkins<br>Univ. | HPTN SDMC<br>Associate director | Lynda Emel<br>SCHARP, FHCRC |
| | Estelle Piwowar-Manning<br>HPTN LC, Johns Hopkins<br>Univ. | HVTN SDMC<br>Program manager | Gina Escamilla<br>SCHARP, FHCRC |
| HVTN<br>Regulatory<br>affairs | Megan Brandon<br>HVTN Core, FHCRC | HVTN Protocol<br>development<br>manager | Carter Bentley<br>HVTN Core,<br>FHCRC |
| Clinic<br>coordinators | Debora Dunbar<br>University of<br>Pennsylvania,<br>Philadelphia, PA, USA | HVTN<br>Communications<br>unit representative | Jim Maynard<br>HVTN Core,<br>FHCRC |

#### HVTN 703/HPTN 081 Version 4.0 / December 14, 2017

Ana Patricia Rimachi HVTN Community Gail Broder HVTN Core, Quiroz engagement unit Asociación Civil Selva representative **FHCRC** Amazónica, Iquitos, Peru Christie Heiberg HPTN Community Jonathan Lucas Desmond Tutu HIV HPTN LOC, FHI360 program Centre, University of Cape associates Town, Cape Town, South Africa Mark Hubbard Community Jontraye Davis Advisory Board Vanderbilt University, HPTN LOC, FHI360 (CAB) members Nashville, TN, USA Likhapha Faku DaShawn Usher Community HVTN Global CAB educator/recruiter New York Blood Member at Large, Center, New York, Rustenberg, South Africa NY, USA Jim Wick Luciana Kamel Bridge HIV. San Instituto de Pesquisa Francisco, CA, USA Clinica Evandro Chagas (IPEC) HVTN Technical Erik Schwab HVTN Core, editor **FHCRC** 

## 2 Background

## 2.1 Rationale for trial concept

Effective biomedical interventions are needed to reduce the acquisition of HIV. The global HIV-1 epidemic continues and while many countries have made progress toward leveling HIV prevalence over the last few years, micro-epidemics of infection continue to occur in nearly all regions, even in countries possessing the full toolkit of proven prevention approaches [1-4]. The World Health Organization (WHO) estimates that there were 2 million new HIV infections worldwide in 2014, the last year for which data are available [5].

Antiretroviral drugs (ARVs) have been shown to be effective for HIV prevention in serodiscordant couples when administered to HIV-infected individuals as treatment as prevention (TasP) and clinical trials are now underway to evaluate the efficacy of TasP at a population level [6]. ARVs have also been shown to be effective as pre- or post-exposure prophylaxis (PrEP or PEP) [7]. At present daily oral emtricitabine (FTC)/tenofovir disoproxil fumarate (TDF) (Truvada) is the only drug approved for PrEP use, but this drug combination has significant known side effects [8]. The requirement for daily use and the side effect profile have made adherence to this drug regimen challenging, especially over long periods of time [9]. As a consequence, the capacity of currently available ARV regimens to reduce HIV incidence or prevalence is less than optimal. Furthermore, sustained use of ARVs for HIV prevention will increase the already significant burden of ARV manufacturing and delivery for HIV treatment, especially in countries bearing the highest burden of HIV disease. For these reasons, a biomedical HIV prevention approach that exhibits sustained activity over an extended time period, that has a safety profile acceptable for healthy persons, and whose effectiveness is less dependent upon individual adherence, is still needed.

An alternative approach to prevention and/or treatment of infectious diseases is passive administration of antibodies, a strategy that has been employed for more than 100 years against diverse disease targets and that is still used for hepatitis A and B prophylaxis [10,11] and for PEP for rabies, measles, varicella zoster, and other infectious diseases [12]. Most notably, palivizumab has been used for respiratory syncytial virus (RSV) prophylaxis in pre-term and other high-risk infants for nearly two decades. In 1998, a multinational, randomized controlled trial showed that palivizumab administered during the RSV season reduced RSVassociated hospitalizations by 39-78% in premature infants and in children with bronchopulmonary dysplasia [13]. Subsequent studies have confirmed palivizumab's safety, efficacy, and clinical benefit for infants at high risk for RSV infection [14,15]. Hence, palivizumab serves as a model for the use of mAbs to block a mucosally-acquired infection. Significantly, passive administration of this antibody has also set a standard by which candidate RSV vaccines are evaluated, by defining antibody levels that effectively inhibit fusion by RSV. This precedent has informed the conceptual framework for this study.

Over the past several years, there has been a concerted and notably successful effort to isolate broadly neutralizing antibodies (bnAb) to HIV-1 from chronically infected donors [16-32]. Subsequent research has provided considerable insight into the sites these antibodies target on HIV-1 and their functionality (ie, the mechanisms by which they neutralize the virus) [19,20,29,33]. This research has informed efforts to design recombinant protein immunogens that can elicit such antibodies [34-37], prompting optimism that vaccines that elicit bnAbs against HIV-1 can be developed [35,38]. In addition, the availability of bnAbs against HIV opens the exciting possibility of antibody-mediated prevention (AMP) of HIV infection.

The Vaccine Research Center (VRC), NIAID, NIH has developed VRC01, a broadly neutralizing human mAb that targets the HIV-1 CD4 binding site [18]. This mAb was originally discovered in a participant infected with HIV-1 for more than 15 years who maintained viral control without use of antiretroviral therapy (ART) [39]. VRC01 has the capacity to neutralize a broad range of HIV-1 strains in vitro (Section 2.3) and has conferred protection against simian-human immunodeficiency virus (SHIV) challenges in nonhuman primate (NHP) studies [40-49] (Section 2.8). It has an acceptable safety profile, as seen in previous phase 1 studies (Section 2.9).

In addition to potentially developing a new HIV prevention modality, evaluating the preventive efficacy of mAbs can be expected to inform future HIV vaccine development. An important requisite for designing vaccines that elicit bnAbs is determining the level of neutralizing activity required to achieve a reasonable degree of protection in humans. It will also be important to know whether such levels vary by route of infection or neutralizing sensitivity of the infecting isolate. Notably, VRC01 contains the Fc portion of IgG1 and has demonstrated other effector functions. Evaluating the role of antibody-mediated effector functions (eg, antibody-dependent cellular cytotoxicity [ADCC], antibody-dependent cellular phagocytosis [ADCP], antibody-dependent cell-mediated viral inhibition [ADCVI], antibody-mediated virion capture in mucus, or inhibition of viral translocation across epithelial barriers, etc.) in protection is also of critical importance (see, eg, [50-53]).

Although it is not anticipated that this trial will lead directly to licensure, further assessment of this VRC01 product will depend on the results of this and other studies.

#### 2.2 bnAbs to HIV-1

The last several years have seen a marked increase in the number of well-characterized bnAbs to HIV-1. Figure 2-1 shows the names and binding sites of many of these.



Figure 2-1 Neutralizing antibody epitopes on native Env timer

As shown in Figure 2-2, several of these antibodies have shown considerable breadth of neutralization in in vitro testing.



Figure 2-2 Percentage of viruses neutralized at different serum concentrations. (A) < 50 mcg/mL; (B) < 10 mcg/mL; (C) < 1 mcg/mL [32,49,54-57].

Two antibodies to the CD4 binding site of the HIV-1 envelope, VRC01 and 3BNC117 (highlighted in red in Figure 2-1), have entered phase 1 clinical trials.

#### 2.3 VRC01: VRC-HIVMAB060-00-AB

VRC01 is a human mAb, developed by VRC/NIAID/NIH, directed against the CD4-binding site of HIV-1. The bulk lot of the drug substance was manufactured under current Good Manufacturing Practice (cGMP) conditions in a Chinese Hamster Ovary (CHO) cell line and the drug product vials were filled and labeled at the VRC Vaccine Pilot Plant (Frederick, Maryland, USA) operated by Leidos Biomedical Research, Inc. (formerly SAIC-Frederick), Frederick, Maryland (USA). Product is vialed at a concentration of 100 mg/mL VRC01 in formulation buffer containing 25 mM sodium citrate, 50 mM sodium chloride, and 150 mM Larginine hydrochloride at pH 5.8. VRC01 was produced using recombinant DNA technology. Briefly, using polymerase chain reaction (PCR) amplification and cloning of the heavy and light chain variable region genes, a mAb was initially isolated from a single B cell from an HIV-1—infected subject who displayed bnAbs. VRC01 is an IgG1 antibody and is highly somatically mutated from the germ-line precursor.

The VRC01 antibody has been well characterized preclinically and has demonstrated favorable characteristics in potency and half-life [19]. In addition, it has demonstrated protection in NHP challenge studies (see Section 2.8.1 below). Figure 2-2 shows graphically the impressive breadth of VRC01, with 90% of 190 HIV-1 isolates across all clades tested showing sensitivity to neutralization by VRC01. As shown in Figure 2-3, VRC01 has a 50% inhibitory concentration (IC<sub>50</sub>) of < 50 mcg/mL against 91% of primary HIV-1 isolates and IC<sub>50</sub> < 1 mcg/mL against 72% of HIV-1 isolates. Notably, the IC<sub>50</sub> for the vast majority of HIV-1 isolates tested is < 1 mcg/mL; the geometric mean IC<sub>50</sub> for HIV-1 strains from all clades tested is 0.33 mcg/mL.



| Virus clade | Number of viruses | IC <sub>50</sub> < 50 mcg/mL | IC <sub>50</sub> < 10 mcg/mL | IC50 < 1 mcg/mL |
|---|---|---|---|---|
| Α | 22 | 100% | 100% | 95% |
| В | 49 | 96% | 94% | 80% |
| С | 38 | 87% | 84% | 66% |
| D | 8 | 88% | 88% | 50% |
| CrRF01_AE | 18 | 89% | 83% | 61% |
| CRF02_AG | 16 | 81% | 75% | 56% |
| G | 10 | 90% | 90% | 90% |
| CRF07_BC | 11 | 100% | 91% | 45% |
| Other | 18 | 83% | 83% | 78% |
| Total | 190 | 91% | 88% | 72% |

Figure 2-3 CD4 binding site antibody: VRC01 [18,19]

Details on VRC01 composition and manufacturing can be found in the investigator's brochure (IB).

## 2.4 Trial design rationale

Several considerations inform the design of this test-of-concept phase 2b study. The first is to establish that passive administration of bnAbs can block HIV acquisition. Based on data from in vitro neutralization studies, the NHP challenge studies described below, and pharmacokinetic (PK) data from the phase 1 clinical trials VRC 602 and HVTN 104, the doses selected are designed to elucidate the activity of the antibody across a range of serum concentrations in a diverse population of at-risk persons in multiple geographic regions of the world. The study is designed to define the optimal dosage for widespread use of the antibody or its subsequent derivatives as well as to benchmark the types of effector functions associated with efficacy, thus constituting an important bridge to other types of bnAbs and other bnAb delivery systems.

Inclusion of different doses (ie, in a 3-arm study) is important for a number of reasons. First, while the in vitro and NHP challenge data are informative, the VRC01 antibody serum level required to provide protection against HIV-1 infection in humans is unknown. Some studies suggest that transmitted-founder HIV strains may be more sensitive to neutralization than other strains (particularly by VRC01) [58,59], and therefore potentially susceptible to even lower antibody

doses than those suggested by SHIV challenge studies in NHP. It must also be recognized that the lowest challenge doses used in the NHP model likely exceed natural exposure in the majority of transmissions in humans.

Defining the lowest efficacious VRC01 dose is essential for establishing a target product profile (TPP), including optimal dosing for clinical use, for this antibody and its derivatives. Typically, higher doses of drug products are associated with lower tolerability due to side effect profiles or operational features such as length of drug administration time (eg, IV infusion time). At present the high dose (30 mg/kg) cannot be administered subcutaneously (SC), limiting the feasibility of long-term clinical use. The extreme difficulty of scaling IV administration to the populations most in need of protection against HIV infection and the complexity and cost of manufacturing mAbs would severely limit implementation of this potentially important HIV prevention tool if higher doses are required for efficacy. Therefore, it is important to evaluate the efficacy achieved at lower antibody concentrations. That lower doses of mAbs may prevent HIV acquisition is supported by the high percentage of isolates susceptible in vitro to antibody concentrations as low as 1 mcg/mL of VRC01, 1/10 the mean trough level anticipated with 30 mg/kg VRC01 dosing every 8 weeks.

Including a range of doses in this study also facilitates evaluation of antibody effector functions, in addition to neutralization, that are associated with protection (eg, virion binding, ADCC, ADCP). Note that the relationship of these important functions to neutralization is not linear and therefore cannot be inferred directly. This information will have important implications for the development of other bnAbs and other biomedical HIV prevention modalities.

Hence, in addition to providing a test of concept for AMP for HIV, if breakthrough infections are observed, the data generated by this trial will help guide development of functionally-enhanced mAbs and of long-term delivery strategies (eg, vaccine immunogen or vectored immunoprophylaxis). This trial affords a unique opportunity to correlate serum antibody levels and the potency of effector functions with protective efficacy in a trial in which these parameters can be measured close to the time of HIV acquisition, providing benchmarks for vaccine development and helping define "targets" of antibody effector mechanisms for protein or viral vector based vaccines. The data will also provide critical information by which to identify which NHP models (eg, SHIV challenge stocks) are most predictive of bnAb efficacy in humans.

#### 2.4.1 Cohort selection

The study will be conducted in 1900 sexually active women in sub-Saharan Africa. The trial sample size is designed to provide 90% power to detect a prevention efficacy (PE) of 60% (rejecting the null hypothesis of 0% PE), based on reasonable assumptions regarding background HIV-1 incidence, retention, and frequency of infusions.

The cohort for this study was selected based on regional epidemiological data. There were approximately 24.7 million people living with HIV in sub-Saharan Africa in 2013, representing over 70% of the global HIV burden. HIV prevalence in sub-Saharan Africa continues to be higher than anywhere else in the world. Women in sub-Saharan Africa are disproportionately impacted, accounting for nearly 60% of all people living with HIV in the region in 2013. There are approximately 16 million women  $\geq$  15 years old who are living with HIV; 80% live in sub-Saharan Africa. Young women 15-24 years old in sub-Saharan Africa are twice as likely as young men to be living with HIV, with acquisition rates among heterosexual women as high as 6-8% annually in some locations [60]. In recent clinical trials in southern Africa, annual HIV-1 incidence rates of 1.9-9.1% have been observed among sexually-active women [61-67]. Yet, there are currently no biomedical HIV prevention tools proven to protect women at high risk of HIV infection in sub-Saharan Africa. Fortunately there are biomedical tools with demonstrated HIV prevention success for men at high risk of HIV infection in sub-Saharan Africa (eg, medical male circumcision, oral PrEP). With this context in mind, and recognizing that we have limited resources for this trial that prevent us from addressing the HIV prevention needs of all populations, this trial in sub-Saharan Africa is designed to: evaluate the effectiveness of AMP, inform future research on AMP and related prevention approaches (eg, HIV vaccines), and develop a biomedical tool to reduce the disproportionate HIV incidence among sub-Saharan African women. Conducting the study in heterogeneous cohorts of overall lesser risk (eg, men as well as women in sub-Saharan Africa), would require larger sample sizes in order to answer the study questions. We look forward to extending what we learn in this trial to other cohorts, including men at high risk of HIV infection in sub-Saharan Africa.

We note that a parallel study assessing the safety and preventive efficacy of VRC01 is being conducted among 2700 men and transgender persons who have sex with men or transgender persons in the Americas and Europe. That study, designated HVTN 704/HPTN 085, will be conducted over approximately the same time period as HVTN 703/HPTN 081.

#### 2.4.2 Dose and schedule

An equal number of study participants will be randomized to receive VRC01 mAb by IV infusion at a dose of 10 mg/kg or 30 mg/kg every 8 weeks, or to receive control infusions every 8 weeks. The 8 week infusion interval represents approximately 4 half-lives of the study drug (half-life ~14 days based on previous clinical testing; see the IB).

Infusions will continue for 72 weeks for all groups, with a final primary follow-up visit (without infusion) at week 80 and an additional 24 weeks of follow-up without infusions. Hence, the study duration for each participant is 104 weeks (2 years).

Projected serum concentrations of VRC01 are shown in Figure 2-4. This figure plots predicted median VRC01 serum concentrations over time based on PK

models for VRC01 administered at 10 mg/kg every 8 weeks (Panel A) and for VRC01 administered at 30 mg/kg every 8 weeks (Panel B). The plots include shaded regions illustrating time regions where the study participants have serum concentrations in low, medium, and high ranges. Based on in vitro neutralization studies (see Section 2.3) and NHP challenge studies (see Section 2.8.1) and assuming that these accurately predict protection in humans, the expected trough levels of VRC01 are projected to be an order of magnitude higher than the levels required to protect against a majority of circulating HIV-1 strains.

See Section 2.9.3 and Figure 2-9 for VRC01 serum concentrations reported to date for participants administered 10mg/kg and 30mg/kg of VRC01 every 8 weeks in HVTN 104.



10 mg/kg VRC01 group: Predict (50%, 40%, 10%) PYRs in (Low, Medium, High) zones



30 mg/kg VRC01 group: Predict (10%, 40%, 50%) PYRs in (Low, Medium, High) zones

Figure 2-4 Predicted VRC01 serum concentrations over time. Panel A: Predicted VRC01 median serum concentration over time (solid lines) for 10 mg/kg IV infusions of VRC01 at Weeks 0, 8, 16, 24, 32, 40, 48, 56, 64, 72, with 95% confidence intervals (CI) (dashed lines). The shaded regions classify the serum concentration marker S(t) into high, medium, and low ranges based on the cut-points 10 and 50 mcg/mL. Panel B: Predicted median VRC01

serum concentration over time for 30 mg/kg IV infusions of VRC01 at Weeks 0, 8, 16, 24, 32, 40, 48, 56, 64, 72. The shaded regions classify the serum concentration marker S(t) into high, medium, and low ranges based on the cut-points 10 and 50 mcg/mL. PYR = personyear at risk.

There is a substantial overlap in the mAb concentrations between the low and high dose groups during a considerable period of time after each infusion. This is shown in Figure 2-5.



Figure 2-5 Projected overlap in serum VRC01 concentrations and PYRs of HIV exposure between high dose (30 mg/kg) and low dose (10 mg/kg) VRC01 administration

#### 2.4.3 Choice of control

Sodium Chloride for Injection 0.9%, USP (referred to as Control) administered IV at a volume of 150 mL will serve as an inert control.

Use of a placebo control in this trial is warranted based on the scientific and public health importance of the questions it seeks to answer, the necessity of a placebo control in order to assess VRC01 efficacy in preventing HIV-1 infection, and an acceptable risk/benefit ratio considering the minimal risk associated with the placebo control selected and its administration via a procedure commonly used in clinical care. In addition, the placebo control is essential to maintain double-blinding to ensure unbiased assessments of study product safety and efficacy, and the use of the placebo control is disclosed fully to study participants (see Section 10 of Appendix A). Hence, this trial meets the standards commonly required for ethical use of placebo controls in clinical trials [68-70].

### 2.4.4 HIV diagnostic testing

HIV diagnostic testing will be scheduled at least every four weeks and at any time following participant report of possible exposure during the study. See Section 8 for further detail on HIV-infection assessment. Participants who are diagnosed with HIV infection after enrollment will not receive additional infusions. Infusions will also be permanently discontinued for participants who have 2 reactive HIV tests, even if subsequent testing indicated that the participant is not HIV infected. Based on the schedule of testing, it is possible that a newly infected participant may receive an infusion of VRC01 (or Control). This does not appear to pose a safety risk for participants based on existing preclinical, clinical, and in vitro data. Specifically, passively-infused VRC01 given to NHP on Day 7 after SHIV SF162P3 infection reduces viremia and does not cause clinical harm (see IB). Additionally, passive transfer of neutralizing antibodies (at non-protective levels) prior to infection improved control of SHIV viremia and was associated with early nAb development in infected infant macaques [71]. Furthermore, VRC01 has been evaluated in viremic and aviremic HIV-infected participants (see Section 2.9.1). VRC01 administration is associated with statistically significant transient reductions in HIV viral load in adults with chronic HIV infection (see IB), and HIV variants that escape from in vitro VRC01 neutralization have reduced viral fitness [72]. Studies evaluating VRC01 in acutely infected subjects are being initiated based on these data.

## 2.4.5 Trial monitoring

As this is the first large-scale phase 2b study with IV administration of a biomedical intervention for prevention of sexual HIV-1 transmission, the trial design includes an early feasibility check. After approximately 120 participants have completed the Week 32 visit, a treatment-blinded analysis of infusion feasibility will be conducted and reported to the DSMB. Enrollment of the remaining study participants will be deemed feasible if  $\geq$  80% of those 120 participants remain engaged in the trial and have not declined further infusions. Enrollment will not be paused for this feasibility assessment.

In addition to the feasibility assessment, the study design includes sequential monitoring for potential harm, non-efficacy, high efficacy, and futility for assessing prevention efficacy. Following similar monitoring procedures developed and implemented for the HVTN 505 phase 2b vaccine efficacy trial, potential harm monitoring is maximally vigilant by testing for a higher HIV infection rate among VRC01 recipients than in the control group after each HIV infection and providing the results to the DSMB after each infection starting with the 20<sup>th</sup> total infection pooled over the study groups. This ensures that any potential risk of increased HIV acquisition (negative prevention efficacy [PE]) would be detected as early as possible, such that infusions of the mAb could be discontinued expeditiously. In addition, the operating characteristics of the trial (Figure 4-3 and Table 4-2) show that this potential harm-monitoring approach has a low risk of stopping the study prematurely if the true PE is 0% or higher. The

non-efficacy monitoring is conducted approximately every 6 months, and is based on a trigger specified in the study monitoring plan.

At the 6-month intervals, statistical interim analysis reports are provided to the DSMB. Gilbert et al [73] describe the conceptual approach to the sequential monitoring of PE, where the implementation for the current trial is slightly different. Additional information is provided in Section 4.7. Full details regarding implementation of monitoring for this trial are contained in a separate trial monitoring plan.

## 2.5 Combination prevention for HIV acquisition

In 2013, sub-Saharan Africa bore more than 70% of the global burden of HIV infections and women accounted for nearly 60% of all those living with HIV in the region. Of all the women in the world who live with HIV, 80% live in sub-Saharan Africa [60]. Hence it is essential that approaches to reducing HIV infection risk be made available to the women participating in this clinical trial.

Participants in all arms of the study will be provided with a comprehensive HIV prevention package consistent with all HIV prevention clinical trials. This package includes evidence-based behavioral risk reduction counseling [74], free condoms and lubricant, counseling and referral for postexposure prophylaxis (PEP) when indicated, and, where appropriate, access to oral drugs for pre-exposure prophylaxis (PrEP, see below). These activities can be expected to reduce HIV acquisition below historical levels. The contribution of these efforts will be monitored. Further details on these efforts are provided in the HVTN 703/HPTN 081 Study Specific Procedures (SSP) and the HVTN 703/HPTN 081 website. It should be emphasized that because the benefit of VRC01 monoclonal antibody is unknown, subjects in each arm of the study will receive the same prevention package.

## 2.5.1 Evidence for PrEP efficacy

Multiple studies in multiple settings have established that daily or pericoital FTC/TDF can be highly efficacious in preventing HIV infection in MSM [7,75-79]. However, aside from women in HIV-discordant couples [80], comparable efficacy has not as consistently been demonstrated in trials evaluating topical or oral tenofovir (TFV)-based regimens among at-risk women in sub-Saharan Africa. While the CAPRISA 004 trial demonstrated a 39% reduction in HIV infection with pericoital application of TFV 1% vaginal gel among at-risk women in South Africa [65], efficacy was not seen in the larger, more recent FACTS 001 trial conducted among young South African women [81]. In 2011 the FEM-PrEP trial was stopped early because of lack of efficacy of once daily oral FTC/TDF among at-risk women in Kenya, South Africa, and Tanzania [66]. In 2011 the VOICE trial, conducted in Uganda, South Africa, and Zimbabwe, reported no efficacy of once daily oral TDF or TFV 1% gel; in 2013, this trial reported no efficacy for once daily oral FTC/TDF [82]A meta-analysis of these trial results

shows that effectiveness correlates strongly with PrEP adherence (see Figure 2-6)[83]; because adherence was poor in the trials that generated the largest number of infection events (FEM-PrEP and VOICE), overall PrEP efficacy in southern African trials appears particularly disappointing. However, in addition to adherence, other factors may also contribute to the conflicting results observed in women, including differences in the study populations (discordant couples versus uninfected individuals), differing demographic and behavioral characteristics, prevalent HIV subtypes, differing transmission modes (mucosal versus parenteral), and underlying host factors such as genital tract inflammation and/or copathogens [83]. In addition, pharmacokinetic studies report lower concentrations of PrEP drug in vaginal as compared to rectal mucosa [84], suggesting that efficacy mediators may differ between men and women and that PrEP efficacy may be more sensitive to adherence in women than in men [85].

Figure 2-6 Forest plot showing point estimates and 95% confidence intervals of PrEP effectiveness, meta-analysis estimates, and meta-analysis regression results for major PrEP trials in women [83]



## 2.5.2 Evolving PrEP guidelines

Guidelines for use of fixed dose FTC/TDF for HIV prophylaxis have evolved rapidly. In 2011, the US Centers for Disease Control and Prevention (CDC) issued interim guidelines for use of FTC/TDF as PrEP for high-risk MSM [86]. In 2012, the US FDA approved FTC/TDF for HIV prophylaxis in persons at high risk for HIV infection. That same year, the World Health Organization (WHO) issued guidance on the use of PrEP for serodiscordant couples and for men and TG women who have sex with men [87]. In 2014, the US CDC issued a further PrEP guidance document and a Clinical Provider Supplement confirming the previous recommendation of FTC/TDF PrEP as a prevention option for sexually-active adult MSM at substantial risk of HIV acquisition and expanding the

recommendation to include adult heterosexually active persons at substantial risk of HIV acquisition [88,89]. PrEP has since been incorporated into WHO guidelines for ARV use for HIV treatment and prevention [90,91]; a revised and more comprehensive WHO PrEP guideline is anticipated in 2016. Notably, the Republic of South Africa and Kenya approved FTC/TDF for use as PrEP in December 2015.

#### 2.5.3 Operationalizing PrEP access in sub-Saharan Africa

Although the WHO released updated guidance documents on universal test and treat and recommendations for PrEP in late 2015, most countries in this region are in the process of regulating antiretrovirals for prevention, and it is envisaged that PrEP use will be scaled up over time in the ensuing 5-10 years. Going to scale in a generalized heterosexual epidemic will require significant financial investment. For this reason, countries are currently investigating the fiscal impacts of the new guidelines and are in discussions to develop demonstration projects to evaluate mechanisms for the successful roll out of PrEP to key populations. The threshold for PrEP roll-out in-country will depend on: 1) the epidemiology context; 2) availability of resources; 3) the cost of the intervention; 4) the feasibility of delivering this service; and 5) demand. There are limited donor-driven demonstration PrEP projects in Africa and countries are working closely with PEPFAR and the Global Fund to design demonstration projects that are potentially sustainable in the long-term.

As an example, South Africa recently registered FTC/TDF for prevention and is developing guidelines for its use. These guidelines stipulate that prep must be delivered in the service delivery setting with the main guiding principal of informed and voluntary choice and equitable access. There is a commitment by the Republic of South Africa to strategically expand the reach and coverage of the antiretroviral programme in such manner of it being equitable and non-discriminatory. Although FTC/TDF is not yet available in the public sector for use in prevention, the South African government through the National Department of Health (NDOH) intends to conduct demonstration projects, in conjunction with key donors, in key populations such as sex workers and MSM, as well as in geographic locations that have a high burden of HIV. However, FTC/TDF for prevention is not yet on the Essential Drug List, which is a prerequisite for use in the public sector through which the vast majority of South Africans secure health care.

Currently an investment case evaluating the new WHO guidelines is being undertaken by the South African government. While the investment case for universal test and treat is clear, and this will be rolled out as a priority, the investment case for PrEP is less certain and is being evaluated. Initially the NDOH plans to evaluate PrEP in key population groups such as sex workers and MSM. The roll-out of PrEP in young women is more complex and the NDOH is developing guidelines as to how this may occur.

For these reasons, the protocol team plans to work collaboratively with national regulatory and other government agencies to develop mechanisms for PrEP access that are supportive of and consistent with national priorities and strategic objectives in the several sub-Saharan African countries where this study is being implemented.

Given the potential of FTC/TDF to prevent HIV acquisition, it could be argued that substantial uptake of PrEP could prevent the HVTN 703/HPTN 081 trial from detecting any benefit of VRC01 beyond the universal prevention package. This possibility is addressed in the sample size and power calculations (see Section 4.4) and in plans for trial monitoring by the DSMB (see Section 4.7 and, specifically, Section 4.7.3). If the background HIV incidence rate is too low to support evaluation of VRC01 prevention efficacy, the DSMB will detect this and will make recommendations to the team accordingly. The study team will monitor PrEP availability and roll-out in-country; and within the protocol, evaluate individual use via questionnaires and blood drug levels. In support of a comprehensive package of prevention, PrEP will be discussed in the informed consent process, in risk reduction counseling sessions, and referral systems into demonstration projects, health service delivery settings, and the private sector will be developed to support those who wish to access PrEP.

## 2.6 Plans for future product development and testing

VRC01 is considered to have potential value for both preventive and therapeutic purposes across broad geographic regions of the HIV-1 epidemic. The product was initially evaluated in phase 1 studies to characterize PK and distribution in HIV-infected and HIV-uninfected adults (VRC 601 and 602, respectively; see Sections 2.9.1 and 2.9.2) and PK and safety for multiple administrations under several route and dosing regimens are being evaluated currently (HVTN 104; see Section 2.9.3). In parallel, IMPAACT P1112 will evaluate the safety of VRC01 in high-risk infants born to HIV-infected mothers; data from this study will support a future evaluation of the efficacy of VRC01 administered to high-risk infants shortly after birth and continued through the period of breast-feeding for prevention of mother-to-child HIV transmission (PMTCT).

The development of VRC01 for clinical use depends on a number of factors, the most critical of which is the level of efficacy demonstrated by the current study. If the antibody proves to be highly effective at preventing HIV-1 infection, its development will depend on identifying a partner able to provide large-scale manufacturing. Other factors that could influence advanced development of VRC01 or similar monoclonal antibodies include: 1) the potential for improving the potency of the product to allow use at a lower dose and perhaps by an SC route, 2) the potential for increasing the half-life of the product to allow less frequent dosing, and 3) the potential to use VRC01 or its derivatives in combination with other neutralizing mAbs to increase potency and breadth of coverage. Efforts to address these issues are proceeding in parallel with the

current study, but the outcome of the current study will have the greatest influence on the future clinical use of VRC01 in adult prevention or PMTCT.

## 2.7 Preclinical safety studies

## 2.7.1 Preclinical toxicology and PK study of VRC01 in rats

Table 2-1 Summary of preclinical studies

| Study<br>number | Product | Type of study | Animal | N | Dose<br>groups | Route | Schedule |
|---|---|---|---|---|---|---|---|
| SRI No<br>M896-11 | VRC-<br>HIVMAB060-<br>00-AB | Repeat dose toxicity | Sprague-<br>Dawley rats | 10m, 10f<br>each<br>50m, 50f<br>total | Vehicle* 4mg/kg IV 40 mg/kg IV 400 mg/kg IV 40 mg/kg SC | IV &<br>SC | D1, D8 |
| SRI No<br>M896-11 | VRC-<br>HIVMAB060-<br>00-AB | Single-dose<br>PK | Sprague-<br>Dawley rats | 9m, 9f<br>each<br>27m, 27f<br>total | 4 mg/kg IV<br>40 mg/kg<br>IV<br>40 mg/kg<br>SC | IV &<br>SC | D1 |

<sup>\*</sup> Vehicle consists of VRC01 formulation buffer.

A repeat dose toxicity study of IV and SC administration and a single dose PK study was performed by SRI International (Menlo Park, CA) with VRC01 in male and female Sprague-Dawley rats in accordance with US FDA "Good Laboratory Practice (GLP) for Nonclinical Laboratory Studies" (Table 2-1). This study was conducted with a pre-GMP pilot lot of VRC01 manufactured at smaller scale using a similar purification process to that of the GMP clinical grade drug product.

For the safety assessment, various doses of VRC01 (4 mg/kg, 40 mg/kg, or 400 mg/kg) or a comparable control vehicle was administered by tail vein infusion on Days 1 and 8 to Groups 1 through 4, respectively. An additional group (Group 5) received 40 mg/kg VRC01 via SC administration to the dorsal scapular region on Days 1 and 8. Each group contained 10 male and 10 female rats. Five animals of each sex were sacrificed on Day 9, one day after the second administration; the remaining animals were sacrificed on Day 30, 22 days after the second administration.

Results obtained showed that both routes of administration were well tolerated in the rats. All animals survived until their scheduled necropsy. No findings or changes were seen in clinical observation, body weight, food consumption, body temperature, infusion site irritation, hematology, coagulation, or organ weight evaluations that are attributed to administration of VRC01. VRC01 administration resulted in small, transient, dose-dependent increases in aspartate

aminotransferase (AST) and alkaline phosphatase (ALP) on Day 9. By Day 30, AST values had returned to normal, and ALP values were returning to normal.

Other than red discoloration of the administration site in one male in the SC group on Day 9, there were no other gross necropsy observations attributable to VRC01 administration. There were no histopathology findings that were considered related to IV administration of VRC01.

The pre-specified IV dose studied in rats was 400 mg/kg and SC was 40 mg/kg, which will greatly exceed the dose levels in the adult clinical studies. A "no observed effect level" (NOEL) was not determined in this study because transient elevations of AST and ALP were observed on Day 9 after IV administration and transient inflammation at the dose site was observed on Day 9 after SC administration. Because the elevated AST and ALP levels were transient and minor and did not correlate with histopathology findings, the no observed adverse effect level (NOAEL) for VRC01 by the IV route of administration in rats was 400 mg/kg, the highest dose used in this study.

For the PK analysis, 3 groups of rats (9 males and 9 females in each group) received VRC01 on Day 1 at 4 mg/kg IV, 40 mg/kg IV, and 40 mg/kg SC respectively. VRC01 levels in serum were determined using an enzyme-linked immunosorbent assay (ELISA) with samples collected predose from each animal and from an additional 3 males and 3 females to provide untreated control serum. Blood was collected from 3 rats/sex/PK group for a total of 4–5 collections per PK animal at each of the following postdose timepoints: 1, 4, 8, 24, 48, and 72 hours and 7, 14, 21, and 29 days.

VRC01 administration by the IV route resulted in dose-proportional exposure. The terminal elimination phase half-life was about 10 days, with clearance of approximately 20 mL/day/kg and volume of distribution that was about 0.28 L/kg, indicating that the drug was distributed primarily in the serum and eliminated slowly. VRC01 administration by the SC route resulted in mean peak serum levels at 7 days for male or 3 days for female animals. The maximum serum concentration and area under the concentration-time curve to the last timepoint values were lower when 40 mg/kg was administered by the SC route compared with the IV route. The bioavailability of 40 mg/kg VRC01 administered by the SC route was estimated to be 31.4% (males) and 42.3% (females). After the peak concentration of VRC01 was achieved in the SC group, the serum levels decreased much more rapidly from 7 to 14 days than they did in the IV groups, and VRC01 concentrations in the SC group were not quantifiable at timepoints after 14 days. These data indicate that clearance of VRC01 in rats was markedly enhanced when it was administered by the SC route. The development of antidrug antibodies that contribute to an increased rate of clearance is often observed in preclinical safety studies of protein-based test articles when they are not tested in the species of origin. Although immunogenicity was not examined in this study, the presence of such antibodies might have contributed to the increased rate of clearance of VRC01 after SC administration that was observed in this study [92,93].

# 2.7.2 Tissue cross reactivity GLP study of VRC01 with human tissues in vitro

A tissue cross-reactivity study of VRC01 using normal adult and neonatal human tissues in vitro (Testing Facility Study No. A255-12) was performed by Charles River Laboratories (Reno, NV) in accordance with U.S. FDA "Good Laboratory Practice for Nonclinical Laboratory Studies" (GLP). The tissue panels used as the test system for this *in vitro* cross-reactivity study included all of the tissues on the "Suggested list of human tissues to be used for immunohistochemical or cytochemical investigations of cross reactivity of monoclonal antibodies" in Annex I of the "European Medicines Agency Guideline on Development, Production, Characterization and Specifications for Monoclonal Antibodies and Related Product, Adopted by the Committee for Medicinal Products for Human Use on December 18, 2008" and all of the tissues recommended in the FDA/Center for Biologics Evaluation and Research "Points to Consider in the Manufacture and Testing of Monoclonal Antibody Products for Human Use (February 28, 1997)." In addition, the tissue cross-reactivity study used additional neonate/infant tissues suggested by the FDA to support future trials in infants.

To determine the cross-reactivity of VRC01 binding, VRC01 was applied to cryosections from a full panel of tissues from normal human adults and a limited panel of human neonatal tissues, immunohistochemically detected using a biotinylated rabbit anti-human IgG secondary antibody, and binding was visualized with a streptavidin-horseradish peroxidase complex and a diaminobenzidine chromogen substrate. VRC01 binding was evaluated at concentrations of 5 and 50 mcg/mL.

Specific VRC01 staining was not observed in any normal adult human or neonatal human tissues evaluated. Therefore, in vitro evaluation of cross-reactivity in tissue specimens did not identify potential tissue sites or organ systems to more thoroughly evaluate in subsequent preclinical studies, and it supports the future use of VRC01 in humans.

## 2.7.3 Other toxicity studies

Several in vitro studies were conducted to assess antibody activity against self-antigens by VRC01. Several anti-HIV neutralizing mAbs will cross-react to lipid or nuclear antigens or Hep-2 cells [94,95]. Anti-lipid binding activity is understandable when considering that the HIV-1 gp41 protein is membrane-spanning and the epitopes (MPER: Membrane-Proximal External Region) recognized by some mAbs (eg, 4E10 and 2F5) are membrane-proximal and likely extend into the membrane itself. Therefore, the ability (or lack thereof) of VRC01 to cross-react with lipids was assessed in collaboration with Dr. Barton Haynes of Duke University. Binding of antibody to cardiolipin was assessed in a luminescent assay, expressed in relative units. VRC01 was compared to 4E10, an anti-gp41 mAb known to bind to cardiolipin and nuclear antigens, and Synagis, a licensed anti-RSV antibody used as a negative control. Synagis is included

because it is the licensed mAb product most analogous to the intended clinical use of the VRC mAb [13].

Individual studies are summarized in Table 2-2. Unlike other anti-HIV neutralizing mAbs, VRC01 does not react to phospholipids or anti-nuclear antigens or Hep-2 cells. Additional details are provided in the IB.

Table 2-2 In vitro preclinical safety studies

| Study Purpose | Study Outcome |
|---|---|
| Assessment of anti-phospholipid reactivity | VRC01 does not react to phospholipids |
| Assessment of anti-nuclear antigen reactivity | VRC01 does not react with nuclear antigens |
| Assessment of anti-phospholipid characteristics by impact on activated partial thromboplastin time (aPTT) | VRC01 does not impact aPTT by binding phospholipids |
| Assessment of Binding to a Human Cell Line by Immunohistochemistry | Fluorescently labeled VRC01 does not bind<br>Hep-2 cells |

## 2.8 Nonhuman primate (NHP) studies of VRC01

Several non-Good Laboratory Practices (ie, non-GLP) studies of VRC01 have been completed in NHP to assess for preclinical evidence of potential efficacy for prevention of HIV infection. Table 2-3 summarizes the studies performed.

Table 2-3 Summary of NHP pharmacology and challenge studies

| Study | ndy Product Animal N Dose/Route | | Infusion schedule | Challenge route | Challenge stock/dose | Challenge schedule | | |
|---|---|---|---|---|---|---|---|---|
| Pharmacology | VRC01<br>(Pilot lot) | Rhesus<br>macaques | 4f<br>4f | 40 mg/kg IV<br>40 mg/kg<br>SC | Day 0 NA | | NA | NA |
| High-dose<br>challenge | VRC01<br>(Research<br>Grade) | Rhesus<br>macaques | 4m<br>4m<br>4m | 5 mg/kg IV<br>20 mg/kg IV<br>Human IgG<br>IV (control) | Day 0 | Intrarectal | SHIV-<br>SF162P3<br>(300<br>TCID <sub>50</sub> *) | Day 2 postinfusion |
| High-dose<br>challenge | VRC01<br>(Research<br>Grade) | Rhesus 4f Human IgO | | 20 mg/kg IV<br>Human IgG<br>IV (control) | Day 0 | Intravaginal | SHIV-<br>SF162P3<br>(300<br>TCID <sub>50</sub> ) | Day 2 postinfusion |
| High-dose<br>challenge | VRC01<br>(Research<br>Grade) | Rhesus<br>macaques | 6m<br>6m<br>4m<br>16m<br>14m | 20 mg/kg IV<br>5 mg/kg IV<br>1.25 mg/kg<br>IV<br>0.3 mg/kg<br>IV<br>Human IgG<br>IV (control) | Day 0 | Intrarectal | SHIV-BaL<br>(TCID <sub>50</sub><br>12,800 in<br>TZM-bl) | Day 2<br>postinfusion |

<sup>\*</sup>TCID<sub>50</sub> = 50% tissue culture infectious dose

In the pharmacology study, plasma and mucosal (ie, rectal, vaginal, and nasal) samples were collected at frequent intervals through Day 28. A dose of 40 mg/kg IV or SC in female rhesus macaques resulted in plasma concentration of VRC01

exceeding 50 mcg/mL in 7 of 8 animals at Day 14 and greater than 10 mcg/mL in 7 of 8 animals at Day 28.

Please see the VRC01 IB for more details.

#### 2.8.1 Protection against challenge in NHP models

Both neutralizing and non-neutralizing antibodies to HIV and SIV have been shown to protect against experimental challenge in the NHP model [40-42,96-100]. In these studies the degree of protection has varied with the neutralizing potency of the antibodies and with the dose, route, and sensitivity of the challenge stocks. Low antibody concentrations have in some instances been quite protective, especially against repeat low-dose mucosal challenges [44,45]. However, neutralization-resistant SHIVs have been developed and have been shown to be resistant to protection [101,102]. This has permitted estimation of neutralization titers for different mAbs against SHIVs representing a broad range of neutralization resistance.

VRC01 has been tested in several NHP challenge experiments (see Table 2-3). In a rectal challenge model with SHIV BaLP4, a dose of 20 mg/kg IV protected 6/6 NHP; a 5 mg/ kg IV dose protected 6/6; and a 0.3 mg/kg IV dose protected 2/6 [47]. Using a more resistant SHIV-162P3 challenge, a 20 mg/kg IV dose protected all 4 male animals from rectal challenge and all 4 female animals from vaginal challenge [47]. Analyses of the combined data from the NHP challenge studies show complete protection against SHIV162P3 challenge at a VRC01 plasma concentration of 50 mcg/ml and partial protection (IC50 [50% inhibitory concentration]) at 20 mcg/mL. For the more sensitive BaLP4 virus the IC50 is only 1.5 mcg/mL. Based on preclinical studies, an antibody serum concentration of about 40 to 50 mcg/mL is projected to provide protection against the vast majority of circulating strains of HIV [103]. In the NHP studies, both the virus sensitivity and serum antibody titers appear to influence protection from mucosal challenge. A summary of serum concentrations associated with protection against diverse SHIV strains of varying resistance to neutralization is shown in Figure 2-7.



Figure 2-7 VRC01 IC<sub>80</sub> values (170 Isolates) and serum concentrations in NHP SHIV challenge studies

It is particularly interesting to note that following administration of VRC01 to NHP, the antibody is found in mucosal tissues (see Figure 2-8). This is likely a product of active antibody transport to mucosal tissues through neonatal Fc receptor (FcRn) binding [48].



· Co-localization of VRC01 with FcRn

Active transport of IgG to mucosal surface

Figure 2-8 VRC01 mucosal pharmacokinetics in rhesus macaques [48]

NHP challenge studies have also shown that, in addition to classic neutralization, bnAbs such as VRC01 often elicit antibody-mediated cellular effector functions [45,104]. As a result, protection against experimental challenge has sometimes been achieved with notably low doses of VRC01 [47,103]. Similar mechanisms of protection have been implicated in studies of other bnAbs showing protection despite barely detectable neutralization activity (1:1) at challenge [44].

Recent NHP studies of VRC01 and other highly potent mAbs, such as PGT121, demonstrate protection at infusion doses of 5 mg/kg and even at 1 mg/kg [46,49,103,105]. There is also evidence that such protection can be durable; a simianized version of VRC01 was shown to protect monkeys against SHIV challenge nearly 8 weeks after their last 5 mg/kg antibody infusion, when plasma concentrations of VRC01 ranged from ~0.5 mcg/ml to undetectable [105]. These data suggest that a 10 mg/kg infusion dose of VRC01 administered every 8 weeks may offer protection against HIV acquisition.

Please see the VRC01 IB for more details on the NHP challenge studies.

## 2.9 Clinical trial experience

Completed phase 1 clinical studies of VRC01 include first-in-humans dose escalation studies for safety, tolerability, and PK assessments in HIV-infected (VRC 601) and HIV-uninfected (VRC 602) adults. Studies to characterize the neutralizing activity and other functional assays as a function of plasma concentration are also underway. As of April 2017, more than 1200 clinical trial participants have received VRC01 in phase 1 trials and in the phase 2b AMP studies.

Both the IV and SC routes of administration have been evaluated. Ultimately, the best route for clinical use may depend upon the age of the recipient (adult or infant), stage of product development, formulation, and important considerations related to volume needed and maintenance of a target VRC01 blood level considered to be in the therapeutic range.

#### 2.9.1 VRC 601

VRC 601 (NCT01950325) titled, "A Phase 1, Open-Label, Dose-Escalation Study of the Safety and Pharmacokinetics of a Human Monoclonal Antibody, VRC-HIVMAB060-00-AB (VRC01), with Broad HIV-1 Neutralizing Activity, Administered Intravenously or Subcutaneously to HIV-Infected Adults."

VRC 601 (Table 2-4) was the first study of the VRC01 mAb in HIV-infected participants [106]. It was a dose-escalation study to examine safety, tolerability, dose, PK, and anti-antibody immune responses. VRC 601 opened in September 2013 as a single site study at the NIH Clinical Center, Bethesda, Maryland and in total, 23 HIV-infected participants, including 15 aviremic ARV-treated participants and 8 viremic non-ARV treated participants, were infused with one or two doses of VRC01 at doses up to 40 mg/kg IV.

Table 2-4 VRC 601 study schema

| VRC 60 | 1 Dose Groups | VRC01 Administration Schedule | |
|---|---|---|---|
| Group | No. of<br>evaluable<br>participants* | Day 0 | Week 4 |
| 1 | 3-5 | 1 mg/kg IV | 1 mg/kg IV |
| 2 | 3-5 | 5 mg/kg IV | 5 mg/kg IV |
| 3 | 3-5 | 5 mg/kg SC | 5 mg/kg SC |
| 4 | 3-5 | 20 mg/kg IV | 20 mg/kg IV |
| 5 | 3-5 | 40 mg/kg IV | 40 mg/kg IV |
| Total | 15-25 | IV doses administered in 100 mL of minutes. SC doses administered in the minim *Only participants who begin infusi evaluable participants per group wil group until the safety review is com available, if needed, to have sufficie to include at least one eligible subje later after the dose escalation is com | num volume at 15 mL/hr. on are evaluable. Only 3 1 be enrolled into the dose pleted. Additional slots are ent data for the safety review or ct with a detectable viral load |

The first infusion at 1 mg/kg IV was administered in the VRC 601 study on September 30, 2013. Beginning on March 28, 2014, the dose escalation proceeded according to the schema. The first 40 mg/kg IV administration in this study occurred May 12, 2014 and the last infusion in VRC 601 occurred on April 6, 2015. All IV and/or SC infusions have been well-tolerated with no serious adverse events (SAEs) or dose limiting toxicity.

VRC 601 demonstrated evidence of VRC01-mediated antiviral effect. An interim analysis of the VRC 601 viral load data obtained from 8 viremic adults through April 30, 2015 shows that VRC01 has a statistically significant in vivo virological effect on HIV viral load when administered as a single 40 mg/kg IV dose. None of these adults were taking antiretroviral therapy (ART) when enrolled into the study and had not started ART during the time period when the viral load data were collected. Six of the eight adult participants had  $\geq 1 \log_{10}$  copies/mL decrease in viral load and two participants had a viral load drop of 0.26 and 0.18  $\log_{10}$  copies/mL respectively. These interim data indicate the following for a single dose of VRC01 at 40 mg/kg IV:

- A statistically significant change from baseline viral load postinfusion days 5 to 16;
- The median time to reach  $\geq 0.5 \log 10$  decrease in viral load is 5 days; and,
- The median time to greatest decrease in viral load is 7 days.

A 0.5 log<sub>10</sub> copies/mL or greater decrease in viral load is considered to be a positive response to ART. To have clinical benefit, such a change would need to be sustained. In VRC 601, participants were administered only one dose of

VRC01 at 40 mg/kg and, thus, a sustained effect on viral load was not expected. However, the data demonstrate a VRC01 mediated anti-viral effect.

#### 2.9.2 VRC 602

VRC 602 (NCT01993706) is titled, "A Phase 1 Dose-Escalation Study of the Safety and Pharmacokinetics of a Human Monoclonal Antibody, VRC-HIVMAB060-00-AB (VRC01), Administered Intravenously or Subcutaneously to Healthy Adults."

VRC 602 was the first study of the VRC01 mAb in HIV-uninfected adults. It was a dose-escalation study to examine safety, tolerability, dose, and PK of VRC01 [107]. VRC 602 opened in December 2013 as a single site study at the NIH Clinical Center, Bethesda, Maryland and the final infusion was administered in August 2014.

As shown in Table 2-5, there were 3 open-label, dose escalation groups (Groups 1, 2, and 3) for IV administration and 1 double-blinded, placebo-controlled group (Group 4) for SC administration.

Table 2-5 VRC 602 study schema

| | VRC 602 G | roups | VRC01 Admini | stration Schedule |
|---|---|---|---|---|
| Group | Initial<br>Enrollments | Additional<br>Enrollments | Day 0 | Week 4 |
| 1 | 3 | 2 | 5 mg/kg IV | 5 mg/kg IV |
| 2 | 3 | 2 | 20 mg/kg IV | 20 mg/kg IV |
| 3 | 3 | 2 | 40 mg/kg IV | 40 mg/kg IV |
| 4 | | SC admi | inistration | |
| 4A | 3 | 2 | 5 mg/kg SC | 5 mg/kg SC |
| 4B | 3 | 2 | Placebo SC | Placebo SC |
| | Total | 25 | 20 participants treat<br>different dosage lev<br>participants treated<br>administered SC | rels and 5 |

IV doses administered in 100 mL of normal saline over 1 hr.

First SC dose administered at about 15 mL/hr via SC infusion pump; subject option for second dose administration (Week 4) by direct SC injection with needle and syringe.

All IV and/or SC infusions were well-tolerated with no SAEs or dose limiting toxicity.

PK analysis from VRC 602 revealed a VRC01 terminal half-life of 15 days across all IV infused dose groups. After the first infusion, 28-day trough levels were 35 mcg/mL and 57 mcg/mL for the 20 mg/kg and 40 mg/kg dose groups, respectively. Following the second infusion, the 28-day trough values rose to 57 mcg/mL and 89 mcg/mL for the 20 mg/kg and 40 mg/kg dose groups, respectively [107].

In addition, after infusion VRC01 retained the expected neutralizing activity in serum and no anti-VRC01 antibodies were detected [107].

#### 2.9.3 HVTN 104

HVTN 104, titled *A phase 1 clinical trial to evaluate the safety and drug levels of a human monoclonal antibody, VRC-HIVMAB060-00-AB (VRC01) administered in multiple doses intravenously and subcutaneously in different dosing schedules to healthy, HIV-uninfected adults,* is examining safety profiles and serum levels of 5 different regimens for the IV and SC administration of VRC01 (Table 2-6). IV administration is being evaluated at doses of 10, 20, 30, and 40 mg/kg; SC administration is being tested at 5 mg/kg.

Table 2-6 HVTN 104 study schema

| Dose<br>Groups | | | | | Study p | roduct adn | ninistrati | on schedul | e in mon | ths (days) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Group | N | 0 | 0.5<br>(14) | 1 (28) | 1.5<br>(42) | 2 (56) | 2.5<br>(70) | 3 (84) | 3.5<br>(98) | 4 (112) | 4.5<br>(126) | 5 (140) | 5.5<br>(154) |
| 1 | 20 | VRC01<br>40mg/kg<br>IV | | VRC01<br>20mg/kg<br>IV | | VRC01<br>20mg/kg<br>IV | | VRC01<br>20mg/kg<br>IV | | VRC01<br>20mg/kg<br>IV | | VRC01<br>20mg/kg<br>IV | |
| 2 | 20 | VRC01<br>40mg/kg<br>IV | | | | VRC01<br>40mg/kg<br>IV | | | | VRC01<br>40mg/kg<br>IV | | | |
| | 20 | VRC01<br>40mg/kg<br>IV | VRC01<br>5mg/kg<br>SC | VRC01<br>5mg/kg<br>SC | VRC01<br>5mg/kg<br>SC | VRC01<br>5mg/kg<br>SC | VRC01<br>5mg/kg<br>SC | VRC01<br>5mg/kg<br>SC | VRC01<br>5mg/kg<br>SC | VRC01<br>5mg/kg<br>SC | VRC01<br>5mg/kg<br>SC | VRC01<br>5mg/kg<br>SC | VRC01<br>5mg/kg<br>SC |
| 3 | 4 | IV<br>placebo<br>for<br>VRC01 | SC<br>placebo<br>for<br>VRC01 | SC<br>placebo<br>for<br>VRC01 | SC<br>placebo<br>for<br>VRC01 | SC<br>placebo<br>for<br>VRC01 | SC<br>placebo<br>for<br>VRC01 | SC<br>placebo<br>for<br>VRC01 | SC<br>placebo<br>for<br>VRC01 | SC<br>placebo<br>for<br>VRC01 | SC<br>placebo<br>for<br>VRC01 | SC<br>placebo<br>for<br>VRC01 | SC<br>placebo<br>for<br>VRC01 |
| 4 | 12 | VRC01<br>10mg/kg<br>IV | | | | VRC01<br>10mg/kg<br>IV | | | | VRC01<br>10mg/kg<br>IV | | | |
| 5 | 12 | VRC01<br>30mg/kg<br>IV | | | | VRC01<br>30mg/kg<br>IV | | | | VRC01<br>30mg/kg<br>IV | | | |
| Total | 88 | | . , | ses admini<br>doses adm | | | | | hr | | | | |

HVTN 104 is a phase 1 clinical trial designed to evaluate the safety and drug levels of VRC01 administered in multiple intravenous or subcutaneous doses and different dosing schedules to 88 healthy, HIV-uninfected adults at 6 HVTN CRSs in 4 US cities: Boston, New York, Philadelphia, and Cleveland. The first participant enrolled in HVTN 104 on September 9, 2014 and the last participant enrolled on July 15, 2015. Study product administration for all participants was complete as of November 30, 2015. The study has 5 arms: Group 1 is evaluating the IV administration of a 40 mg/kg loading dose, with 2 subsequent 20 mg/kg doses given at 8 week intervals. Groups 2, 4, and 5 are evaluating 3 infusions of 40 mg/kg, 10 mg/kg, or 30 mg/kg, respectively, given 8 weeks apart. Group 3 is evaluating 5 mg/kg given every 2 weeks subcutaneously for 24 weeks after an initial IV administration at 40 mg/kg; this will inform the design of perinatal

prophylaxis studies. Secondary aims of HVTN 104 are: (1) to evaluate the kinetics of *in vitro* neutralization in serum of a single VRC01 sensitive virus isolate (TZM.bl assay); (2) to determine whether anti-idiotypic antibody (AIA) can be detected and whether there is a correlation of VRC01 levels and AIA levels in serum; (3) to determine if measurable levels of VRC01 can be found in genital, rectal, and oral secretions; (4) to evaluate the kinetics of *in vitro* neutralization in mucosal secretions of a single VRC01 sensitive virus isolate; and (5) to assess binding of VRC01 to multiple Env proteins.

A total of 249 IV infusions and 208 SC injections of VRC01 were administered in HVTN 104. The infusions and injections were well tolerated, with 28% of infusions and 14% of injections associated with mild pain and/or tenderness. 55% of VRC01 and 50% of placebo recipients experienced mild pain and/or tenderness at the infusion or injection site sometime during the trial. One participant experienced moderate pain and/or tenderness following a SC injection of VRC01. Mild infusion site erythema/induration reactions were reported for 2 VRC01 participants and 1 placebo recipient. Two moderate erythema/induration reactions were reported. 1 following IV VRC01 and 1 following VRC01 SC injection. For 76% of the infusions and injections administered in the trial, no systemic reactogenicity symptoms were reported. 56% of VRC01 and 75% of placebo recipients experienced systemic reactogenicity symptoms following at least one study product administration. These were all graded as mild in the placebo recipients; of VRC01 recipients who experienced any systemic symptoms, the maximum severeity was mild in 70%, moderate in 23%, and severe in 6% (3 participants). The most commonly reported symptoms were malaise/fatigue, headaches, and myalgias.

The severe systemic reactogenicity symptoms reported in 3 VRC01 recipients are detailed as follows:

- 1 participant developed severe malaise, myalgia, headache and chills, mild nausea, and moderate arthralgia symptoms within 3 days after the first infusion of study product. These symtoms had resolved by Day 7. The participant had a concomitant AE of laboratory confirmed Influenza A infection diagnosed on Day 2 and was treated with Ibuprofen.
- 1 participant reported a viral illness AE of moderate intensity beginning 3 days prior to the 9<sup>th</sup> SC injection (10th study product administration), characterized by nausea and vomiting, sore throat, runny nose but no fevers; a household contact was also ill. At baseline on Day 0 of the 9<sup>th</sup> SC injection, mild malaise/fatigue was still present. At the early assessment timepoint on Day 0, this was still present and also grade 1 nausea. Within 3 days of the injection, the participant developed severe malaise, myalgia, headache, chills, and arthralgia; these all resolved on Day 6, which was the date the AE for viral illness was resolved. There was no reported use of concomitant medications for these symptoms.
• 1 participant reported severe malaise/fatigue on the day of the first infusion, resolving spontaneously the next day. During this reactogenicity period, this participant also reported a grade 1 headache on Day 1, resolving the next day.

There were no study product discontinuations due to reactogenicity symptoms.

There were 235 AEs occurring in 70 participants (79.5%), with similar rates of occurrence across all treatment groups. 74% of AEs were graded as mild, 22.5% as moderate, and 3.4% as severe. 9 AEs (3.8% of all AEs) occurring in 8 participants were deemed product-related by the investigators; all were mild and transient. Those occurring following VRC01 administration included elevations of hepatic transaminases (AST and ALT in 1 individual), elevated creatinine, neutropenia, localized injection site pruritus, diarrhea, generalized rash, and Varicella zoster infection. No VRC01-related hypersensitivity reactions or CRS symptoms were observed during the study.

Study product administration was discontinued in 8 participants. Reasons for discontinuing study product included: AEs (3 participants), relocation from study site (2), unable to adhere to visit schedule (1), unable to contact (1), and pregnancy (1). Of those participants for whom study product was discontinued due to an AE, 1 participant developed a mild, localized pruritic, maculopapular rash 3 days after receiving the first SC injection of VRC01, which resolved within 4 hours after applying inert lotion; this was deemed related to study product. Another participant had a brief syncopal episode several hours after receiving a VRC01 infusion; this was deemed not related to study product. A third participant had mild, brief chest tightness following the first SC injection that resolved spontaneously; this was deemed related to study product, however this participant was determined after unblinding to have received the placebo. In sum, VRC01 was well-tolerated when administered IV or SC.

Of note, safety experience with VRC01 has remained consistent whether 1-2 doses were administered, as in VRC 601 and 602, or multiple doses were administered, as in HVTN 104. No trends toward recurrence of lab abnormalities or AEs deemed related to study product or increase in frequency or severity of local or systemic reactogenicity symptoms has been observed with multiple administrations of VRC01.

Figure 2-9 shows serum VRC01 levels following the first 2 infusions (samples collected as of October 19, 2015) for participants in Group 4 (10 mg/kg of VRC01) and Group 5 (30 mg/kg) of HVTN 104. The number of study participants with samples assayed at each time point is shown on the X axis of each graph. As expected, trough levels following the second infusion are somewhat higher than following the first infusion. The median antibody concentration in the 10 mg/kg group is above 10 mcg/mL for approximately 37 of the 56 days (66%) following the second infusion with a median trough concentration of 4.6 mcg/mL (25-75% interquartile range 2.6-6.3). For the 30mg/kg group the median trough level is 9 mcg/mL (25-75% interquartile range 6.5-9.4).

These levels are quite similar to those modeled for the study and they show the desired overlap in concentrations achieved with the two doses selected for the study.





Figure 2-9 VRC01 serum levels through month 4 observed in HVTN 104 Group 4 (10mg/kg IV) and Group 5 (30mg/kg IV)

# 2.9.4 Safety summary of VRC01

As of February 23. 2016, approximately 130 adult participants received one or more VRC01 administrations, including 23 in VRC 601, 23 in VRC 602 (5 additional participants received placebo), and 84 in HVTN 104 (4 additional participants received placebo). 249 VRC01 infusions and 208 SC injections were given in HVTN 104.

Cumulatively, there have been no expedited safety reports to the FDA or study safety pauses for adverse events and no reactions during the VRC01 or

placebo/control product administration that resulted in an incomplete administration.

VRC01 SC or IV administrations are generally associated with mild or moderate local reactions of pruritus, redness, and pain/tenderness, which resolve within a few minutes to a few hours after the administration is completed. When present, most systemic reactions after administration of VRC01 SC or IV are mild and include: malaise, myalgia, headache, chills, nausea, and joint pain.

Unsolicited AEs of grade 3 or higher severity and deemed related to study product have not been reported.

Other AEs attributed to study product administration have included mild or moderate AST elevation, alanine aminotransferase (ALT) elevation, creatinine elevation, and decreased neutrophil count. Mild or moderate elevated transaminases were reported in 4 of 21 (19%) HIV-infected participants in VRC 601 (all of whom were taking ARVs). These laboratory changes resolved spontaneously and did not require discontinuation of study product administration. Among HIV-uninfected participants in VRC 602 or HVTN 104, 1 participant had grade 1 (mild) transiently elevated ALT assessed as possibly attributed to VRC01 in the VRC 602 study and 2 participants had grade 1 (mild) transiently elevated ALT/AST values assessed as related to VRC01 in HVTN 104. These 3 participants all received VRC01.

In the HVTN 104 trial, there were 3 product discontinuations for AEs, 2 of which were deemed related to study product infusion or injection. One discontinuation was for a 20-minute episode of chest tightness occurring approximately 25 minutes after SC injection of placebo in a participant who is a chronic smoker on nicotine replacement while smoking. One discontinuation was in a participant who reported a generalized rash that began three days after SC injection of VRC01, and resolved within 4 hours with ibuprofen and the application of an over-the-counter non-steroidal cream. The third discontinuation was in a young, otherwise healthy participant who experienced a brief episode of syncope, deemed not related to study product, approximately 4 hours after IV infusion of VRC01. In addition, one person in HVTN 104 had study product discontinued due to pregnancy occurring during the trial.

Overall, VRC01 administration in the dose range from 10 to 40 mg/kg IV and at 5 mg/kg SC has been assessed as well-tolerated and safe for further evaluation.

#### 2.9.5 Particle formation

VRC01 is a highly concentrated protein solution and may develop white, opaque to translucent particles after thawing. When particles are observed, they may disappear after a few hours at room temperature or storage at 2°C to 8°C. For additional information, see the IB.

# 2.10 Potential risks of study products and administration

In a preclinical study performed in rats, there was a small dose-dependent, but transient, increase in AST and ALP, but not in ALT following IV administration. In rats, there were no histopathology findings following IV administration.

Thus far in VRC 601, VRC 602, and HVTN 104 there have been no SAEs deemed related to study product (see Section 2.9.4). Administration of mAb may have a risk of immune reactions such as acute anaphylaxis, serum sickness, and the generation of auto-reactive antibodies; however, these reactions are rare and more often associated with mAbs targeted to human proteins or with the use of murine mAbs, which would have a risk of human anti-mouse antibodies [106]. In this regard, as VRC01 is targeted to a viral antigen and is a human mAb, it is expected to have a low risk of such side effects.

Typically, the side effects of mAbs are mild but may include fever, flushing, chills, rigors, nausea, vomiting, pain, headache, dizziness, shortness of breath, bronchospasm, hypotension, hypertension, pruritus, rash, urticaria, angioedema, diarrhea, tachycardia, or chest pain. Clinical use of mAbs that are targeted to cytokines or antigens associated with human cells may be associated with an increased risk of infections [108]; however, this is not expected to be a risk for a mAb targeted to a viral antigen.

It is known from published experience with human mAbs directed against the cell surface targets on lymphocytes that infusion of a mAb may be associated with cytokine release, causing a reaction known as cytokine release syndrome [109]. Cytokine release syndrome and other immune reactions such as tumor lysis syndrome have been observed with administration of chimeric and humanized mAb [108]. Most infusion-related events occur within the first 24 hours after beginning administration. Specifically, with regard to cytokine release syndrome reactions, these most commonly occur within the first few hours of beginning the infusion and are more common with the first mAb infusion received. This is because the cytokine release is associated with lysis of the cells targeted by the mAb and the burden of target cells is greatest at the time of the first mAb treatment. With licensed therapeutic mAbs, cytokine release syndrome is managed by temporarily stopping the infusion, administering histamine blockers, and restarting the infusion at a slower rate [110]. Severe reactions such as anaphylaxis, angioedema, bronchospasm, hypotension, and hypoxia are infrequent and more often associated with mAbs targeted to human proteins or with a non-human mAb, such as a murine mAb [108].

Delayed allergic reactions to a mAb may include a serum sickness type of reaction, which is characterized by urticaria, fever, lymph node enlargement, and joint pains. These symptoms may not appear until several days after exposure to the mAb and are noted to be more common with chimeric types of mAb [108]. Serum sickness has not been described with administration of licensed fully human mAbs.

There are several FDA-licensed mAbs for which reactions related to the rate of infusion have been described. Some symptoms may be treated by slowing or stopping the infusion.

Other side effects of licensed mAbs include infections, thrombocytopenia, autoimmune diseases, cancer, dermatitis, and cardiotoxicity [108].

The HVTN laboratory tested plasma from HIV-uninfected individuals that was spiked with VRC01 in a range of concentrations that encompasses those likely to be observed in this clinical trial. VRC01 did not cause a reactive test result using several standard antibody-based HIV-1/2 diagnostic tests used in the US. However, VRC01 is an antibody to an HIV protein, so, it may be theoretically possible for a standard antibody-based HIV diagnostic test to detect VRC01 for a short time period postinfusion or postinjection. This has not been observed in clinical studies to date.

Risks of Blood Drawing: Blood drawing may cause pain and bruising and may, infrequently, cause a feeling of lightheadedness or fainting. Rarely, it may cause infection at the site where the blood is taken. Problems from use of an IV for blood drawing are generally mild and may include pain, bruising, minor swelling, or bleeding at the IV site and, rarely, infection, vein inflammation (phlebitis), or blood clot.

Risks of IV Infusion: The placement of an IV catheter can allow for the development of bacteremia because of the contact between the catheter and unsterile skin during insertion. Risk of infection from IV infusion will be minimized through careful decontamination of skin prior to catheter placement and through the use of infection control practices during infusion. The risk of product contamination will be minimized through the use of aseptic techniques during product preparation and administration.

# 3 Objectives and endpoints

# 3.1 Primary objectives and endpoints

*Primary objective 1:* 

To evaluate the safety and tolerability of VRC01 mAb administered through IV infusion in sub-Saharan African women

Primary endpoint 1:

Local and systemic reactogenicity signs and symptoms, laboratory measures of safety, AEs, SAEs, and rates of discontinuation

Primary objective 2:

To determine if the VRC01 mAb prevents HIV-1 infection and to estimate the level of efficacy in sub-Saharan African women

Primary endpoint 2:

Documented HIV-1 infection by the Week 80 study visit

## 3.2 Secondary objectives and endpoints

Secondary objective 1:

To develop a marker(s) of the VRC01 mAb that correlates with the level and antigenic specificity of protection against HIV-1 infection and to provide insight into the mechanistic correlates of protection

Secondary endpoints 1:

Serum concentration of VRC01 in participants assigned to receive the mAb (ELISA, neutralizing assay)

Serum mAb effector functions to HIV-1 Envs representing variability of the VRC01 antibody footprint

Sequences of breakthrough HIV infections from the earliest available HIV-positive plasma samples

VRC01 neutralization-sensitivity of, and effector function against, HIV strains from infected trial participants from the earliest available post–HIV-infection serum samples

# 3.3 Exploratory objectives

Exploratory objective 1:

To assess use of FTC/TDF in the study cohort

Exploratory objective 2:

To assess if prevention efficacy is modified by FTC/TDF use

Exploratory objective 3:

To understand changes in risk behavior and the potential for risk compensation for all study participants

Exploratory objective 4:

To measure anti-idiotype antibodies to VRC01

# 4 Statistical considerations

#### 4.1 Outline of the statistical considerations section

The statistical considerations section is organized as follows. Section 4.2 states the primary and secondary efficacy objectives in terms of the target prevention efficacy (PE) parameters that are estimated in the trial, and describes the hypothesis tests regarding these efficacy parameters. Section 4.3 summarizes a statistical rationale for using a 3-arm design, which adds to the scientific rationale provided in Section 2.4. Section 4.4 describes sample size and power considerations for the primary efficacy objectives, which justify the sample size of the trial. Section 4.4 also provides operating characteristics of the trial design for addressing the primary efficacy objective. Section 4.5 describes statistical power available for the secondary objective that compares PE between the two mAb dose groups. Section 4.6 describes statistical power available for detecting safety problems of the mAb in terms of SAEs. Section 4.7 summarizes the approach to monitoring the trial including interim analysis reports provided to the DSMB. Sections 4.8, 4.9, and 4.10 describe ARV assessments, randomization, and blinding, respectively. Section 4.11 describes the approach to statistical analysis, ordered first by the approach to the analysis of PE, and secondly by the approach to the assessment of correlates of protection.

# 4.2 PE parameters for measuring mAb efficacy and associated primary and secondary hypothesis tests

Let PE denote the overall PE of the 10 mg/kg and 30 mg/kg mAb groups pooled together compared to the control group. This PE parameter is defined as

PE =  $[1 - \text{Cumul. incid. ratio (pooled mAb grp/control) of HIV-1 Dx by 80 Wks}] \times 100\%$ ,

where the cumulative incidence ratio is the probability of HIV-1 diagnosis by the Week 80 visit for participants assigned to receive the mAb divided by the probability of HIV-1 diagnosis by the Week 80 visit for participants assigned to receive control. PE is the target parameter for the primary analysis of overall PE.

The primary analysis tests the null hypothesis

H0: PE = 0% versus the alternative hypothesis H1: PE  $\neq 0\%$ 

using a 2-sided alpha = 0.05 level test that accounts for sequential monitoring for potential harm, non-efficacy, and high efficacy.

Secondary analyses assess PE parameters for the mAb dose groups separately. Let PE10 be the overall PE of the 10 mg/kg mAb group and let PE30 be the overall PE of the 30 mg/kg mAb group, defined as

PE10 =  $[1 - \text{Cumul. incid. ratio (mAb-10 mg/kg grp/control) of HIV-1 Dx by 80 Wks}] \times 100\%$ 

and

PE30 =  $[1 - \text{Cumul. incid. ratio (mAb-30 mg/kg grp/control) of HIV-1 Dx by 80 Wks}] \times 100\%$ .

Secondary analyses test the null hypotheses

```
H0: PE10 = 0% versus the alternative hypothesis H1: PE10 \neq 0% and
```

H0: PE30 = 0% versus the alternative hypothesis H1: PE30  $\neq$  0%

using 2-sided alpha = 0.05 level tests. Both unadjusted p-values and Holm-Bonferroni p-values will be reported for each of the individual dose versus placebo group analyses.

In addition, the following secondary analyses of PE are conducted:

• Assess a dose-response effect by testing the null hypothesis

H0: Cumul. HIV-1 incidence by 80 Wks equal in the 3 groups versus H1:  $0\% \le PE10 \le PE30$  with at least one strict inequality

- Test the complete null hypothesis that the HIV-1 incidence is the same in the three treatment groups versus the alternative hypothesis that there are some differences
- Test for different HIV-1 incidence between the two mAb groups, where a finding of PE30 significantly greater than PE10 would demonstrate that assignment to a higher mAb dose level causes higher PE

## 4.3 Statistical rationale for the 3-arm design compared to a 2-arm design

An alternative design would compare a single dose and schedule of the VRC01 mAb versus control. However, the 3-arm design allows addressing additional scientific questions and improves the assessment of correlates of protection, without requiring more participants by virtue of the primary analysis being based on the pooled mAb groups versus control. Specifically, consider a 2-arm design with 2:1 allocation to a single dose of VRC01 versus placebo, compared to the 3-arm design in the protocol with 1:1:1 allocation. For scenarios where the average of PE10 and PE30 equal PE set to a number greater than 0 and less than 1, power to reject H0: PE  $\leq$  0% in favor of H1: PE > 0% is very similar between the two trial designs, for the same total number of study participants. By providing results

about estimated PE10 and estimated PE30 as well as about pooled estimated PE, the trial provides data for modeling of how PE would change given a new dose and/or schedule.

A second advantage of the 3-arm design is that it allows a direct assessment of the causal effect of different mAb infusion doses on HIV-1 incidence based on randomization of treatment assignments (a so-called 'group-level' correlate of protection), which can directly prove the concept that a higher mAb dose causes a greater level of protection. In contrast, with a 2-arm design the association between mAb marker characteristics and the level of PE can only be inferred with non-randomized epidemiological analysis approaches for which the results cannot be guaranteed to be free from postrandomization selection bias [111,112]. That is, without a randomization to multiple mAb interventions a result that a mAb characteristic is associated with reduced incidence of HIV-1 infection may not imply that mAb recipients with the characteristic have a higher level of PE. For instance, the implication may fail if participants tend to have fewer HIV-1 exposures during the few weeks after infusion visits compared to during the few weeks before infusion visits, which could possibly occur related to the counseling and informed consent process. Or, the implication may fail if the mAb characteristic marks an intrinsic HIV-1 susceptibility factor that is not caused by administration of the mAb [113-115]. A third advantage of the 3-arm design is that the random assignment of two mAb doses creates greater inter-individual variability in mAb characteristics, which improves statistical power for the assessment of individual-level correlates of protection.

In sum, the dose-response 3-arm design has the advantages of allowing more insightful and rigorous inferences about causal effects of the mAb and greater resolution of correlates of protection, and allows addressing the additional question of whether a higher dose confers greater PE than a lower dose.

# 4.4 Sample size calculations for testing for overall PE (Primary objective 2)

The trial is designed to have 90% power to test

H0: PE  $\leq$  0% versus the alternative hypothesis H1: PE > 0%

if the level of overall pooled PE is 60% (with a 1-sided 0.025  $\alpha$ -level test); the design fits the paradigm of an intermediate-sized phase 2b screening efficacy trial proposed for HIV-1 vaccine efficacy trials by Rida, Fleming et al [116].

The sample size calculations are based on the power of a 1-sided 0.025-level Wald test for comparing log-transformed cumulative incidences of HIV-1 infection by the Week 80 visit between randomized groups, in the presence of the sequential monitoring described below. Power is computed based on simulating 10,000 efficacy trials under assumptions described below using the R package seqDesign.

# 4.4.1 Assumptions of the sample size calculations including sequential monitoring for PE

The following assumptions are made for the sample size calculations:

- 10% annual dropout incidence in each of the three study groups
- 27 month uniform accrual with halved accrual during the first three months (approximating current accrual projections)
- visits every 4 weeks for HIV-1 diagnostic tests through Week 80 and HIV-1 status at Week 80 is known
- 4.0% annual HIV-1 incidence in the control group
- For each of the mAb treatment groups, average PE versus control within an 8-week infusion interval is assumed to be the same for each of the 10 infusion intervals
- Sequential monitoring of the mAb groups versus control to stop early for:
  - Potential harm [Establish that PE (pooled over the mAb groups) < 0% based on a 2-sided monitoring adjusted 90% CI lying below 0%]</li>
  - o Non-efficacy [Establish that PE (pooled over the mAb groups) ≤ 40% based on a 2-sided 95% nominal CI lying below 40%]
  - High efficacy [Establish that PE (pooled over the mAb groups) > 70% based on a 2-sided 95% nominal CI lying above 70%]

With the exception of the potential harm monitoring, the sequential monitoring of PE does not use critical values adjusted for the number of analyses. Examination of the design operating characteristics (reported in the figures and tables below) was used to ensure that this approach provides a fitting trade-off of the control of false negative and false positive error rates.

Justification for the incidence assumptions is provided in Section 4.4.6.

We also show power calculations allowing for lower levels of HIV-1 incidence. In particular, we show power calculations assuming 3.3% annual HIV-1 incidence in the control group, which would account for lower than expected incidence rates due to increased PrEP usage.

# 4.4.2 Power curves and operating characteristics of the design (Primary objective 2)

Required sample sizes to achieve 90% power to reject H0: PE  $\leq$  0% in favor of H1: PE > 0% for different values of PE are determined based on 1-sided 0.025 level Wald tests as described above. The power calculations are repeated for a

range of sample sizes to determine the required sample size to achieve 90% power as reported in Figure 4-1. These power calculations are conducted using the open source R package seqDesign developed by the protocol statisticians [117], which computes power based on simulating many thousands of efficacy trials, applying the sequential monitoring procedures to each trial, and computing power as the fraction of the trials where the 1-sided 0.025-level Wald test rejects the null hypothesis. The calculations are based on a large number of simulated efficacy trials.

Figure 4-1 shows the total sample size required to have 90% power to reject H0:  $PE \le 0\%$  in favor of H1: PE > 0% for different values of PE = PE10 = PE30. The results show that about N = 1800 total participants are needed to achieve 90% power to detect PE = 60%; the sample size N = 1900 total participants (~634 per arm) is selected to build in a provision of robustness to the control group annual incidence being lower than 4.0%.



Figure 4-1 Total sample size for 90% power to reject H0: PE ≤ 0% in favor of H1: PE > 0% in a 1:1:1 allocation design with 80 weeks of follow-up for HIV-1 infection for each trial participant

Table 4-1 shows power available to reject the null hypothesis under different levels of true PE.

Table 4-1 Power for rejecting H0: PE ≤ 0% in favor of H1: PE > 0% under different effect sizes PE = PE10 = PE30

| | Unconditional Power (× 100) |
|-----|-----------------------------|
| 0% | 2.7 |
| 10% | 7.4 |
| 20% | 18.7 |
| 30% | 37.0 |
| 40% | 60.5 |
| 50% | 82.1 |
| 60% | 95.1 |
| 70% | 99.4 |
| 80% | >99.9 |
| 90% | >99.9 |
| 95% | >99.9 |

The power calculations for the primary analysis of prevention efficacy were done assuming PE10 = PE30, and it is of importance to also understand power available in the primary analysis in the event that PE10 differs from PE30. Power for rejecting H0:  $PE \le 0\%$  in favor of H1: PE > 0% when PE equals a fixed constant PE<sub>0</sub> greater than 0 and less than 1 is very similar for different values of (PE10, PE30) subject to the constraint of average value (PE10 + PE30)/2 = PE<sub>0</sub>. For example, power to test H0 vs. H1 is very similar for (PE10, PE30) = (60%, 60%) and for (PE10, PE30) = (30%, 90%). This result attains because all of these scenarios have the same number of expected HIV-1 infection events among study participants assigned to receive VRC01. Power tends to be slightly greater for differential scenarios like (PE10, PE30) = (30%, 90%) compared to the equal scenario (PE10, PE30) = (60%, 60%), because the hypothesis testing procedure stratifies by VRC01 dose group, gaining efficiency by accounting for a baseline variable that predicts HIV infection. Therefore, the trial is powered to detect the design alternative of a dose-pooled VRC01 efficacy PE equal to 60%, regardless of whether VRC01 efficacy differs by dose group.

# 4.4.3 Additional operating characteristics of the design for assessing primary objective 2

For the selected sample size (N = 1900), Figure 4-2 shows the power curves for rejecting H0:  $PE \le 0\%$  in favor of H0: PE > 0% for a range of fixed values of the pooled PE. The power for rejecting H0 when the HIV-1 incidence rate is lower than projected is included in the figure. At the lower incidence of 3.3%, there is 90.5% power to detect PE = 60%. Section 4.4.6 describes the rationale for the incidence assumptions in this trial.



Figure 4-2 Unconditional power to reject H0: PE  $\leq$  0% in favor of H1: PE > 0% for a range of fixed values of pooled PE based on primary assumptions for HIV-1 incidence and dropout rate. A power curve is also shown for a lower than expected HIV-1 incidence rate.

# 4.4.4 Additional operating characteristics of the primary analysis accounting for the sequential monitoring

For the selected sample size (N = 1900), Figure 4-3 shows probabilities of reaching each possible trial monitoring outcome, pooling over the two mAb treatments (under the primary assumptions about HIV-1 incidence and dropout rates). More specifically, the monitoring outcomes include potential harm, non-efficacy, and high efficacy. Table 4-2 provides the same information in tabular form. In addition, the figure and table show unconditional power in the primary

analysis to reject the null hypothesis H0:  $PE \le 0\%$  in favor of the alternative hypothesis H1: PE > 0%.



Figure 4-3 Probabilities of reaching each possible trial monitoring outcome, and unconditional power to reject the primary null hypothesis H0: PE ≤ 0% with 634 control recipients and 1268 mAb recipients (1-sided 0.025-level tests)

Table 4-2 Probabilities (x 100) of reaching each possible trial monitoring outcome, and unconditional power (x 100) to reject the null hypothesis H0:  $PE \le 0\%$  in favor of the alternative hypothesis H1: PE > 0%, pooling over the two mAb groups (1-sided 0.025-level tests)

| | | Weed Out at Interim Analysis | | | |
|---|---|---|---|---|---|
| | | Potential Harm | Non-Efficacy | High Efficacy | <b>Unconditional Power</b> |
| PE | HR | PE < 0% | PE < 40% | PE > 70% | PE > 0% |
| | 3.0 | 95.5 | 4.5 | 0.0 | 0.0 |
| | 2.5 | 87.7 | 12.3 | 0.0 | 0.0 |
| | 2.0 | 67.7 | 32.3 | 0.0 | 0.0 |
| | 1.5 | 34.3 | 65.7 | 0.0 | 0.0 |
| 0% | 1.0 | 5.1 | 92.2 | 0.0 | 2.7 |
| 10% | 0.9 | 2.4 | 90.3 | 0.0 | 7.4 |
| 20% | 8.0 | 1.0 | 80.3 | 0.0 | 18.7 |
| 30% | 0.7 | 0.3 | 62.6 | 0.0 | 37.0 |
| 40% | 0.6 | 0.1 | 39.4 | 0.0 | 60.5 |
| 50% | 0.5 | 0.0 | 17.9 | 0.0 | 82.1 |
| 60% | 0.4 | 0.0 | 4.9 | 0.0 | 95.1 |
| 70% | 0.3 | 0.0 | 0.6 | 2.1 | 99.4 |
| 80% | 0.2 | 0.0 | 0.0 | 21.4 | >99.9 |
| 90% | 0.1 | 0.0 | 0.0 | 82.6 | >99.9 |
| 95% | 0.0 | 0.0 | 0.0 | 98.6 | >99.9 |

N = 634:1268 Control:mAb group

4.0% annual incidence in the Control group

10% annual dropout

Cumulative incidence-based non-efficacy monitoring

Cumulative incidence-based high-efficacy monitoring

Cumulative incidence-based unconditional power

Table 4-3 shows the numbers of HIV-1 infection endpoints during the trial expected under the null hypothesis scenario PE = PE10 = PE30 = 0% and under the design alternative hypothesis scenario PE = PE10 = PE30 = 60%. Under the design alternative hypothesis scenario, the calculations show that 35 HIV-1 infection endpoints are expected in the control group and 28 HIV-1 infection endpoints are expected in the two mAb groups combined after 80 weeks of follow-up.

Table 4-3 Cumulative number of HIV-1 infection endpoints over 80 weeks of follow-up under the null hypothesis scenario PE10 = PE30 = 0% and under the design alternative hypothesis scenario PE = PE10 = PE30 = 60%. Medians are computed based on simulating a large number of efficacy trials.

| PE10 = PE30 | Weeks since first person in | Median number of control endpoints | Median number of pooled mAb group endpoints |
|---|---|---|---|
| 0% | 0 | 0 | 0 |
| 0% | 26 | 1 | 1 |
| 0% | 52 | 4 | 8 |
| 0% | 78 | 10 | 20 |
| 0% | 104 | 18 | 35 |
| 0% | 130 | 23 | 47 |
| 0% | 156 | 26 | 51 |
| 0% | 182 | 26 | 53 |
| 0% | 197 | 26 | 54 |
| 60% | 0 | 0 | 0 |
| 60% | 26 | 1 | 0 |
| 60% | 52 | 4 | 3 |
| 60% | 78 | 10 | 8 |
| 60% | 104 | 18 | 14 |
| 60% | 130 | 26 | 21 |
| 60% | 156 | 31 | 25 |
| 60% | 182 | 34 | 28 |
| 60% | 197 | 35 | 28 |

# 4.4.5 Power curves for secondary hypothesis tests about PE in each mAb group

Figure 4-4 shows unconditional power to reject the null hypothesis H0:  $PE10 \le 0\%$  versus the alternative hypothesis H1: PE10 > 0% (or, equivalently, the null hypothesis H0:  $PE30 \le 0\%$  versus the alternative hypothesis H1: PE30 > 0%), where PE10 and PE30 measure prevention efficacy in each mAb group separately.



Figure 4-4 Unconditional power to reject H0: PE10  $\leq$  0% in favor of H1: PE10 > 0% (or H0: PE30  $\leq$  0% in favor of H1: PE30 > 0%) based on primary assumptions about HIV-1 incidence rate and dropout rate. A power curve is also shown for a lower than expected HIV-1 incidence rate.

### 4.4.6 Rationale for the HIV-1 incidence assumptions

The assumption of 4.0% annual HIV-1 incidence for the control group is based on recent data directly measuring HIV-1 incidence in women at several African sites [6,61,64-67,81,82,118]. The overall annual incidence rate in the VOICE study was 5.7%, which pools over all intervention groups given the similar incidence rates and the lack of significant differences. The annual incidence rate of female control recipients in the Phambili study, at 5.1%. The Fem-Prep and ASPIRE studies had annual incidence rates of 5.0% and 4.5%, respectively, in the control groups. The FACTS-001 trial showed no efficacy and the annual incidence was 4.0% for both study arms.

The total sample size N=1900 builds in a conservative margin, where the smallest control group annual incidence under which there is at least 90% power to detect PE = 60% is 3.3%. Moreover, power is 81.9% to detect PE = 60% if the control group annual incidence is 2.56%. This scenario of 2.56% annual incidence is consistent with the following scenario in which many study participants choose to use Truvada PrEP: 60% of person-years at-risk are without PrEP use and a 4.0% control group annual incidence, and the other 40% of person-years at-risk are with PrEP use at 90% PrEP efficacy and thus a 0.4% control group annual incidence. In this scenario, an assumption of 75% (instead of 90%) PrEP efficacy yields the control-group annual incidence of 2.8% (instead of 2.56%).

Based on a synthesis of the above-cited references using control arms or active arms in trials that showed no efficacy, we assume that the background annual incidence of HIV-1 in sub-Saharan African women in the absence of any PrEP

use is 5.1%. It is difficult to predict the degree of PrEP use that will occur in sub-Saharan African women. Given that the South African Medicines Control Council (MCC) approved fixed-dose emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) for use as PrEP only recently (December 2015) and the drug is not yet available in the public sector on which the vast majority of South Africans depend for health care and pharmaceuticals. While the government of South Africa is committed to rolling PrEP out as part of its HIV prevention efforts and is currently undertaking a limited number of narrowly targeted demonstration projects, when PrEP will be available more broadly in South Africa is unclear. The situation is equally uncertain in the other sub-Saharan countries in which this trial will be conducted. Assuming 15% of the PYRs under PrEP use with 90% (75%) PrEP efficacy leads to 4.4% (4.5%) control-group annual incidence. This protocol assumes conservatively 4.0% annual incidence in the control group.

Higher than expected use of PrEP will be reflected in lower than expected annual incidence rates. As shown in Figure 4-2, however, the trial would still provide enough statistical information to be powered to detect highly relevant prevention efficacy effect sizes if annual incidence rates are lower than we have estimated here due to higher than expected use of PrEP.

# 4.5 Power for the secondary analysis comparing HIV-1 incidence between the 10 mg/kg mAb group versus the 30 mg/kg mAb group

Table 4-4 reports power calculations for comparing HIV-1 incidence between the 10 mg/kg and 30 mg/kg mAb groups. The calculations assume the scenarios for true values of PE10 and PE30 indicated in the first two columns of the table. The results show that the study is moderately powered to detect large differences (eg, 65.6% power to discriminate 30% vs 70% PE) but may miss moderate differences (eg, 37% power to discriminate 30% vs 60% PE). In contrast, the study has high power to correctly select the best mAb dose group given moderate efficacy differences. Specifically, if the true PE30 is moderately greater than the true PE10, then there is high probability that the estimated PE30 would be greater than the estimated PE10, such that the 30 mg/kg mAb dose group would be selected.

Table 4-4 Statistical power for comparing the 10 versus 30 mg/kg mAb groups: Power to select the best mAb group and power to correctly select the best mAb group

| | | Power to Select Best mAb | Power to Detect PE10 |
|------|------|--------------------------|----------------------|
| PE10 | PE30 | Dose Group <sup>\$</sup> | Different from PE30# |
| 20% | 60% | 84.1 | 55.2 |
| 30% | 60% | 82.4 | 37.7 |
| 40% | 60% | 77.7 | 19.0 |
| 30% | 70% | 96.0 | 65.6 |
| 50% | 85% | 99.0 | 72.5 |

<sup>§</sup> Probability that the mAb dose group that is truly better (the 30 mg/kg dose group in the scenarios considered in the table) is correctly selected based on the point estimate for PE30 exceeding that for PE10. Specifically, correct selection entails that the estimated PE30 is greater than the estimated PE10 and that PE30 is significantly > 0% (1-sided  $\alpha = 0.025$ )

<sup>#</sup> Cumulative hazard-based 2-sided Wald tests comparing HIV-1 incidence between the 10 mg/kg and 30 mg/kg mAb groups. Rejection of the null hypothesis requires that PE30 is significantly > 0% (1-sided  $\alpha = 0.025$ )

## 4.6 Sample size calculations for safety

We consider the statistical power of Fisher's exact test to detect a higher rate of SAEs in a mAb group (Group 1 or 2 with n=634) versus the control group (Group 3 with n=634). Based on HVTN vaccine trials from December 2000 through April 2014, about 4% of participants who received placebos experienced an SAE. The tests use a 2-sided  $\alpha$ -level of 0.05. This level does not correct for the 4 comparisons; however this is appropriate because it is desirable to maximize power to detect a safety problem. For the safety calculations, we assume no missing data as almost all participants will have some follow-up data for safety.

To describe the precision of the study to characterize differences in SAE rates between groups, Table 4-5 shows 2-sided 95% CIs for different levels of observed differences (mAb group-control) of event rates between a mAb group of size n1 = 634 (or the combined mAb groups n2 = 1268) and a control group of size n0 = 634.

Table 4-5 Two-sided 95% CIs for different observed event rate differences of safety endpoints between the mAb recipient and control groups\*

| Observed<br>event rate in<br>controls<br>(n0 = 634) | Observed event<br>rate in single<br>mAb group<br>(n1 = 634) | Observed event<br>rate in<br>combined mAb<br>groups<br>(n1 = 1268) | Rate<br>difference<br>(mAb group<br>– control) | 95 % CI<br>(n1 = 634) | 95% CI<br>(n1 = 1268) |
|---|---|---|---|---|---|
| 0% | 2% | 2% | 2% | (0.0116, 0.0341) | (0.0136, 0.0293) |
| | 4% | 4% | 4% | (0.0273, 0.0582) | (0.0305, 0.0523) |
| | 10% | 10% | 10% | (0.0790, 0.1258) | (0.0847, 0.1177) |
| | 20% | 20% | 20% | (0.1707, 0.2329) | (0.1789, 0.2229) |
| 2% | 2% | 2% | 0% | (-0.0164, 0.0164) | (-0.0155, 0.0126) |
| | 4% | 4% | 2% | (0.0013, 0.0403) | (0.0032, 0.0351) |
| | 10% | 10% | 8% | (0.0553, 0.1075) | (0.0598, 0.1000) |
| | 20% | 20% | 18% | (0.1482, 0.2114) | (0.1554, 0.2049) |
| 4% | 2% | 2% | -2 % | (-0.0403, -0.0013) | (-0.0394, -0.0044) |
| | 4% | 4% | 0% | (-0.0222, 0.0222) | (-0.0205, 0.0177) |
| | 10% | 10% | 6% | (0.0325, 0.0891) | (0.0365, 0.0822) |
| | 20% | 20% | 16% | (0.1261, 0.1957) | ( 0.1327, 0.1867) |

<sup>\*95%</sup> CIs are computed using the method of Miettinen and Nurminen [119]. Entries are bolded where significantly more events are observed among mAb recipients than among control recipients based on the 95% CI.

Figure 4-5 shows the power to detect an elevated SAE rate as a function of the true rate in the mAb group under consideration.



Figure 4-5 Power to detect a greater SAE rate in a mAb group versus the control group given a 4% SAE rate in the control group (2-sided 0.05-level test)

Figure 4-5 shows that there is 80% power to detect a higher SAE rate in a mAb arm if the true SAE rate is 7.8% and 90% power if the true rate is 8.5%.

# 4.7 Monitoring of the trial

#### 4.7.1 Role of the Data and Safety Monitoring Board (DSMB)

The study DSMB will review study data at 6-monthly interim analyses to evaluate safety, integrity, and efficacy of the ongoing trial. Following each DSMB meeting, the DSMB reports to the Oversight Committee (OC) a summary of the trial review, which may include recommendations to modify or terminate the trial. The DSMB is guided by a trial monitoring plan, and reviews and approves the monitoring plan before the trial initiates.

Each 6-monthly DSMB report will include a complete analysis of safety data. If a total of N=20 participants reach the Week 12 study visit before the first DSMB report is generated, then a safety report based on these data will be provided to the DSMB as soon as possible and before the first DSMB meeting. The contents of the early report are the same as the contents in the scheduled 6-monthly DSMB reports.

In addition, as soon as 10 grade 2 or higher AEs occur, a report will be generated describing these AEs and will be provided to the DSMB. The DSMB reports will also tabulate occurrence of SAEs, and of AEs judged related to product, accounting for the number of infusions received.

# 4.7.1.1 Sequential monitoring for potential harm, non-efficacy, and high efficacy

The trial uses sequential monitoring of the mAb groups versus control to stop early for:

- Potential harm [Establish that PE (pooled over the mAb groups) < 0% based on a 2-sided monitoring-adjusted 90% CI lying below 0%]
- Non-efficacy [Establish that PE (pooled over the mAb groups) < 40% based on a 2-sided 95% nominal CI lying below 40%]
- High efficacy [Establish that PE (pooled over the mAb groups) > 70% based on a 2-sided 95% nominal CI lying above 70%]

The sequential monitoring is based on CIs in order that the result of the study that would be reported would convey evidence supporting the conclusion of potential harm, non-efficacy, or high efficacy. Freidlin, Korn, and Gray [120] discuss a rationale for this approach to non-efficacy monitoring. The sequential monitoring for potential harm is based on monitoring-adjusted 1-sided 0.05-level tests (instead of 1-sided 0.025-level tests) for prudence to protect the safety of study participants (ie, less precision is required to meet a guideline for potential harm than to meet guidelines for non-efficacy or high-efficacy). Once non-efficacy monitoring commences, the potential harm monitoring after each infection ceases, as the non-efficacy monitoring now provides the function of detecting an elevated rate of HIV-1 infection. The non-efficacy monitoring is supplemented with conditional power calculations that report estimates of the probability of rejecting the null hypothesis of zero PE under different assumptions about the estimated PE if the trial were to continue to the end. The sequential monitoring plan is summarized in Table 4-6 and Figure 4-6.

Table 4-6 Summary of sequential monitoring of PE

| Monitoring<br>Type | Hypotheses | Testing Approach | Size of Test | Stopping Boundary | Timing of Interim Analyses |
|---|---|---|---|---|---|
| Potential<br>Harm | H0: PE ≥ 0%<br>vs<br>H1: PE < 0% | Exact 1-sided binomial<br>test of the fraction of<br>infections assigned to<br>receive the mAb | Specified in<br>the<br>monitoring<br>plan | Near-constant 1-sided p-<br>value cut-off controlling<br>the FWER at α = 0.05* | After every infection from 20 <sup>th</sup> total until first non-efficacy analysis |
| Non-<br>Efficacy | H0: PE ≥ 40%<br>vs<br>H1: PE < 40% | 2-sided Wald test and<br>1:1 corresponding 2-<br>sided 95% CI | 1-sided<br>α = 0.025 | Nominal 2-sided 95% CI<br>below 40% supplemented<br>with conditional power<br>(specified in the<br>monitoring plan) | 6-monthly starting<br>based on an event-<br>driven trigger<br>specified in the<br>monitoring plan |
| High<br>Efficacy | H0: PE ≤ 70%<br>vs<br>H1: PE > 70% | 2-sided Wald test and<br>1:1 corresponding 2-<br>sided 95% CI | 1-sided<br>α = 0.025 | Nominal 2-sided 95% CI<br>above 70% | 6-monthly starting at the same time as for non-efficacy |

<sup>\*</sup> Equivalently, a monitoring-adjusted 2-sided 90% CI based on inversion of the test statistic lies below 0%. The 1-sided p-value significance threshold stopping boundaries after each infection event are specified in the study monitoring plan.



Figure 4-6 Stopping boundaries for the sequential monitoring based on 2-sided CIs (or on the corresponding 1-sided p values)

Details of the sequential monitoring plan will be provided in a separate trial monitoring plan. The sequential monitoring is closely related to what was done for the HVTN 505 HIV-1 vaccine efficacy trial [121] (background discussion in [73]).

# 4.7.2 Feasibility check and guideline for continuing enrollment as planned

In addition to the sequential monitoring of PE, feasibility monitoring is done for the first 120 enrolled participants. This feasibility monitoring is based on the first four 8-week intervals (Weeks 1 through 32) and evaluates whether an adequately high percentage of participants attend clinical visits and receive the infusions per the protocol. The guideline is based on an adequately high rate of study participation (participants remain engaged in the trial and have not declined further infusions) supplemented by data on visit attendance, which corresponds to adherence to receipt of infusions. Additional details will be provided in the trial monitoring plan.

The feasibility monitoring based on the first 120 enrolled participants will use the following guideline for continuing enrollment as planned: continued participation by the Week 32 visit pooled over the 3 groups is greater than 80%.

If the blinded criterion fails to be met, the Protocol Team, in discussions with the DSMB and OC, will discuss whether modification or termination of the trial is warranted.

## 4.7.3 Monitoring for futility to assess PE

The objective of monitoring the trial for futility to assess PE is to monitor progress toward the minimal needed target number of treatment arm-pooled HIV-

1 primary endpoint infections by the Week 80 visit in the MITT cohort. Two targets are monitored for:

- 1. the total number of HIV-1 infections needed to achieve the planned 90% power to detect PE = 60%, and
- 2. the total number of HIV-1 infections needed to achieve 50% power to detect PE = 60%,

each using a 1-sided 0.025-level Wald test of H0: PE  $\leq$  0% against H1: PE > 0%, assuming proportional hazards of HIV-1 infection in the pooled VRC01 and control groups. The target numbers in (1) and (2) are 57 and 21, respectively (calculated by solving equation (1) in Schoenfeld [122]. The rationale for considering the two targets is as follows: (i) if the trial cannot achieve the planned 90% power to detect PE = 60%, considerations about enrollment modification or expansion are warranted, and (ii) if the trial cannot achieve even 50% power to detect PE = 60%, considerations about completing the trial early for futility to assess PE are warranted.

Two versions of the futility monitoring report will be generated. A report provided to the DSMB will be included in 6-monthly closed DSMB reports, starting in November 2017, and will report:

- a. the estimated distribution of the total (i.e., treatment arm-pooled) number of HIV-1 infections, with corresponding power to reject H0:  $PE \le 0\%$  using a 1-sided 0.025-level Wald test under the alternative hypothesis PE = 60% throughout the trial,
- b. the estimated probability that the total number of HIV-1 infections is  $\geq 57$  (target 1) with 95% credible intervals,
- c. the estimated probability that the total number of HIV-1 infections is  $\geq 21$  (target 2) with 95% credible intervals,
- d. the estimated distribution of the number of HIV-1 infections in each of the three treatment arms.

The distributions in (a) and (d) will also be summarized by the mean number of HIV-1 infections with a Wald 95% confidence interval. The estimation procedure for (a)–(d) will be conducted under each of the following two scenarios:

• the treatment arm-pooled infection rate in (a)–(c) and the three treatment armspecific infection rates in (d) used for generating future data are based on a Bayesian model and the prior assumption that PE = 60% (the design alternative), and • the treatment arm-pooled infection rate in (a)–(c) and the three treatment arm-specific infection rates in (d) used for generating future data are based on a Bayesian model and the prior assumption that PE = 0% (the null hypothesis).

The reason for conducting the estimation procedure twice is that the purpose of the results for the 57 endpoint target (b) is to trigger considerations for trial modifications, whereas the purpose of the results for (c) is to trigger considerations for early trial completion due to futility, where it is desired to reach the guideline (b) more easily/readily than the guideline (c). Accordingly, the results for (b) are interpreted focusing on the prior of PE = 60%, which makes it more likely to reach a guideline than the prior of PE = 0%, and the results for the 21 endpoint target (c) are interpreted focusing on the prior of PE = 0%, which makes it less likely to reach a guideline than the prior of PE = 60%.

Furthermore, a treatment-blinded report will be generated for distribution to the OC after each DSMB meeting takes place and will report estimates listed in (a)–(c) above calculated based only on treatment-blinded data. The reported results pertaining to estimates (a)–(c) will be identical to those in the DSMB report.

While it is the primary responsibility of the OC to make decisions regarding trial operations and modifications based on the monitoring of treatment-blinded primary endpoints, given the resource issues involved, DSMB review is also needed because issues of scientific integrity are also involved. More specifically, the DSMB can evaluate the progress toward primary endpoint targets in the context of the treatment-unblinded data, and based on this review may recommend to the OC to complete the trial early due to reaching a guideline for futility to assess PE (specified below).

The monitoring for futility to assess PE includes the following guidelines for trial modifications:

- [Guideline for enrollment modifications] If, in the PE = 60% scenario for the prior distribution, the estimated probability of reaching at least 57 total infections is less than 25%, the Oversight Committee may consider enrollment modifications with the intention to be able to conduct the primary PE analysis with adequate power.
- [Guideline for futility] If, in the PE = 0% scenario for the prior distribution, the estimated probability of reaching at least 21 total infections is less than 25%, the DSMB may recommend completing the trial early based on the inability to conduct the primary PE analysis with adequate power. However, since this is a proof-of-concept trial, a high bar is desired for completing the trial early for futility, and therefore if this event occurs yet the non-efficacy monitoring has not started or the non-efficacy boundary has not been reached, then this guideline for futility also requires that the estimated PE for the pooled VRC01 vs. control arm is < 30% and the estimated PE for the VRC01 30 mg/kg vs. control arm is < 30%.

If enrollment is incomplete at the time of an interim futility analysis, then the outlined estimation procedures will use the average observed enrollment rate in approximately the last 6 months for generating future enrollment data. In addition, a Bayesian approach will be used for generating future HIV-1 incidence data, conditional on observed data to-date. More specifically, the estimates in (a)–(c) will condition on the observed to-date treatment arm-pooled HIV-1 incidence rate, whereas the estimates in (d) will condition on the observed to-date (three) treatment arm-specific HIV-1 incidence rates. All estimates in (a)–(d) will also use the observed to-date treatment arm-pooled dropout rate for generating future dropout data.

If, at any time, these guidelines for futility to assess PE are met and yet it appears that value exists in continuing the trial, the statisticians will provide the DSMB and the OC with additional information, as appropriate, for use in their consideration of whether to recommend early trial completion.

#### 4.8 Assessment of PrEP use

The use of oral FTC/TDF as PrEP (either off-study or provided in the study) may impact study outcomes (eg, by lowering HIV incidence with a loss of study power). Dried blood spot samples will be collected and stored for assessment of quantitative concentrations of intracellular TFV (see Section 9.6), using a calendar based selection of visits that will ensure representative sampling of participants across the entire visit schedule at all sites throughout the study. A detailed testing plan, specified in the study monitoring plan, has been developed to prospectively monitor FTC/TDF use during the trial to inform the DSMB, and assess the potential impact of FTC/TDF use on PE of the study product. Prevalence of PrEP will be reported both as the estimated proportion of participant visits with highly adherent PrEP use (above the concentration of TFV designated as consistent with daily dosing) and the proportion of participant visits with any detectable PrEP use (concentration of TFV above the lower limit of detection for the dried blood spot assay). Additionally, we will use knowledge of PK quantitative levels to estimate the proportion of study person years protected by highly adherent use of FTC/TDF. PrEP use measures will be reported by arm to the DSMB; in addition both the OC and the protocol team leadership will see pooled estimates of FTC/TDF use.

#### 4.9 Randomization

The randomization sequence will be obtained by computer-generated random numbers and provided to each CRS through a Web-based randomization system. The randomization will be done in blocks to ensure balance across arms. At each institution, the pharmacist with primary responsibility for dispensing study products is charged with maintaining security of the treatment assignments (except in emergency situations as specified in the SSP).

# 4.10 Blinding

Participants and site staff (except for site pharmacists) will be blinded as to participant treatment arm assignments. Study product assignments are accessible to those CRS pharmacists, DAIDS protocol pharmacists and contract monitors, and SDMC staff who are required to know this information in order to ensure proper trial conduct. Any discussion of study product assignment between pharmacy staff and any other CRS staff is prohibited.

When a participant leaves the trial prior to study completion, the participant will be told he or she must wait until all participants are unblinded to learn his or her treatment assignment.

Emergency unblinding decisions will be made by the site investigator. If time permits, the HVTN 703/HPTN 081 PSRT should be consulted before emergency unblinding occurs.

### 4.11 Statistical analyses

This section describes the final study analyses, unblinded as to treatment arm assignment. All data from enrolled participants will be analyzed according to the initial randomization assignment regardless of how many infusions they received. In the rare instance that a participant receives the wrong treatment at a specific infusion visit, the Statistical Analysis Plan will address how to analyze the participant's safety data. Analyses are modified intent-to-treat (MITT) in that individuals who are randomized but not enrolled do not contribute data and hence are excluded. Because of blinding and the brief length of time between randomization and enrollment—typically no more than 4 working days—very few such individuals are expected.

Analyses for primary endpoints will be performed using SAS and R. All other descriptive and inferential statistical analyses will be performed using SAS, StatXact, or R statistical software.

# 4.11.1 Analysis variables

The analysis variables consist of baseline participant characteristics, safety, efficacy, and markers of mAb characteristics for primary- and secondary-objective analyses.

#### 4.11.2 Baseline comparability

Treatment arms will be compared for baseline participant characteristics using descriptive statistics.

## 4.11.3 Safety/tolerability analysis

Since enrollment is concurrent with receiving the first infusion, all participants will have received at least 1 infusion and therefore will provide some safety data.

## 4.11.3.1 Reactogenicity

The number and percentage of participants experiencing each type of reactogenicity sign or symptom will be tabulated by severity and treatment arm and the percentages displayed graphically by arm. For a given sign or symptom, each participant's reactogenicity will be counted once under the maximum severity for all injection visits. In addition, to the individual types of events, the maximum severity of local pain or tenderness, induration, or erythema, and of systemic symptoms will be calculated. Kruskal-Wallis tests will be used to test for differences in severity between arms.

#### 4.11.3.2 AEs and SAEs

AEs will be summarized using MedDRA System Organ Class and preferred terms. Tables will show by treatment arm the number and percentage of participants experiencing an AE within a System Organ Class or within preferred term category by severity or by relationship to study product. For the calculations in these tables, a participant with multiple AEs within a category will be counted once under the maximum severity or the strongest recorded causal relationship to study product. Formal statistical testing comparing arms is not planned since interpretation of differences must rely heavily upon clinical judgment.

A listing of SAEs reported to the DAIDS Regulatory Support Center (RSC) Safety Office will provide details of the events including severity, relationship to study product, time between onset and last infusion, and number of infusions received.

# 4.11.3.3 Local laboratory values

Box plots of local laboratory values will be generated for baseline values and for values measured during the course of the study by treatment arm and visit. Each box plot will show the first quartile, the median, and the third quartile. Outliers (values outside the box plot) will also be plotted. If appropriate, horizontal lines representing boundaries for abnormal values will be plotted.

For each local laboratory measure, summary statistics will be presented by treatment arm and timepoint, as well as changes from baseline for postenrollment values. In addition, the number (percentage) of participants with local laboratory values recorded as meeting Grade 1 AE criteria or above as specified in the DAIDS AE Grading Table (see Section 10.2.2) will be tabulated by treatment arm for each postinfusion timepoint. Reportable clinical laboratory abnormalities without an associated clinical diagnosis will also be included in the tabulation of AEs described above.

## 4.11.3.4 Reasons for infusion discontinuation and early study termination

The number and percentage of participants who discontinue infusions and who terminate the study early will be tabulated by reason and treatment arm.

### 4.11.4 Efficacy analysis

### 4.11.4.1 General approach

For the statistical analysis of prevention efficacy, data from enrolled participants will be used according to the initial randomization assignment regardless of how many infusions they received. Given that all or almost participants will receive the first infusion, the analyses are MITT, where all participants HIV-1 negative at entry receiving the initial infusion are included in the analysis, participants are analyzed according to their randomized treatment assignment, and participants retrospectively determined to be HIV-1 infected at entry based on treatment blinded procedures are excluded from the analysis. Additional analyses may be performed, limited to participants who received most or all infusions per protocol.

Cumulative incidences of HIV-1 infection over time for different treatment arms and pooled treatment arms will be estimated by a transformation of Nelson-Aalen estimators [123] for the respective cumulative hazard functions of HIV-1 infection. PE parameters will be estimated by one minus the ratio (mAb/control group) of these cumulative incidence estimators. Point estimates and 95% Wald CIs about cumulative incidence curves and PE(t) curves will be plotted. For the final timepoint of 80 weeks, 2-sided Wald p-values will be reported. These procedures will be used to test the hypotheses listed in Section 4.2.

As a supportive analysis for the hypotheses listed in Section 4.2, targeted maximum likelihood estimation (tMLE) will be used to estimate cumulative incidences of HIV-1 infection over time for different treatment arms and pooled treatment arms [124,125]. The Statistical Analysis Plan will describe the details of implementation of the tMLE estimators in an automated and objective fashion. PE parameters will be estimated by 1 minus the ratio (mAb group/control) of these tMLE estimators. Point estimates and 95% Wald CIs about cumulative incidence curves and PE(t) curves will be plotted. For the final timepoint of 80 weeks, 2-sided Wald p-values will be reported.

In addition to studying PE based on cumulative incidences of HIV-1 infection over time, complementary secondary analyses will assess hazard-ratio based PE using Cox proportional hazards models with score tests stratified by VRC01 dose group for testing whether PE differs from zero. This analysis uses as the failure time the time from the most recent infusion to the estimated date of HIV infection, entered in the Cox model as a time-dependent covariate. This analysis can have increased power to detect prevention efficacy compared to the primary analysis of the cumulative incidence based parameter PE, if instantaneous prevention efficacy is higher when VRC01 concentrations are lower. Goodness-of-fit diagnostics will be applied to assess veracity of the proportional hazards

assumption. The Cox models are selected for the secondary analysis instead of the primary analysis in order that the validity of the primary analysis does not depend on the proportional hazards assumption. The Cox model will also be used for a secondary analysis of PE in subgroups defined by the level of cumulative infusion adherence over time included in the model as a time-varying covariate.

Sensitivity analyses of the primary analysis will test H0: PE = 0% with a log-rank test and with a Gehan-Wilcoxon test stratified by VRC01 dose group. To explore potential time-variations in prevention efficacy, instantaneous prevention efficacy over time defined based on the instantaneous hazard ratio (VRC01 vs. placebo) will be estimated with pointwise and simultaneous confidence bands using nonparametric kernel smoothing [126].

## 4.11.5 Analyses prior to end of scheduled follow-up visits

Any analyses conducted prior to the end of the scheduled follow-up visits should not compromise the integrity of the trial in terms of participant retention or safety or efficacy endpoint assessments.

# 4.11.6 Specific approach for assessing PE, PE10, PE30

Primary objective 2 is addressed based on comparing cumulative HIV-1 incidence between the group of participants assigned to receive the VRC01 mAb (at either dose pooling over the two doses) and the group of participants assigned to the control group, and secondarily between each individual mAb dose group and the control group. For each prevention efficacy parameter PE, PE10 and PE30, point and 2-sided 95% CI estimates will be reported, along with the 2-sided p-values for testing the respective null hypotheses (with 2-sided p = 0.05 the threshold for a significant effect). Unadjusted and Holm-Bonferroni p-values will be reported for testing of the secondary endpoint efficacy parameters PE10 and PE30.

# 4.11.7 Assessment of individual-level markers of VRC01 mAb that correlate with protection against HIV infections (Secondary objective 1)

Secondary objective 1 is addressed based on the measurement of VRC01 mAb markers over time in mAb group breakthrough HIV-1—infected cases and in a random sample of HIV-1—uninfected mAb group participants (marker subset), integrated with the genotypic and phenotypic sieve analysis of breakthrough HIV-1 viruses accounting for knowledge of the VRC01 antibody footprint. The main analyses of the secondary objective 1 pool over the two mAb doses to maximize statistical power.

The design and results requirements for successful identification of correlates of protection in secondary objective 1 are:

1. Sufficient sample size to observe enough participants diagnosed with incident HIV-1 infection during the primary follow-up period of 80 weeks postenrollment in the mAb arms

- 2. A result of significant beneficial overall mAb PE > 0%
- 3. Sufficiently frequent HIV-1 testing schedule and accurate HIV-1 diagnostics
- 4. Wide variability in the concentration and effector functions of the mAb over time and/or individuals, and the ability to measure these characteristics such that their timing relative to the timing of HIV-1 acquisition is estimated with adequately low measurement error
- 5. mAb marker sampling design that allows sufficiently accurate PK modeling of mAb characteristics over time

Note that the serum concentration mAb markers (secondary endpoints 2) are defined without reference to a particular HIV-1 Env sequence. The effector function markers (also secondary endpoints 2) are relative to specific HIV-1 Envs or panels of Envs, and thus may be linked to immunogenicity endpoints (and the antigen reagents for those endpoints) that would be used in future trials of candidate HIV-1 vaccines. Correlates of protection analyses directly assess how mAb PE depends on markers.

# 4.11.7.1 Sampling of mAb markers

Characteristics of the mAb or immune responses to the mAb are measured in participants assigned to the mAb treatment groups, and in a small number of participants assigned to the control group. The sampling design determining the set of participants for measuring the markers will be finalized after the primary analysis results. This sampling design will include measuring the markers in all mAb group primary endpoint cases with a minimal number of samples available prior to diagnosis of HIV-1 infection, and on a random sample of participants from each mAb group who complete follow-up to the Week 96 visit HIV-1 negative (mAb group control participants). The random sample of HIV-1 uninfected controls is chosen to create a common control:case ratio across participant strata defined by factors such as dose group, infusion adherence, and calendar period of enrollment. For participants assigned to the control group, a smaller number of cases and HIV-1 negative controls will be sampled for measurement of markers. The timing of marker measurements is as follows:

- mAb group and control group cases: visits every 4 weeks up until the time of HIV-1 diagnosis and Day 61 (5 days post second infusion) if before diagnosis, plus the first positive visit and additional time-points post HIV-1 infection
- mAb group and control group marker subset controls: visits every 4 weeks through Week 80 plus Day 61 and Weeks 88 and 96

The Day 5 post-second infusion visit is included because it occurs shortly after the end of the distributive phase of the mAb, which together with the samples drawn just before infusions (Week 0, 8, ..., 72), the samples drawn 4 weeks post-

infusions (Week 4, 12, ..., 76), and the Week 80, 88, and 96 samples 8–24 weeks post last infusion constitute the basis for modeling marker curves over time.

# 4.11.7.2 Overview of the analysis of a mAb marker as a correlate of protection

A correlates of protection statistical analysis plan will be finalized not using any information on case-control status of participants; this plan will contain details of the statistical analysis. We provide a brief summary here. For a given mAb recipient, let S(t) be a marker characteristic at time t postenrollment in days, for example the time-concentration curve. The entire curve S(t) cannot be known exactly given that the marker is measured at a grid of time-points. A PK model will be used to express S(t) as a function of the measured marker readouts and error terms. One approach to the correlates of protection analysis will estimate the "prevention efficacy curve" PE(S(t) = s) defined as

$$PE(S(t) = s) = [1 - (hazard-mAb(S(t) = s))/(hazard-control(S(t) = s))] \times 100\%$$

where hazard-mAb(S(t) = s) is the hazard rate of HIV-1 infection at time t for a participant assigned to either mAb group with S(t) = s and hazard-control(S(t) = s) is the hazard rate of HIV-1 infection at time t for a participant assigned to the control group who would have had S(t) = s had s/he been assigned to the same mAb group (thus S(t) is a counterfactual random variable for control recipients). Similar parameters are used for assessing time-dependent correlates of protection in vaccine efficacy trials. A time-dependent parameter is used because interest centers on understanding how the current value of a mAb marker associates with the level of instantaneous PE given exposure with an HIV-1 virus at that time. The statistical analysis plan will describe the methods used to estimate PE(s) over the range of values s of a mAb marker characteristic. In addition to estimation, hypothesis testing will be performed to assess whether a mAb marker modifies PE, ie, testing

H0: 
$$PE(S(t) = s) = PE$$
 versus H1:  $PE(S(t) = s)$  varies in s. (1)

Rejecting H0 in favor of H1 supports the role of the marker in protection. The correlates of protection analysis pools over the two mAb groups, for the purpose of improving power both through a larger sample size and through greater interindividual variability of the mAb markers. Given that the exact dates of infusions have a major impact on mAb markers S(t) such as concentration over time (eg, notice the profound influence of missed infusions on S(t) in Figure 2-9), the analysis accounts for the exact dates of infusions that are expected to show considerable heterogeneity across trial participants.

#### 4.11.7.3 A time-window approach to assessing mAb correlates of protection

To explain the concept of this approach, first suppose all participants received all scheduled infusions and rigidly followed the visit schedule. Then this approach compares HIV-1 incidence during the first 4 weeks of the infusion intervals (ie, weeks 1-4, 9-12, 17-20, ..., 73-76) to HIV-1 incidence during the second 4 weeks

of the infusion intervals (ie, weeks 5-8, 13-16, 21-24, ..., 77-80), aggregating over the ten 8-week infusion intervals. Because the mAb has much higher concentration during the first halves of the infusion intervals compared to the second halves (eg, demonstrated in Figure 2-9), detection of higher HIV-1 incidence in the second halves of visit windows would imply that higher concentrations are associated with a lower rate of HIV-1 infection.

However, because of missed infusions and the heterogeneity among participants of infusion dates (which is allowable as specified by broad visit windows), a better approach accounts for the set of exact infusion dates of each participant. As such, our approach to implementing the time-window approach compares the mean time between the last infusion and infection for VRC01 group cases, with the mean of the participant-specific weighted average time between infusions of VRC01 group control participants, where the weights allow for changing HIV-1 incidence over time. The analysis stratifies by the 10 mg/kg and 30 mg/kg dose groups and aggregates estimates over these two dose groups. In addition, an important element of the analysis uses predictions of the HIV-1 infection times for all VRC01 group cases. Models for these predictions are built using information on HIV-1 diagnostic tests, intra-host diversity of HIV-1 sequences, HIV-1 viral loads, and perhaps other factors. Initial research to build predictors of HIV-1 infection time based on HIV-1 sequence information has been conducted using validation data sets of acutely HIV-1 infected individuals [127].

A related approach to assessing correlates or protection integrates a pharmacokinetic model of the serum concentration of VRC01 over time, comparing the mean VRC01 concentration at the time of HIV infection for VRC01 group cases with the mean of participant-specific weighted average VRC01 concentrations over follow-up time. The participant-specific average VRC01 concentration over follow-up time is intended to reflect the expected concentration at the time of a random HIV exposure, with weighting used as above to allow for changing HIV-1 incidence over time. Details of these statistical methods will be provided in the statistical analysis plan.

#### 4.11.7.4 mAb markers

For effector function markers measured based on a sample from a mAb recipient, the markers are measured to each of a panel of HIV-1 Envelope proteins. The most relevant HIV-1 Env panel represents the VRC01 antibody footprint diversity of viruses exposing trial participants. For example, relevant for the study population that is mostly exposed to subtype C HIV-1, Figure 4-7 shows a logo plot of the VRC01 antibody footprint motifs comprising 35 amino acid sites [19] based on 444 subtype C sub-Saharan African sequences deposited in the Los Alamos National Laboratory (LANL) sequence database between 2006 and 2014.



Figure 4-7 Logo plot of the VRC01 antibody footprints that occur in 444 subtype C sub-Saharan African sequences deposited in the LANL sequence database between 2006 and 2014

During the conduct of the trial the research team will determine a minimal set of Envs constituting a panel capturing most of the VRC01 mAb footprint diversity of exposing viruses. One effector function marker of interest for assessing as a correlate of protection is the weighted area under the magnitude-breadth neutralization curve of the mAb footprint Env panel, where the weighting is by the estimated prevalence of mAb footprints in HIV-1s circulating at the trial sites during the trial.

For mAb group participants with a primary study endpoint (breakthrough HIV-1 infection during the first 80 weeks), an important marker is the level at which his/her pre-infection sample at the time of HIV-1 acquisition neutralizes his/her particular breakthrough virus. (This analysis requires modeling the marker at the time of HIV-1 acquisition based on the available grid of marker measurements.) A result where sera from infected participants generally fail to neutralize their founding viruses would support neutralization as a correlate of protection. This analysis is repeated for other effector functions as a way to discriminate which effector functions are or are not correlates of protection, and to rank the effector functions by their contribution to explaining the level of protection.

## 4.11.7.5 Statistical power for assessing a mAb marker as a correlate of protection

The marker S(t) must vary within mAb recipients over time and/or among mAb recipients in order to detect a correlate of protection, with more variability in one or both components providing greater statistical power to detect a correlate of protection via testing the null hypothesis of equation/panel (1) above. In essence, to detect correlates of protection it is necessary that a large fraction of person-years at risk are in high protection zones and a large fraction of person-years at risk are in low protection zones. (A "high protection zone" is a period of time during which a mAb recipient has high levels of a marker and high levels of efficacy.) Data from VRC 601, VRC 602, and HVTN 104 show wide variability in the mAb concentration over time, and more limited variability among mAb recipients. HVTN 104 will provide more data on these two aspects of marker variability. The limited among-mAb recipient variability motivates the study design that randomly assigns participants to 2 different mAb doses in order to create inter-individual variability.

Achieving adequate power to detect correlates of protection requires that the HIV-1 diagnostic testing is more frequent than the infusion schedule. This is why diagnostic visits every 4 weeks are advantageous given infusions every 8 weeks, and procedures may be determined and applied to test for HIV-1 infection more frequently than every 4 weeks. The data from all of the employed diagnostic testing kits is incorporated into the modeling of S(t) and of HIV-1 infection times, and is integrated into the statistical analysis for estimation and testing of PE(S(t) = s). Lastly, achieving adequate power to detect correlates of protection requires studying markers that can be measured with a high ratio of potentially protection relevant variability versus protection irrelevant variability, where the latter variability could stem from technical measurement error of the assay or to error in estimation of the timing of infection. Because of this fact the trial design relies on parallel assay studies to qualify marker variables for the analysis and relies on development and characterization of models for S(t) over continuous time t.

We provide one power calculation for assessing a trichotomous marker S(t), the concentration of the mAb at time t post enrolment, as a correlate of protection, which divides the pooled mAb group at a given time t by two thresholds of marker response  $[S(t) = 0 \text{ indicates Low}, S(t) = 1 \text{ indicates Medium}, \text{ and } S(t) = 2 \text{ indicates High for some pre-set definitions of Low}, Medium}, High]. Thus at any given time t after entry, <math>S(t)$  divides the pooled mAb group into three subgroups. In our illustration we take "0" to be a VRC01 serum concentration  $\leq 50 \text{ mcg/mL}$ , "2" to be a VRC01 serum concentration > 10 mcg/mL, and "1" to be an intermediate serum concentration.

Based on Figure 2-4, we conduct a power calculation indexed by the percentage of person-years at-risk of mAb recipients that are in the (Low, Medium, High) zones, and indexed by the level of PE within each of these zones. As indicated in the figure, we expect that about (50%, 40%, and 10%) of the PYRs at risk in the 10 mg/kg mAb group are in the (Low, Medium, and High) regions whereas about (10%, 40%, and 50%) of the PYRs at risk in the 30 mg/kg mAb group are in the (Low, Medium, and High) regions. We consider power calculations pooling data across both mAb groups, assuming 30 mAb HIV-1—infected cases with data and 150 mAb group HIV-1—uninfected controls with data, assuming the design alternatives PE10 = PE30 = 60% approximating the numbers displayed in Table 4-3. The detailed mathematical assumptions of these power calculations will be provided in the statistical analysis plan.

Figure 4-8 shows power curves for the scenario that (30%, 40%, 30%) of PYRs at risk are in the (Low, Medium, High) zones (which we approximately expect to occur based on Figure 2-4) and PE10 = PE30 = (15%, 60%, 85%) in these zones. The power curves also account for noise in the measurement of S(t) via a parameter rho that equals the proportion of the inter-individual marker variability that is potentially protection relevant. The results show that the noise level majorly affects power, underscoring that only assays meeting qualification criteria will be studied as correlates. The parameter rho also reflects noise due to uncertainty in the exact times t of HIV-1 acquisition at which values of S(t) are

needed. For the scenario that this extra variability reduces rho to 0.7, there is about 80% power to detect a correlate of protection (with effect size 15%, 60%, 85% efficacy) at the selected trial sample size. Note that the parameter rho also reflects noise due to uncertainty in the exact times t of HIV-1 acquisition at which values S(t) are needed. A more extensive set of power calculations will be conducted based on HVTN 104 study data.

Power to Discriminate (Lo, Med, Hi) PE = (15%, 60%, 85%) [Overall PE = 60%] 30% with Lo and 30% with Hi Marker Response



2-phase logistic regression; 2-sided alpha = 0.05; controls:cases = 5:1

Figure 4-8 Power of the trial for detecting that PE varies over the three mAb marker-defined subgroups S(t) = Low, S(t) = Medium, and S(t) = High at level PE = 15%, 60%, 85%, respectively, for a marker with assay noise parameter rho = 1 (perfect marker), 0.9, 0.7, and 0.5 and percentages of person-years at risk in the (Low, Medium, High) marker regions set at (30%, 40%, 30%). The calculations at 1900 total participants assume 30 mAb group HIV-1–infected cases and 150 mAb group HIV-1–uninfected controls with data on S(t) and pool over both mAb groups. The dashed vertical line represents the sample size of the study.

Figure 4-9 shows the same power analysis as Figure 4-8, fixing rho = 0.9 (indicating a qualifying assay) and varying the percentage of PYRs at risk that are in the (Low, Medium, High) zones. The results show that power increases sharply with the percentage of mAb recipients that are in the Low and High regions, demonstrating the principle that variability in the marker is a strong determinant of power to detect a correlate of protection.

Power to Discriminate (Lo, Med, Hi) PE = (15%, 60%, 85%) [Overall PE = 60%; rho = 0.9]



2-phase logistic regression; 2-sided alpha = 0.05; controls:cases = 5:1

Figure 4-9 Power of the trial for detecting that PE varies over the three mAb marker-defined subgroups S(t) = Low, S(t) = Medium, and S(t) = High at level PE = 15%, 60%, 85%, respectively, for a marker with assay noise parameter rho = 0.9 and percentages of person-years at risk in the Low and High marker regions varied from 10%, 15%, 20%, 25%, 30%. The calculations at 1900 total participants assume 30 mAb group HIV-1-infected cases and 150 mAb group HIV-1-uninfected controls with data on S(t) and pool over both mAb groups.

### 4.11.7.6 Genotypic and phenotypic sieve analysis

Genotypic sieve analysis analyzes sequences of breakthrough HIV-1 infecting viruses from the earliest available postinfection sample and seeks to identify amino acid "signatures" that differentiate breakthrough sequences in the mAb groups versus the control group, in terms of differential PE against HIV-1s according to some genotypic characteristics. For example, the genotypic sieve analysis assesses differential PE against different genotypes of HIV-1 with genotype defined by:

- Number of mismatches to the VRC01 mAb footprint of the subtype C consensus sequence (subtype selected to match the circulating HIV-1s)
- Number of known mAb neutralization escape mutations in the mAb footprint
- Number of known mAb effector function escape mutations in the mAb footprint for non-neutralization effector functions such as ADCC, virion capture, and phagocytosis
- Number of potential N-linked glycosylation (PNG) sites within a given radius of the mAb footprint
- Length of variable loops in proximity to the mAb footprint

To illustrate the utility of genotypic sieve analysis, we consider a hypothetical result that would support that the mAb protects via specific neutralization targeting of the mAb's epitope. In this illustration, the HIV-1 genotype is defined by four ordered genotypes according to whether there are 0, 1, 2, or >2 neutralization escape mutations in the VRC01 mAb antibody footprint. The hypothetical result would be an estimated PE of 95% against HIV-1s with zero
escape mutations and a PE of 0% against HIV-1s with >2 neutralization escape mutations, and intermediate and monotone decreasing level of estimated PE against HIV-1 with one mutation and two mutations, respectively.

A second type of sieve analysis, phenotypic sieve analysis, compares breakthrough viruses between the mAb versus control groups using an immunological assay. Specifically, data from an "effector function checkerboard" is filled out, with the rows representing serum samples from a random sample of mAb recipients HIV-1 uninfected at the time of sampling, and the columns representing HIV-1 Env VRC01 footprint targets created from the breakthrough viruses. The phenotypic sieve analysis compares the sensitivity of the breakthrough viruses to mAb recipient sera between the mAb and control treatment groups. A second version of the phenotypic sieve analysis compares the sensitivity of the breakthrough viruses to the VRC01 mAb between the treatment groups; this latter analysis is simpler, based on a single column of data instead of a matrix, because it does not use mAb recipient sera. For an example of the second type of phenotypic sieve analysis, the TZM-bl neutralization assay could be performed on all control breakthrough HIV-1s versus VRC01 and on all mAb group breakthrough HIV-1s (pooled over the two mAb groups) versus VRC01, and a Wilcoxon rank sum test applied to assess a difference. Reduced TZM-bl neutralization sensitivity of the mAb breakthrough group viruses would support that neutralization had a role in protection and that the TZM-bl assay was able to detect this role, and would support using the TZM-bl assay as a tool for evaluating future candidate HIV-1 vaccines. The HVTN has previously conducted neutralization sieve analysis [128]. Figure 4-10 illustrates a genotypic and phenotypic sieve analysis.



Figure 4-10 Illustration of genotypic (left panel) and phenotypic (right panel) sieve analysis, where the left panel shows the distribution of the number of known neutralization escape mutations in breakthrough control and mAb group HIV-1 sequences, and the right panel shows the percentage of the panel of breakthrough HIV-1s that are neutralized at level 50% (IC<sub>50</sub>) by the given concentration of the VRC01 mAb.

Another phenotypic sieve analysis focuses on mAb group cases, and measures different effector functions of closest-to-infection participant serum samples or of the VRC01 mAb against the participant-matched breakthrough HIV-1s. The effector functions that tend to have low readouts against participant-matched breakthrough viruses compared to against the panel of control group HIV-1s or compared to an historic panel of HIV-1s are implicated as potential correlates of protection.

In addition, an important sieve analysis will assess PE against HIV-1s that are sensitive to neutralization by VRC01 as measured using the first post-infection sample (sensitive is defined by positive neutralization based on IC<sub>50</sub> or IC<sub>80</sub>). This PE parameter measuring prevention efficacy against neutralization sensitive HIV-1s is estimated (with confidence intervals and p-values) in the same way as genotype-specific PE described above. In addition, the same hypothesis testing procedure for detecting differential PE by two HIV-1 genotypes is applied for assessing differential PE by neutralization sensitive versus resistant HIV-1. Moreover, this sieve analysis of sensitive versus resist HIV-1 is also conducted with sensitive/resistant defined by positive/negative response of other assays besides neutralization (eg, ADCC, ADCP).

## 4.11.7.7 Illustration of power to detect a phenotypic sieve effect

We conduct power calculations based on TZM-bl neutralization IC<sub>50</sub> values (in mcg/mL) of VRC07 (a close cousin of VRC01) to approximately 100 viruses representing global HIV-1 diversity (data provided by Mark Louder, Robert Bailer, and John Mascola from the VRC). From the control group we sample 35 HIV-1 infections with IC<sub>50</sub> from the VRC07 data set, and from the pooled mAb group we sample 30 HIV-1 infections with IC<sub>50</sub> values bias sampled based on IC<sub>50</sub>-dependent PE, with PE(x) the probability an infected control recipient would be infected had she received the mAb with IC<sub>50</sub> value of x to the exposing virus. Figure 4-11 shows power for comparing the VRC01 IC<sub>50</sub> distribution of the pooled mAb group HIV-1s versus the control group HIV-1s, based on a twosample Wilcoxon rank sum test. The effect size indexing a difference between the two groups is equivalently expressed in terms of the PE(x) function (where a horizontal line indicates the null hypothesis of no difference) or in terms of a different cumulative distribution function of the IC<sub>50</sub> in the two groups. Four correlates effect sizes are considered, ranging from the weakest (Effect Size 1) to the strongest (Effect Size 4). The results show that there is moderate power to detect Effect Size 3 phenotypic sieve effects (second steepest curve in Figure 4-11, power = 0.793).



Figure 4-11 Power calculations for comparing IC<sub>50</sub> distributions between mAb group breakthrough HIV-1s and control group breakthrough HIV-1s, with difference equivalently expressed in terms of the PE(x) curve or the cumulative IC<sub>50</sub> distribution functions, where in the right panel the black/highest curve represents the distribution for the control group breakthrough HIV-1s.

Effect Size 3 is biologically plausible based on the following argument. Under the design alternative of 60% PE we expect a transition between full protection against the most sensitive viruses and zero protection against the most resistant viruses. Table 4-7 shows the percentage of susceptible viruses that are completely blocked by the VRC01 antibody and the percentage of viruses that are completely resistant to the antibody for each of the four specified effect sizes PE(x) in Figure 4-11. For example, for Effect Size 3, the most susceptible 11.6% of viruses are completely blocked (PE = 100%) while the most resistant 2.8% of viruses are completely resistant (PE = 0%) and there is a gradient of protection for the 85.6% of intermediate viruses between the two poles (Table 4-7). The wide range of neutralization (and Fc effector function) sensitivities of HIV-1s suggests that this range of prevention efficacies is plausible. For this effect size there is 79.3% power to detect a phenotypic sieve effect and hence a correlate of protection.

Table 4-7 Percentages of HIV-1s fully susceptible to VRC01 (PE = 100%) and fully resistant to VRC01 (PE = 0%) for the four different effect sizes studied in Figure 4-11

| PE(x) Effect Size in Figure 1-16 | Susceptible<br>[PE = 100%] | Resistant $[PE = 0\%]$ |
|---|---|---|
| Effect Size 4 | 41.9% | 23.3% |
| Effect Size 3 | 11.6% | 2.8% |
| Effect Size 2 | 1.0% | <0.1% |
| Effect Size 1 | <0.1% | <0.1% |
| Null Hypothesis | NA | NA |

The sieve analyses will be done including all MITT infected participants, as well as only including mAb group infected participants who received an infusion at the beginning of the 8-weekly interval during which HIV-1 infection was diagnosed.

# 5 Selection and withdrawal of participants

Participants will be healthy, HIV-uninfected (seronegative) adults who comprehend the purpose of the study and have provided written informed consent. Volunteers will be recruited and screened; those determined to be eligible, based on the inclusion and exclusion criteria, will be enrolled in the study. Final eligibility determination will depend on information available at the time of enrollment, including results of laboratory tests, medical history, physical examinations, and answers to self-administered and/or interview questions.

Investigators should always use good clinical judgment in considering a volunteer's overall fitness for trial participation. Some volunteers may not be appropriate for enrollment even if they meet all inclusion/exclusion criteria. Medical, psychiatric, occupational, or other conditions may make evaluation of safety and/or serum mAb concentration and efficacy difficult, and some volunteers may be poor candidates for retention.

Determination of eligibility, taking into account all inclusion and exclusion criteria, must be made within 56 days prior to enrollment unless otherwise noted in Sections 5.1 and 5.2.

#### 5.1 Inclusion criteria

#### General and Demographic Criteria

- 1. **Age** of 18 to 40 years
- 2. **Access to a participating CRS** and willingness to be followed for the planned duration of the study
- 3. Ability and willingness to provide **informed consent**
- 4. **Assessment of understanding**: volunteer demonstrates understanding of this study and completes a questionnaire prior to first infusion with verbal demonstration of understanding of all questionnaire items answered incorrectly
- 5. **Agrees not to enroll in another study** of an investigational research agent for the duration of the participant's trial participation
- 6. **Good general health** as shown by medical history, physical exam, and screening laboratory tests

#### **HIV-Related Criteria:**

7. Willingness to receive HIV test results

- 8. Willingness to **discuss HIV infection risks** and amenable to HIV risk reduction counseling
- 9. Persons born Female (assigned female sex at birth) and identifying as female, who, in the 6 months prior to randomization, has had vaginal and/or anal intercourse with a male partner

Volunteers who have been in a mutually monogamous relationship with an HIV-1 seronegative partner for > 1 year are excluded.

#### **Laboratory Inclusion Values**

#### **Hematology**

- 10. **Hemoglobin** (Hgb)  $\geq$  10.5 g/dL
- 11. Platelets  $\geq 100,000 \text{ cells/mm}^3$

#### **Chemistry**

12. ALT < 2.5 times the institutional upper limit of normal and creatinine  $\leq$  1.25 times the institutional upper limit of normal

#### **Virology**

13. HIV uninfected, as defined in the SSP, within 30 days prior to enrollment

#### **Urine**

14. Negative, trace, or 1+ (30 g/L for semi-quantitative) urine protein by dipstick

#### **Reproductive Status**

- 15. **Volunteers capable of becoming pregnant**: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed at the screening visit and prior to infusion on the day of initial infusion. Persons who are NOT capable of becoming pregnant due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records) are not required to undergo pregnancy testing.
- 16. **Reproductive status**: A volunteer who is capable of becoming pregnant must agree to consistently use effective contraception (see Appendix B and SSP) for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit.
- 17. Volunteers capable of becoming pregnant must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

#### 5.2 Exclusion criteria

#### General

- 1. **Investigational research agents** received within 30 days before first infusion
- 2. Body mass index (BMI)  $\geq 40$
- 3. Pregnant or breastfeeding
- 4. **Any reactive, indeterminate, or positive HIV test**, even if subsequent testing indicates that the individual is not HIV infected, except as permitted by the HVTN 703/HPTN 081 PSRT

#### Vaccines

5. **HIV vaccine(s)** received in a prior HIV vaccine trial. For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN 703/HPTN 081 PSRT will determine eligibility on a case-by-case basis.

#### **Immune System**

- 6. Serious adverse reactions to VRC01 formulation components such as sodium citrate, sodium chloride, and L-arginine hydrochloride, including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain.
- 7. **Autoimmune disease**, including Type I diabetes mellitus (Not excluded from participation: Volunteer with mild, stable and uncomplicated autoimmune disease that does not require consistent immunosuppressive medication and that, in the judgment of the site investigator, is likely not subject to exacerbation and likely not to complicate reactogenicity and AE assessments)
- 8. Immunodeficiency syndrome

#### Clinically significant medical conditions

- 9. Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:
  - Any contraindication to repeated infusions or blood draws, including inability to establish venous access;
  - A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period; or

- A condition or process for which signs or symptoms could be confused with reactions to VRC01.
- 10. **Any medical, psychiatric, occupational, or other condition** that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or infusion reactions, or a volunteer's ability to give informed consent
- 11. **Psychiatric condition that precludes compliance with the protocol**. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
- 12. **Asthma**, other than mild, well-controlled asthma
- 13. **Bleeding disorder** diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
- 14. **Malignancy** (Not excluded from participation: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure. or who is unlikely to experience recurrence of malignancy during the period of the study)
- 15. **Seizure disorder:** History of seizure(s) within past three years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
- 16. History of hereditary **angioedema**, acquired angioedema, or idiopathic angioedema
- 17. History of **receiving transplantation of life-saving organs or tissue** (includes heart, kidney, pancreas, lungs, liver, and intestines)
- 18. Known hepatic or renal dysfunction

#### 5.3 Participant departure from infusion schedule or withdrawal

This section concerns an individual participant's departure from the infusion schedule. Pause rules for the trial as a whole are described in Section 10.3.

#### 5.3.1 Delaying infusions for a participant

Under certain circumstances, a participant's scheduled infusion will be delayed. The factors to be considered in such a decision include but are not limited to the following:

• Prior to infusion, abnormal vital signs or clinical symptoms that may mask assessment of a study product reaction

- Intercurrent illness that is assessed by the site principal investigator (or designee) to require delay or withdrawal from the infusion schedule. The investigator may consult with the HVTN 703/HPTN 081 PSRT.
- Pregnancy: for participants who become pregnant infusions will be stopped. If
  the participant is no longer pregnant (as demonstrated by a negative urine or
  serum pregnancy test) and wants to continue with infusions, the HVTN
  703/HPTN 081 PSRT will be consulted to determine whether the participant
  may resume infusions or whether infusions should be permanently
  discontinued.

## 5.3.2 Participant departure from infusion schedule

Every effort should be made to follow the infusion schedule per the protocol. If a participant misses an infusion and the visit window period for the infusion has passed, then sites may consult the SSP.

## 5.3.3 Discontinuing infusions for a participant

Under certain circumstances, an individual participant's infusions will be permanently discontinued. Specific events that will result in stopping a participant's infusion schedule include:

- Co-enrollment in a study with an investigational research agent (rare exceptions allowing for the continuation of infusions may be granted with the unanimous consent of the HVTN 703/HPTN 081 PSRT);
- Clinically significant condition (ie, a condition that affects the immune system or for which continued infusions and/or blood draws may pose additional risk), including but not limited to the following:
  - Any grade 4 local or systemic reactogenicity symptom or AE that is subsequently considered to be related to study product;
  - An SAE that is subsequently considered to be related to study product;
  - Any grade 3 clinical AE (exception: fever or vomiting and subjective local and systemic symptoms) that is subsequently considered to be related to study product;
  - Any grade 3 or 4 lab abnormality confirmed by a repeated value that is subsequently considered to be related to study product;
  - Clinically significant hypersensitivity reaction including but not limited to type 1 hypersensitivity reaction and/or serum sickness associated with study product. Consultation with the HVTN 703/HPTN 081 PSRT is required prior to subsequent infusion following any hypersensitivity reaction associated with study product; or

• Investigator determination in consultation with Protocol Team leadership (eg, for repeated nonadherence to study staff instructions).

Infusions will be permanently discontinued for a participant diagnosed with HIV infection or with 2 reactive HIV tests, even if subsequent testing indicates that the participant is not HIV infected.

Participants for whom infusions are discontinued for reasons other than HIV infection should be counseled on the importance of continuing with the study and strongly encouraged to participate in Schedule 4 follow-up visits and protocol-specified procedures (see Appendix I and Appendix M), unless medically contraindicated.

## 5.3.4 Participant termination from the study

Under certain circumstances, an individual participant may be terminated from participation in this study. Specific events that will result in early termination include:

- Participant refuses further participation
- Participant relocates and remote follow-up or transfer to another CRS is not possible
- CRS determines that the participant is lost to follow-up
- Investigator decides, in consultation with Protocol Team leadership, to terminate participation (eg, if participant exhibits inappropriate behavior toward clinic staff)
- Any condition where termination from the study is required by applicable regulations.

# 6 Study product preparation and administration

CRS pharmacists should consult the Pharmacy Guidelines and Instructions for DAIDS Clinical Trials Networks for standard pharmacy operations. The protocol schema is shown in Table 1-1. See the IBs for further information about study products.

## 6.1 Study product regimen

The schedule of study product administrations is shown in Section 1 and additional information is given below.

Group 1 [Note – participants randomized under Version 1.0 were enrolled in this same treatment but under the assignment "Treatment 4(T4)"]

Treatment 1 (T1): VRC-HIVMAB060-00-AB 10 mg/kg in sufficient Sodium Chloride for Injection USP, 0.9% to prepare a final total volume of 150 mL IV at Weeks 0, 8, 16, 24, 32, 40, 48, 56, 64, and 72.

Group 2 [Note – participants randomized under Version 1.0 were enrolled in this same treatment but under the assignment "Treatment 5(T5)"]

Treatment 2 (T2): VRC-HIVMAB060-00-AB 30 mg/kg in sufficient Sodium Chloride for Injection USP, 0.9% to prepare a final total volume of 150 mL IV at Weeks 0, 8, 16, 24, 32, 40, 48, 56, 64, and 72.

Group 3 [Note – participants randomized under Version 1.0 were enrolled in this same treatment (control) but under the assignment "Control 6(C6)"]

Control 3 (C3): Control for VRC01 (Sodium Chloride for Injection USP, 0.9%) to be prepared as a final total volume of 150 mL IV at Weeks 0, 8, 16, 24, 32, 40, 48, 56, 64, and 72.

For all participants originally enrolled under Version 1.0, a new prescription must be written and sent to the pharmacy once the participant has consented under Version 2.0 with the appropriate 4-digit CODE written on the prescription as well as a way for the pharmacist to verify that the participant has consented under Version 2.

#### 6.2 Study product formulation

VRC-HIVMAB060-00-AB [VRC01, Labeled as VRC01 HIV MAb Drug Product VRC-HIVMAB060-00-AB]

VRC01 will be provided as a sterile clear, colorless to yellow isotonic solution, essentially free of visible particles; some white, opaque particles may be present. Each vial contains 100 mg / mL of VRC-HIVMAB060-00-AB in formulation buffer. The formulation buffer is composed of 25 mM sodium citrate, 50 mM sodium chloride, and 150 mM L-arginine hydrochloride at pH 5.8. Vials are intended for single use only and do NOT contain a preservative. The product should be stored frozen -35°C to -15°C with excursions permitted between -45°C and -10°C. The study products are described in further detail in the IB.

VRC01 is a highly concentrated protein solution and may develop white, opaque to translucent particles after thawing. When particles are observed, they may disappear after a few hours at room temperature or storage at 2°C to 8°C (36°F to 46°F).

Prior to preparation, vials containing VRC01 must be removed from the freezer and thawed for a minimum of 1 hour at controlled room temperature (maximum 27°C). Following this 1 hour thaw, the unopened vials of VRC01 may be stored for up to 24 hours at controlled room temperature (maximum 27°C) and/or up to 4 weeks at 2°C to 8°C. Product may NOT be thawed or stored in direct sunlight. Once thawed, product may NOT be refrozen.

Prior to preparation, vials should be swirled for 30 seconds with sufficient force to resuspend any visible particles, yet avoiding foaming. DO NOT SHAKE THE VIALS.

If particles are observed, return the vials to 2°C to 8°C storage.

If the particles re-dissolve within the maximum storage time of up to 4 weeks at 2°C to 8°C, the vials may be used for product preparation. Refrigerated product in the vial must be equilibrated at controlled room temperature (maximum 27°C) for a minimum of 30 minutes before preparation and must be used within 8 hours of removal from the refrigerator.

If particles continue to be observed after 4 weeks at 2°C to 8°C, do not use the vialed product for IV bag preparation. These vials must be quarantined until they are returned to the NIAID Clinical Research Products Management Center (CRPMC) or to the manufacturer upon request of the CRPMC or destroyed if directed by the CRPMC.

#### Control for VRC01 [Sodium Chloride for Injection USP, 0.9%]

Sodium Chloride for Injection USP, 0.9% will be used as the Control for VRC01. It must be stored as directed by the manufacturer. For sites who do not have access to Sodium Chloride for Injection USP, 0.9%, the Sodium Chloride for Injection, 0.9% that they use must meet the following criteria: a sterile solution of Sodium Chloride in Water for Injection which contains no antimicrobial agents. It is nonpyrogenic and is intended for intravenous administration.

#### 6.3 Preparation of study products

Prior to preparation of the first infusion (enrollment visit), a new prescription will be sent to the pharmacy. The prescription MUST contain the participant's weight based upon the participant's weight at the most recent visit where weight was measured (this includes screening) and randomization code (this may NOT be communicated verbally). If this information is NOT on the prescription, the prescription will be returned to the clinic from the pharmacy to be completed appropriately prior to the pharmacist beginning preparation of study product. Subsequent visit weights (based upon the participant's weight at the most recent visit where weight was measured) must be communicated to the pharmacy in writing prior to the day of the visit. Any changes in weight of more than 10% (between the prior weight and the weight on the day of the infusion visit) will require an updated visit weight communication to the pharmacy in writing so that product can be prepared based on that weight change.

Pharmacists should keep in mind that the preparation instructions below are considered medium risk per USP 38 General Chapter Physical Tests / <797> Pharmaceutical Compounding - Sterile, and should follow the requirements of their country, their institution, and their pharmacy regulatory authority regarding these procedures.

## 6.3.1 VRC-HIVMAB060-00-AB (10mg/kg IV) - (Group 1)

To prepare an IV infusion, the pharmacist will calculate the dose [total milligrams needed (10 mg/kg x participant's weight in kg)] and remove the total number of vials needed as well as a 100 mL IV bag of Sodium Chloride for Injection USP, 0.9% from storage. If the product has been stored at 2°C to 8°C, the vials should be equilibrated to room temperature for 30 minutes and may be held at room temperature (not to exceed 27°C) for up to 8 hours prior to product preparation. The pharmacist will also calculate the additional amount of Sodium Chloride for Injection USP, 0.9% needed to prepare a final total volume of 150 mL and remove this from storage.

Prior to preparation, the pharmacist should gently swirl the vials containing VRC01 and then inspect for particles. DO NOT SHAKE VIALS. If visible particles are present, the product will not be used (see Section 6.2 for more information). The pharmacist, using aseptic technique, will add the appropriate amount of Sodium Chloride for Injection USP, 0.9% to the 100 mL IV bag of Sodium Chloride for Injection USP, 0.9%. The pharmacist, still using aseptic technique will then add the appropriate volume of VRC01 to that same bag for a final total volume of 150 mL. The IV bag will be labeled as "VRC01 or Control in Normal Saline Total Volume = 150 mL". The weight used for calculating the dose should be written on the label. A bag cover will be placed over the bag and should not be removed by the clinic staff. The IV bag will be labeled with a DO NOT INFUSE after date and time as follows:

o 24 hours if stored at 2°C to 8°C

 8 hours, including completion of infusion, if stored at controlled room temperature (not to exceed 30°C)

Product may NOT be stored in direct sunlight.

Note: Site pharmacists must follow their institutional policies for expiration dates (ie, DO NOT INFUSE after date and time), if shorter than the timeframes above.

Any empty vials, unused portion of entered vials, or unused IV solution that contains study product should be discarded in a biohazard containment bag and incinerated or autoclaved in accordance with institutional or pharmacy policy.

## 6.3.2 VRC-HIVMAB060-00-AB (30mg/kg IV) - (Group 2)

To prepare an IV infusion, the pharmacist will calculate the dose [total milligrams needed (30 mg/kg x participant's weight in kg)] and remove the total number of vials needed as well as a 100 mL IV bag of Sodium Chloride for Injection USP, 0.9% from storage. If the product has been stored at 2°C to 8°C, the vials should be equilibrated to room temperature for 30 minutes and may be held at room temperature (not to exceed 27°C) for up to 8 hours prior to product preparation. The pharmacist will also calculate the additional amount of Sodium Chloride for Injection USP, 0.9% needed to prepare a final total volume of 150 mL and remove this from storage.

Prior to preparation, the pharmacist should gently swirl the vials containing VRC01 and then inspect for particles. DO NOT SHAKE VIALS. If visible particles are present, the product will not be used (see Section 6.2 for more information). The pharmacist, using aseptic technique, will add the appropriate amount of Sodium Chloride for Injection USP, 0.9% to the 100 mL IV bag of Sodium Chloride for Injection USP, 0.9%. The pharmacist, still using aseptic technique will then add the appropriate volume of VRC01 to that same bag for a final total volume of 150 mL. The IV bag will be labeled as "VRC01 or Control in Normal Saline Total Volume = 150 mL". The weight used for calculating the dose should be written on the label. A bag cover will be placed over the bag and should not be removed by the clinic staff. The IV bag will be labeled with a DO NOT INFUSE after date and time as follows:

- 24 hours if stored at 2°C to 8°C
- 8 hours, including completion of infusion, if stored at controlled room temperature (not to exceed 30°C)

Product may NOT be stored in direct sunlight.

Note: Site pharmacists must follow their institutional policies for expiration dates (ie, DO NOT INFUSE after date and time), if shorter than timeframes above.

Any empty vials, unused portion of entered vials, or unused IV solution that contains study product should be discarded in a biohazard containment bag and incinerated or autoclaved in accordance with institutional or pharmacy policy.

## 6.3.3 Control for VRC01 (Groups 3)

To prepare an IV infusion, the pharmacist, using aseptic technique, will add 50 mL of Sodium Chloride for Injection USP, 0.9% to a 100 mL bag of Sodium Chloride for Injection USP, 0.9%. The IV bag will be labeled as "VRC01 or Control in Normal Saline Total Volume = 150 mL". The weight used for calculating the dose should be written on the label. A bag cover will be placed over the bag and should not be removed by the clinic staff. The IV bag will be labeled with a DO NOT INFUSE after date and time as follows:

- o 24 hours if stored at 2°C to 8°C
- 8 hours, including completion of infusion, if stored at controlled room temperature (not to exceed 30°C)

Product may NOT be stored in direct sunlight.

Note: Site pharmacists must follow their institutional policies for expiration dates (ie, DO NOT INFUSE after date and time), if shorter than timeframes above.

#### 6.4 Administration

#### **VRC01** or Control (Intravenously)

Prior to infusion, if the VRC01 or Control IV bag has been stored at 2°C to 8°C, the bag must be equilibrated to room temperature (maximum of 30°C) for 30 minutes or longer and may be held for up to 8 hours, including equilibration time and completion of product administration. (NOTE: This 8 hour period may NOT exceed the DO NOT INFUSE after date and time on the IV bag label.)

The IV bag prepared by the pharmacy will include the weight that was used for preparation of the IV bag (VRC01 or Control). The clinician responsible for administration will check the bag label and confirm that the participant identifier is correct and that the weight on the bag label is within 10% of the participant's current actual weight (see Section 6.3 for more information).

An in-line filter infusion set must be used for IV administration (see SSP for specifications and additional details).

The entire contents of the investigational study product solution will typically be administered IV over about 15 to 60 minutes using a volumetric pump. The total time needed to administer the dose may be longer based on factors such as participant tolerance.

#### 6.5 Acquisition of study products

VRC-HIVMAB060-00-AB is provided by the VRC/DAIDS/NIAID.

Control for VRC01 (Sodium Chloride for Injection USP, 0.9%) will not be provided through the protocol and must be obtained by the site.

Once a CRS is protocol registered, the pharmacist can obtain study products from the CRPMC by following the ordering procedures given in Pharmacy Guidelines and Instructions for DAIDS Clinical Trials Networks.

## 6.6 Pharmacy records

The CRS pharmacist is required to maintain complete records of all study products. The pharmacist of record is responsible for maintaining randomization codes and randomization confirmation notices for each participant in a secure manner.

## 6.7 Final disposition of study products

All unused study products must be returned to the CRPMC after the study is completed or terminated unless otherwise instructed by the CRPMC. The procedures and relevant form are included in the Pharmacy Guidelines and Instructions for DAIDS Clinical Trials Networks.

# 7 Clinical procedures

The schedules of clinical procedures are shown in Appendix J through Appendix M.

#### 7.1 Informed consent

Informed consent is the process of working with participants so that they fully understand what will and may happen to them while participating in a research study. The informed consent form documents that a participant (1) has been informed about the potential risks, benefits, and alternatives to participation, and (2) is willing to participate in this study. Informed consent encompasses all written or verbal study information CRS staff provide to the participant, before and during the trial. CRS staff will obtain informed consent of participants according to HVTN and HPTN policies and procedures.

The informed consent process continues throughout the study. Key study concepts should be reviewed periodically with the participant and the review should be documented. At each study visit, CRS staff should consider reviewing the procedures and requirements for that visit and for the remaining visits. Additionally, if any new information is learned that might affect the participants' decisions to stay in the trial, this information will be shared with trial participants. If necessary, participants will be asked to sign revised informed consent forms.

A CRS may employ recruitment efforts prior to the participant consenting. For example, some CRSs use a telephone script to prescreen people before they come to the clinic for a full screening visit. Participants must sign a screening or protocol-specific consent before any procedures are performed to determine eligibility. CRSs must submit recruitment and prescreening materials to their Institutional Review Board/Ethics Committee (IRB/EC) and any applicable Regulatory Entity (RE) for human subjects protection review and approval.

Note: As defined in the DAIDS Protocol Registration Manual, an RE is "Any group other than the local IRB/EC responsible for reviewing and/or approving a clinical research protocol and site-specific ICFs [informed consent forms] prior to implementation at a site." CRSs are responsible for knowing the requirements of their applicable REs.

## 7.1.1 Screening consent form

Without a general screening consent, screening for a specific study cannot take place until the site receives protocol registration from the DAIDS RSC Protocol Registration Office.

Some CRSs have approval from their IRB/EC and any applicable RE to use a general screening consent form that allows screening for an unspecified HIV prevention trial. In this way, CRS staff can continually screen potential

participants and, when needed, proceed quickly to obtain protocol-specific enrollment consent. Sites conducting general screening or prescreening approved by their IRB/EC and any applicable RE may use the results from this screening to determine eligibility for this protocol, provided the tests are conducted within the time period specified in the eligibility criteria.

#### 7.1.2 Protocol-specific consent forms

The protocol-specific consent forms describe the study products to be used and all aspects of protocol participation, including screening and enrollment procedures. A sample protocol-specific consent form for the main study is located in Appendix A. A separate sample consent form for other uses of specimens is located in Appendix C.

Each CRS is responsible for developing a protocol-specific consent form(s) for local use, based on the sample protocol-specific consent forms in Appendix A and Appendix C. The consent form(s) must be developed in accordance with requirements of the following:

- CRS's IRB/EC, and any applicable RE
- CRS's institution, and
- Elements of informed consent as described in Title 45, CFR Part 46 and Title 21 CFR, Part 50, and in the International Conference on Harmonisation (ICH) E6, Good Clinical Practice: Consolidated Guidance 4.8.

Study sites are strongly encouraged to have their local CABs review their sitespecific consent forms. This review should include, but should not be limited to, issues of cultural competence, local language considerations, and the level of understandability.

The sample informed consent form includes instructions throughout the document for developing specific content.

Sites should follow the instructions in the Protocol-specific Official Memo distributed along with this protocol regarding when they may begin using their site-specific protocol consent forms.

Regarding protocol registration, sites should follow procedures outlined in the current version of the DAIDS Protocol Registration Manual.

#### 7.1.3 Assessment of Understanding

Study staff are responsible for ensuring that participants fully understand the study before enrolling them. This process involves reviewing the informed consent form with the participant, allowing time for the participant to reflect on the procedures and issues presented, and answering all questions completely.

An Assessment of Understanding is used to document the participant's understanding of key concepts in this clinical trial. The participant must complete the Assessment of Understanding before enrollment. Staff may provide assistance in reading and understanding the questions and responses, if necessary. Participants must verbalize understanding of all questions answered incorrectly. This process and the participant's understanding of the key concepts should be recorded in source documentation at the site.

IRB/EC and any applicable RE may require that a participant has signed either a screening or protocol-specific consent document prior to administering the Assessment of Understanding. The consent process (including the use of the Assessment of Understanding) should be explained thoroughly to the IRB/EC and any applicable RE, whose recommendations should be followed.

#### 7.2 Pre-enrollment procedures

Screening may occur over the course of several contacts/visits, up to and including before infusion on Day 0. All inclusion and exclusion criteria must be assessed within 56 days before enrollment, with the exception of HIV testing, which must be performed within 30 days before enrollment (see Section 5.1), unless otherwise specified in the eligibility criteria (or below in this section).

After the appropriate informed consent has been obtained and before enrollment, the following procedures are performed:

- Medical history, documented in the case history record;
- Complete physical examination, including height, weight, vital signs, and clinical assessments of head, ears, eyes, nose, and throat; neck; lymph nodes; heart; chest; abdomen; extremities; neurological function; and skin;
- Assessment of concomitant medications the volunteer is taking, including
  prescription and nonprescription drugs, vitamins, topical products,
  alternative/complementary medicines (eg, herbal and health food
  supplements), recreational drugs, vaccinations, and allergy shots;
- Laboratory tests as defined in the inclusion and exclusion criteria, including:
  - Screening HIV testing at local lab (see SSP)
  - CBC with differential
  - ALT
  - Creatinine
  - Urine dipstick
  - Urine or serum pregnancy test (volunteers capable of becoming pregnant);
     Persons who are not capable of becoming pregnant due to having

undergone total hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing;

- Assessment of participant risk for HIV infection
- Obtaining of volunteer demographics in compliance with the NIH Policy on Reporting Race and Ethnicity Data: Subjects in Clinical Research, Aug. 8, 2001 (available at http://grants.nih.gov/grants/guide/notice-files/NOT-OD-01-053.html);
- Counseling on HIV testing and risk reduction, performed in compliance with US CDC current guidelines or other local guidelines for HIV counseling, testing, and referral as described in Section 7.5; and
- Discussion of pregnancy prevention. A pregnant or breastfeeding person may
  not be enrolled in this trial. Specific criteria and assessment of contraception
  and pregnancy status are described in the study inclusion criteria and in
  Appendix B. Discussion of pregnancy prevention includes advising a
  participant who reports no current sexual activity that could lead to pregnancy
  to have a plan to begin adequate birth control. This plan would be put to use
  if, during the study, the participant becomes sexually active in a way that
  could lead to that participant becoming pregnant.

## 7.2.1 Use of screening results from another HVTN or HPTN study

If a participant screens for an HVTN or HPTN study at the same CRS but then does not join that study, screening results from that effort may be applied to the screening for this protocol, as long as the screening was done under participant consent, the participant has signed a consent form to begin screening for this study, and the tests were conducted within the time periods specified in the eligibility criteria (see Section 5).

#### 7.3 Enrollment and infusion visits

Enrollment is simultaneous with first infusion. The time interval between randomization and enrollment should not exceed 4 working days. The CRS requests the randomization assignment from the Web-based randomization system. Circumstances may require a participant's enrollment visit to be changed. This may exceed the 4-day randomization time limit.

At all infusion visits, the following procedures are performed before infusion:

 Abbreviated physical examination, including weight, vital signs, and a symptom-directed evaluation by history and/or appropriate physical exam based on participant self-reported symptoms or complaints (see SSP for more detail);

- Assessment of baseline reactogenicity parameters;
- Assessment of any new or unresolved AEs/intercurrent illnesses;
- Assessment of concomitant medications (as described in Section 7.2);
- ALT;
- Creatinine;
- CBC with differential;
- Urine or serum pregnancy test (for participants who are capable of becoming pregnant). Persons who are NOT capable of becoming pregnant due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing; and
- Blood collection for HIV testing and sample storage.

Following completion of all procedures in the preceding list, and if results indicate that infusion may proceed, infusion is administered (see Sections 6.3 and 6.4).

Administration of an infusion and infusion-related procedures must be accomplished within 1 calendar day.

Immediately following the first infusion, the participant remains in the clinic for observation and initial reactogenicity assessment. See the SSP for details regarding infusion visit procedures and subsequent infusion observation and reactogenicity assessment procedures that CRSs must follow. The site will make arrangements to obtain a report of reactogenicity events from the participant after the 3-day reactogenicity period (as described in Section 7.10 and in the SSP).

The following procedures will be performed at all infusion visits. These procedures may be performed prior to, during, or following infusion:

- Administration of the participant questionnaire which may include acceptability, behavioral risk, study product belief, motivations, and social impact domains (must be done prior to risk reduction counseling);
- HIV infection assessment including pre-test counseling. A subsequent followup contact is conducted to provide post-test counseling and to report results to participant;
- Risk reduction counseling (as described in Section 7.5);
- Pregnancy prevention assessment (as described in Section 7.2 and 7.6);

- Assessment of new or unresolved social impacts (site staff will ask participant about the status of any unresolved social impacts and if s/he has experienced any new social impacts as a result of the trial participation);
- Confirm that participants received HIV test results from previous visit. If not, provide test results and post-test counseling as appropriate; and
- Ship samples to HVTN Central Laboratory for HIV diagnostic testing.

Additional procedures will be performed at scheduled visits as specified in Appendix J:

- Syphilis serology testing,
- Gonorrhea (GC)/chlamydia (CT) testing by urine or cervical/vaginal swab,
- Trichomonas by cervical/vaginal swab, and
- Urine dipstick (see Section 7.9).

## 7.4 Post-infusion visits for HIV-uninfected study participants

The following procedures are performed at all post-infusion follow-up visits for HIV-uninfected study participants:

- HIV infection assessment including pre-test counseling. A subsequent followup contact is conducted to provide post-test counseling and to report results to participant;
- Confirm that participants received HIV test results from previous visit. If not, provide test results and post-test counseling as appropriate;
- Blood collection for HIV testing and sample storage; and
- Ship samples to HVTN Central Laboratory for HIV diagnostic testing.

Additional procedures will be performed at scheduled follow-up visits as specified in Appendix F and Appendix J:

- Assessment of new or unresolved social impacts (site staff will ask participant about the status of any unresolved social impacts and if s/he has experienced any new social impacts as a result of the trial participation);
- Administration of participant questionnaire, which may include acceptability, behavioral risk, study product belief, motivations, and social impact domains (must be done prior to risk reduction counseling)

- Risk reduction counseling (as described in Section 7.5);
- Urine or serum pregnancy test (for participants who are capable of becoming pregnant). Persons who are NOT capable of becoming pregnant due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing;
- Pregnancy prevention assessment (as described in Section 7.2 and 7.8);
- Assessment of new or unresolved AEs/intercurrent illnesses;
- Urine dipstick (see Section 7.9); and
- Complete physical examination, including weight, vital signs, and clinical assessments of head, ears, eyes, nose, and throat; neck; lymph nodes; heart; chest; abdomen; extremities; neurological function; and skin.

#### 7.5 HIV counseling and testing

HIV counseling will be performed in compliance with the CDC's guidelines or other local guidelines for HIV counseling and referral. HIV testing will be performed in accordance with the protocol-specific HIV testing algorithm following enrollment.

Participants will be counseled routinely during the trial on the avoidance of HIV infection. In addition, study participants will be provided with HIV prevention supplies and referral to providers of PrEP per local and regional guidelines. Study investigators will ensure that participants have access to standards of care for HIV prevention in their local settings. As new data emerge and standards of care for HIV prevention evolve, both the content of risk reduction counseling and referrals for biomedical interventions will be updated to conform to current best practices for the population enrolled in this trial.

## 7.5.1 Study product-related seroreactivity

Human sera containing purified VRC01 at concentrations up to 1600 mcg/mL have been tested using a variety of commercially available HIV test kits without any indication of reactivity. For this reason, we do not anticipate that receipt of VRC01 will cause a reactive result on currently available HIV test kits, but this remains a theoretical possibility.

Because this possibility cannot be categorically eliminated, study staff will advise study participants to confine their HIV testing while in the study to that provided through the CRS. Staff will also inform study participants of the likelihood of routine HIV testing being offered or performed outside the study CRS at emergency rooms, clinics, and medical offices and will inform participants of their right to opt out of HIV testing outside the study site. CRS staff should

inform study participants if local and/or state/regional policies and regulations permit medical providers to perform HIV testing without first informing patients. If this is the case, then CRS staff should advise study participants that they may decline HIV testing preemptively. CRS staff should also inform participants if positive HIV test results must be reported to local public health authorities. CRS staff should also inform participants of the need to maintain study blinding by getting HIV testing only at the study CRS. CRS staff should provide participants with CRS contact information and should encourage participants to ask medical providers to contact the CRS. The CRS can verify that the participant is in an HIV mAb clinical trial and should only be tested for HIV at the study CRS.

Study staff should also stress that the study product is completely cleared from the body within a few months, so even the theoretical risk of VRC01 causing a misleading HIV test result will disappear before their final scheduled clinic visit.

#### 7.6 Follow-up visits for HIV-infected participants

The following procedures are performed at scheduled follow-up visits as specified in Appendix G, Appendix H, Appendix K, and Appendix L:

- Counseling on HIV testing and diagnosis;
- Abbreviated physical exam including weight, vital signs, and a symptomdirected evaluation by history and/or appropriate physical exam based on participant self-reported symptoms or complaints (see SSP for more detail);
- ART assessment;
- Assessment of concomitant medications (as described in Section 7.2);
- Assessment of any new or unresolved AEs/intercurrent illnesses;
- HIV transmission risk reduction counseling;
- Behavioral risk assessment questionnaire;
- Assessment of new or unresolved social impacts (site staff will ask participant about the status of any unresolved social impacts and if s/he has experienced any new social impacts as a result of the trial participation);
- Blood collection for HIV testing, viral load testing, VRC01 Ab levels, functional assays, viral isolation/sequencing, and sample storage (see Appendix G and Appendix H);
- Blood collection for CD4+ T cell counts;

- Urine or serum pregnancy test (for participants who are capable of becoming pregnant). Persons who are NOT capable of becoming pregnant due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing; and
- Complete physical examination, including weight, vital signs, and clinical assessments of head, ears, eyes, nose, and throat; neck; lymph nodes; heart; chest; abdomen; extremities; neurological function; and skin.

# 7.7 Follow-up visits for participants who discontinue infusions for reasons other than HIV infection

Participants for whom infusions are discontinued for reasons other than HIV infection should be encouraged to continue in the study. For such participants, the following procedures are performed at approximately quarterly scheduled follow-up visits as specified in Appendix I and Appendix M:

- Abbreviated physical exam including weight, vital signs, and a symptomdirected evaluation by history and/or appropriate physical exam based on participant self-reported symptoms or complaints (see SSP for more detail);
- Risk reduction counseling (as described in Section 7.5);
- Assessment of concomitant medications (as described in Section 7.2);
- Assessment of any new or unresolved AEs/intercurrent illnesses;
- HIV infection assessment including pre-test counseling. A subsequent followup contact is conducted to provide post-test counseling and to report results to participant;
- Confirm that participants received HIV test results from previous visit. If not, provide test results and post-test counseling as appropriate;
- Behavioral risk assessment questionnaire;
- Assessment of new or unresolved social impacts (site staff will ask participant about the status of any unresolved social impacts and if s/he has experienced any new social impacts as a result of the trial participation);
- Blood collection for HIV testing, CBC/differential, ALT, creatinine, VRC01
   Ab levels, functional assays, and sample storage (see Appendix I and
   Appendix M);
- Urine dipstick (see Section 7.9);

- Urine or serum pregnancy test (for participants who are capable of becoming pregnant). Persons who are NOT capable of becoming pregnant due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing; and
- Complete physical examination, including weight, vital signs, and clinical assessments of head, ears, eyes, nose, and throat; neck; lymph nodes; heart; chest; abdomen; extremities; neurological function; and skin.

## 7.8 Contraception status

Contraception status is assessed and documented at screening and infusion visits for a participant who is capable of becoming pregnant. Prior to enrollment and throughout the study, staff will ask participants to verbally confirm their use of adequate contraceptive methods. These participants should be reminded regularly of the importance of using contraception and should be referred to specific counseling, information, and advice as needed (see Appendix B for further detail.) This reminder should be documented in the participant's study record.

Infertility—including having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation—must be documented in the participant's study record.

## 7.9 Urine testing

Urine dipstick testing may be performed in the clinic or the lab. The following analytes should be analyzed and recorded: specific gravity, protein, blood/hemoglobin, pH, urobilinogen, bilirubin, ketone, leucocyte esterase, nitrite, and glucose. The examination is performed on urine obtained by clean catch. Urine microscopy is required when the protein result is 1+, 2+, 3+, or 4+ (or semi-quantitative 30, 100, 300, or 2000 g/L) and/or the blood/hemoglobin result is trace, 1+, 2+, 3+, or 4+, but not required (unless otherwise clinically indicated) if the dipstick result is abnormal due to non-urinary bleeding.

If the dipstick performed for screening is transiently abnormal with an exclusionary result (eg, 2+ proteinuria), then repeat the dipstick and, if within the eligibility limits specified in the protocol, the participant may be enrolled (see SSP for further detail).

A follow-up urine test should be deferred if a participant is experiencing non-urinary bleeding (eg, menstruation), but should be performed as soon as possible. If a follow-up dipstick is abnormal due to non-urinary bleeding (eg, a participant's menstrual period), document in the comment section of the CRF and repeat the dipstick once the participant is no longer experiencing non-urinary bleeding. In this case, a urine microscopy is not required (see SSP for further

detail). If a follow-up dipstick is abnormal due to infection, document this issue in the participant's chart and provide appropriate treatment and/or referral.

## 7.10 Assessments of reactogenicity

For all participants, baseline assessments are performed before and reactogenicity assessments are performed after each infusion per the SSP. All reactogenicity symptoms are graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017, except as noted in Section 10.2.2.

The reactogenicity assessment period is 3 full days following each infusion. The site staff and the participant will be in contact after the 3-day reactogenicity period, or sooner if indicated. At that time, site staff will discuss reactogenicity events with the participant and record the relevant information on either the appropriate CRF(s) or participant chart note as source (for more details, see the SSP). Clinic staff will follow new or unresolved reactogenicity symptoms present at day 3 to resolution. Participants are instructed to contact the clinic for events that arise during the period between infusion and the next scheduled visit. In general, a participant who self-reports any postinfusion reaction greater than mild is seen by a clinician within 48 hours after onset, unless the reaction is improving and/or has completely resolved.

Reactogenicity assessments include assessments of specific systemic and local signs and symptoms and IV infusion-related site reactions. Events not listed on a CRF, or with an onset after the reactogenicity assessment period (day of infusion and 3 full days after), or those meeting SAE/adverse events requiring expedited reporting to DAIDS criteria, are recorded on an adverse event log form.

For more detailed information and instructions on reactogenicity assessments, see the SSP.

## 7.10.1 Assessment of systemic and local signs and symptoms

Systemic signs and symptoms include increased body temperature, malaise and/or fatigue, myalgia, headache, chills, arthralgia, nausea, and vomiting. Local symptoms include pain and/or tenderness proximal to the infusion site. The maximum severity reached for each symptom during the assessment period per the SSP is reported.

#### 7.10.2 Assessment of infusion site

IV infusion-related site reactions may include redness/erythema and induration/swelling. The maximum horizontal and maximum vertical measurements for IV infusion-related site redness/erythema and induration/swelling are recorded.

All infusion site reactions are monitored until resolution. Areas greater than 25 cm<sup>2</sup> are followed daily; otherwise, the frequency of follow-up is based on clinician judgment.

#### 7.11 Visit windows and missed visits

Visit windows are defined in the SSP. For a visit not performed within the window period, a Missed Visit form is completed.

If a participant misses a scheduled visit, CRS staff should attempt to bring the participant in as soon as possible to complete the required safety assessments and other procedures. See the SSP for more details. If a participant missed an infusion visit or if infusions must be permanently discontinued, see Section 5.3.2 and Section 5.3.3 for resolution.

## 7.12 Early termination visit

In the event of early participant termination, site staff should consider if the following assessments are appropriate: a final physical examination, clinical laboratory tests (including urine dipstick, CBC with differential, ALT, and Creatinine), pregnancy testing, social impact assessment, and HIV test.

## 7.13 Pregnancy

If a participant becomes pregnant during the course of the study, no more infusions of study product will be given during the pregnancy, but remaining visits and study procedures should be completed unless medically contraindicated. For participants who are no longer pregnant, see Section 5.3.1. If the participant terminates from the study prior to the pregnancy outcome, the site should make every effort to keep in touch with the participant in order to ascertain the pregnancy outcome.

# 8 HIV infection assessment and clinical response

## 8.1 HIV symptom assessment

At all scheduled visits and at unscheduled visits due to illness or suspected exposure, if necessary, information will be collected about any signs or symptoms suggestive of acute HIV infection. Participants will be counseled about signs and symptoms of acute HIV infection and at visits following recent high-risk exposure, participants will be queried about any signs/symptoms suggestive of acute HIV infection. Presence of signs/symptoms suggestive of acute HIV infection, an intercurrent illness consistent with acute retroviral syndrome, or history of high-risk exposure would prompt a diagnostic work-up per the protocol-specific algorithm for recent exposure to determine HIV infection.

#### 8.2 HIV screening test (prior to randomization)

Prior to randomization, participants will be screened for HIV-1/2 infection by FDA-approved blood tests (non-US sites may use locally available assays that have been approved by HVTN and HPTN Laboratory Operations [see SSP]). Volunteers identified as being HIV infected during screening will be referred for medical treatment and management of the HIV infection. These individuals may also be referred to appropriate ongoing clinical trials or observational studies. For volunteers who have one or more reactive/positive HIV tests, but whose HIV status is inconclusive, any further testing will be performed locally.

## 8.3 HIV testing postinfusion

Following enrollment, HIV testing will take place at scheduled clinic visits (Appendix F).

HIV testing will be performed using the protocol-specific HIV testing algorithms (see SSP). At scheduled visits that include HIV testing, specimens will be tested with an FDA-approved 4<sup>th</sup> generation HIV 1/2 enzyme immunoassay (EIA) or chemiluminescent microparticle immunoassay (CMIA). If the participant has a reactive test result, an HIV RNA test and an HIV 1/2 discriminatory test will be performed as indicated in the algorithm. Further HIV testing is required using a second specimen drawn on a later date to confirm a diagnosis of HIV infection. The second specimen may be collected at an interim visit (ie, visit #.X specified in Appendix G and Appendix H). Samples to be stored for future studies will also be collected at this time (see Appendix G).

A 'case' will be defined as a participant who is confirmed to have acquired HIV-1 infection after enrollment based on the protocol-specific diagnostic algorithms (see SSP). Before informing a participant that they are infected at or after

enrollment, all HIV test results will be reviewed by a blinded, independent Endpoint Adjudicator(s) or designee(s) (Section 8.4).

The HVTN Laboratory Program is responsible for all in-study diagnostic testing.

## 8.4 Endpoint adjudication

The general diagnostic criteria for HIV infection are well accepted. However, definitive diagnosis of HIV infection in the context of having received a study product that is even partially effective may be more difficult. Specifically, if VRC01 is capable of completely suppressing viral replication, or if the antibody alters the normal serological response upon exposure to HIV, standard diagnostic tests may be more difficult to assess. Therefore, this study will have an endpoint adjudication process to review all serological and virological test results in a blinded manner for each participant who tests positive per the HVTN 703/HPTN 081 HIV diagnostic testing algorithms. Adjudicators will also review HIV test results in cases where HIV infection status is not clearly resolved using the HIV testing algorithm. The assessment of the Endpoint Adjudicator(s) or designee(s) will be reported to the SDMC and to the HIV diagnostics laboratory.

The Endpoint Adjudicator(s) or designee(s) must notify the SDMC within 1 working day of any confirmed HIV infection. The HIV diagnostics lab will inform the clinic of the outcome of the HIV testing algorithm (ie, HIV-infected, HIV-uninfected, or redraw required).

The Endpoint Adjudicator(s) or designee(s) will be expert in the fields of infectious diseases or laboratory medicine independent of the VRC and clinical investigators participating in this trial. A separate Standard Operating Procedure will govern the activities of the Endpoint Adjudicator(s) or designee(s).

## 8.5 HIV infection during the study

It is critical to the success of the study that HIV-infected participants be properly identified and all data postdiagnosis be carefully recorded. Information obtained from these cases of HIV-1 infection will form the basis of the primary endpoint assessment.

Participants who develop HIV infection following the initial infusion of study product may remain in the study for follow-up but will receive no further infusions. This includes participants for whom infusions were discontinued for reasons other than HIV infection but for whom HIV-1 infection has subsequently been confirmed, All participants who become HIV-1—infected following enrollment through their final study visit will be monitored as indicated in Appendix G and Appendix K.

If a participant is confirmed to have become HIV infected after enrollment, plasma HIV-1 RNA will be measured on archived samples prior to the first positive screening test. HIV-1 RNA testing will also be performed at 2-week intervals up to 8 weeks postdiagnosis, then at 12 and 24 weeks postdiagnosis. In addition to plasma HIV-1 RNA testing, participants will also have specimens drawn for measurements of VRC01 Ab serum levels, neutralization and other antibody functions, viral isolation and sequencing; physical exams, recording of AEs, counseling to reduce HIV transmission risk, and social impact assessments will also be performed at most of these visits.

Longer-term follow-up for these participants may be accomplished through enrollment in another protocol. Archived samples from earlier visits may also be tested to determine the earliest date of HIV infection.

If enrollment visit HIV testing indicates that a participant was HIV infected at enrollment (ie, prior to the first infusion of study product) or a participant is diagnosed with HIV-2 infection following enrollment, then the procedures indicated in the preceding paragraph do not apply. Such participants should be followed as indicated in Appendix H and Appendix L. This also applies to participants for whom infusions are discontinued for reasons other than HIV infection and who subsequently are diagnosed with HIV-2 infection.

## 8.6 Medical care for participants who become HIV infected

It is anticipated that some study participants, whether they are randomized to receive VRC01 or control, will become HIV infected during the course of the trial. It is critical that these HIV-infected participants receive appropriate medical care.

The investigators associated with this trial will refer participants who develop HIV infection while participating in this trial to medical professionals for care.

# 9 Laboratory

#### 9.1 CRS laboratory procedures

The SSP provides further guidelines for operational issues concerning the clinical and processing laboratories. This document includes guidelines for general specimen collection, special considerations for phlebotomy, specimen labeling, whole blood processing, HIV screening/diagnostic testing, and general screening and safety testing.

Tube types for blood collection are specified in Appendix F through Appendix I. For tests performed locally, the local lab may assign appropriate tube types.

In specific situations, the blood collection tubes may be redirected to another laboratory or may require study-specific processing techniques. In these cases, laboratory special instructions will be posted on the protocol-specific section of the HVTN website.

#### 9.2 Total blood volume

Required blood volumes per visit are shown in Appendix F through Appendix I. Not shown is any additional blood volume that would be required if a safety lab needs to be repeated, or if a serum pregnancy test needs to be performed. The additional blood volume would likely be minimal. The total blood volume drawn for each participant will not exceed 500 mL in any 56-day (8-week) period.

#### 9.3 Assay timepoints

Endpoint assays are performed on participants at the timepoints shown in Appendix F through Appendix I may be performed at baseline. Assays for humoral and cellular responses may be performed on participants or a subset of participants at other timepoints; the schedules are shown in Appendix F through Appendix I.

#### 9.4 VRC01 mAb levels

VRC01 levels will be measured in serum. An ELISA will be used to determine the concentration of the VRC01 antibody in the serum. The ELISA employs the VRC01 Fab-specific 5C9 mAb, which is an anti-idiotype antibody cloned from a single B cell that was sorted by flow cytometry using a VRC01 scFv probe. The 4-parameter logistic curve regression of a standard curve of VRC01 covering the range from 0.031 to 1.0 mcg/mL is utilized in this assay to quantitate the sample concentrations based upon the average of sample dilutions within the range of the assay. This assay has been qualified but not formally validated. The functional

sensitivity for the generation of the ELISA assay format, which is currently used at NVITAL, is 2 mcg/mL and as the technology for this assay continues to develop, an updated assay may be utilized.

#### 9.5 Endpoint assays: humoral

## 9.5.1 Anti-VRC01 antibody assay

Assessment for development of anti-VRC01 antibodies in participants will be performed using the Meso Scale Discovery (MSD) platform based on electrochemiluminescence. The assay uses biotin-labeled VRC01 immobilized on a streptavidin-coated MSD plate as the capture molecule, and the SULFO-TAG labeled VRC01 as the reporter molecule. This assay is independent of the anti-VRC01 antibody isotype, and permits the detection of both high and low affinity antibodies.

## 9.5.2 Neutralizing antibody assay

Depending upon the VRC01 concentrations measured in collected specimens, their capacity to neutralize HIV in blood and mucosal secretions may be evaluated by an in vitro cell-based virus neutralization assay [129-131] using pseudotyped viruses. All specimens testing positive for anti-VRC01 antibodies will be tested for HIV-1 neutralizing activity.

One or more viruses that are among the most sensitive to VRC01 (eg, MN.3 and MW965.26) will be assayed. The IC<sub>50</sub> of VRC01 against both of these viruses is 0.01 - 0.03 mcg/ml and the TZM-bl assay is validated for this level of sensitivity.

#### 9.6 ARV detection

A direct, biomedical measure is used to assess ARV use in this study. This approach is used because self-report of ARV use for PrEP or PEP and other purposes has been shown to be unreliable in a variety of settings [82,132,133]. For this study, ARV testing will be performed using a test that measures the amount of tenofovir-diphosphate (a metabolite of tenofovir) in red blood cells. This test utilizes a dried blood spot as the sample source and analyzes for tenofovir diphosphate by liquid chromatography and tandem mass-spectroscopy, as previously described [134,135]. Because of a long half-life, high amounts of the metabolite in the dried blood spot correspond with consistent dosing of Truvada and low amounts correspond with inconsistent dosing [75]. Samples are collected and stored on regularly scheduled calendar days throughout the study and testing will be performed periodically on batched samples. In addition, both serum and plasma samples are collected from all participants at all timepoints. This will allow additional assessment of PrEP use by selected participants if warranted by the results of the dried blood spot assay. Individual test results will not be returned to study sites or study participants.

#### 9.7 Host (human) genotyping

Various markers, such as genes associated with host immune functions or HIV disease progression may also be assessed.

#### 9.8 Lab assay algorithm

The HVTN Lab Assay Algorithm lists assays that characterize various types of immunologic activity as well as host genetics that may be conducted to characterize the drug activity in this study. Various types of assays may be employed to assess maintenance of functional drug activity at multiple timepoints selected based on drug level outcomes. Please note that the Lab Assay Algorithm will be updated periodically to include new assays.

#### 9.9 Possible additional studies

Samples may be used for other testing and research related to furthering the understanding of HIV immunology, monoclonal antibodies, or vaccines. In addition, cryopreserved samples may be used to perform additional assays to support standardization and validation of existing or newly developed methods.

## 9.10 Other use of stored specimens

The Networks store specimens from all study participants indefinitely, unless a participant requests that specimens be destroyed or if required by IRB/EC or RE.

Other use of specimens is defined as studies not described in the protocol.

This research may relate to HIV, vaccines, monoclonal antibodies, the immune system, and other diseases. This could include limited genetic testing and, potentially, genome-wide studies. This research is done only to the extent authorized in each study site's informed consent form, or as otherwise authorized under applicable law. Other testing on specimens will occur only after review and approval by the HVTN, the HPTN, the IRB/EC of the researcher requesting the specimens, and the CRS's IRBs/ECs if required.

The protocol sample informed consent form is written so that the participant either explicitly allows or does not allow their samples to be used in other research when they sign the form. Participants who initially agree to other use of their samples may rescind their approval once they enter the study; such participants will remain in this study and their samples will only be used for the studies described in this protocol. If a participant decides against allowing other research using his or her samples, or at any time rescinds prior approval for such other use, the study site investigator or designee must notify HVTN Regulatory

Affairs in writing. In either case, HVTN Regulatory Affairs directs the HVTN Lab Program not to use samples from these participants for such other uses.

CRSs must notify HVTN Regulatory Affairs if institutional or local governmental requirements pose a conflict with or impose restrictions on other use of specimens.

#### 9.11 Biohazard containment

As the transmission of HIV and other blood-borne pathogens can occur through contact with contaminated needles, blood, and blood products, appropriate precautions will be employed by all personnel in the drawing of blood and shipping and handling of all specimens for this study, as currently recommended by the CDC and the NIH or other applicable agencies.

All dangerous goods materials, including Biological Substances, Category A or Category B, must be transported according to instructions detailed in the International Air Transport Association Dangerous Goods Regulations.

# 10 Safety monitoring and safety review

## 10.1 Safety monitoring and oversight

#### 10.1.1 HVTN 703/HPTN 081 PSRT

The HVTN 703/HPTN 081 PSRT is composed of the following members:

- DAIDS medical officer representatives,
- Protocol chairs and cochairs,
- Protocol Team leader,
- Core medical monitor,
- Clinical safety specialist (CSS), and
- Regional medical liaison (RML).

A medical officer from an organization(s) designated by the study sponsor will also participate in the PSRT.

The clinician members of HVTN 703/HPTN 081 PSRT are responsible for decisions related to participant safety.

The Protocol Team clinic coordinators, project managers, study product developer representatives, clinical research manager, clinical trial manager, and others may also be included in HVTN 703/HPTN 081 PSRT meetings.

#### **10.1.2 NIAID DSMB**

The NIAID DSMB assesses the effects of the study product during the trial, provides other monitoring as described in Section 4.7.1.1, and may give advice to the HVTN 703/HPTN 081 OC.

## 10.1.3 Roles and responsibilities in safety monitoring

The roles and responsibilities of the SDMC in relation to safety monitoring include:

- Maintaining a central database management system for clinical data;
- Providing reports of clinical data to appropriate groups such as the HVTN 703/HPTN 081 PSRT and NIAID DSMB.
The roles and responsibilities of the HVTN CSS or HVTN Core designee in relation to safety monitoring include:

- Daily monitoring of clinical data for events that meet the safety pause and HVTN 703/HPTN 081 PSRT AE review criteria (see Section 10.3);
- Notifying CRSs and other groups when safety pauses are instituted and lifted (see Section 10.3);
- Querying CRSs for additional information regarding reported clinical data; and
- Providing support to the HVTN 703/HPTN 081 PSRT.

#### 10.2 Safety reporting

# 10.2.1 Submission of safety forms to SDMC

Sites must submit all safety forms (eg, reactogenicity, adverse experience, urinalysis, local lab results, concomitant medications) before the end of the next business day after receiving the information. The forms should not be held in anticipation of additional information at a later date. If additional information is received at a later date, the forms should be updated and resubmitted before the end of the next business day after receiving the new information.

# 10.2.2 AE reporting

An AE is any untoward medical occurrence in a clinical investigation subject administered a study product/procedure(s) and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational study product/procedure(s), whether or not related to the investigational study product/procedure(s). The AE reporting period for this study comprises the entire study period for each individual participant (from study enrollment until study completion or discontinuation of the study). All AEs are graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1. dated July 2017, available on the RSC website at http://rsc.tech-res.com/clinical-research-sites/safety-reporting/daids-grading-tables, except that the AEs below will be reported according to the SSP:

- Unintentional weight loss
- Infusion Site Erythema or Redness and Infusion Site Induration or Swelling
- Infusion reactions

#### • Uterine bleeding secondary to contraception

As detailed in the SSP, two additional parameters, cytokine release syndrome and serum sickness, have been added to the DAIDS AE Grading Table for HVTN 703/HPTN 081.

AEs are reported to the SDMC on the appropriate CRF. Clinic staff should evaluate every AE to determine if (1) the AE meets the requirements for expedited reporting to DAIDS (Section 10.2.3) and (2) if the AE meets the criteria for a safety pause/prompt AE review (Section 10.2.4).

Sites are expected to notify the CSS or RML of any serious safety concern requiring their attention (see Table 10-1). Telephone numbers and email addresses are found on the HVTN703/HPTN 081 protocol-specific website. Concerns requiring immediate attention should be communicated by calling the clinical safety phone.

In the case of email notification, the CSS or RML will reply during working hours (ie, US Pacific Time, South Africa Standard Time, or Central Africa Time) to confirm that the email has been received and reviewed. If email service is not available, the CRS should notify the CSS or RML of the event by telephone, then submit CRFs.

In addition, site investigators are required to submit AE information in accordance with IRB/EC and any applicable RE requirements.

## 10.2.3 Expedited reporting of adverse events to DAIDS

Requirements, definitions and methods for expedited reporting of AEs are outlined in Version 2.0 (January 2010) of the *Manual for Expedited Reporting of Adverse Events* to DAIDS (DAIDS EAE Manual), which is available on the RSC website at http://rsc.tech-res.com/clinical-research-sites/safety-reporting/manual. The SAE Reporting Category will be used for this study.

The internet-based DAIDS Adverse Experience Reporting System (DAERS) must be used for expedited AE reporting to DAIDS. In the event of system outages or technical difficulties, expedited AE reports may be submitted via the DAIDS EAE Form. This form is available on the DAIDS RSC website at http://rsc.techres.com/clinical-research-sites/safety-reporting/daids/paper-eae-reporting

For questions about DAERS, please contact NIAID CRMS Support at CRMSsupport@niaid.nih.gov or from within the DAERS application itself.

For questions about expedited AE reporting, please contact the RSC (DAIDSRSCSafetyOffice@tech-res.com).

Under ICH E2A (*Clinical Safety Data Management: Definitions and Standards for Expedited Reporting*), an SAE is defined as any untoward medical occurrence that at any dose:

- results in death,
- is life-threatening (Note: The term "life-threatening" in the definition of "serious" refers to an event in which the patient was at risk of death at the time of the event; it does not refer to an event, which hypothetically might have caused death, if it were more severe),
- requires patient hospitalization or prolongation of existing hospitalization,
- results in persistent or significant disability/incapacity,
- is a congenital anomaly/birth defect, or
- is a medically important event or reaction.

Medical and scientific judgment should be exercised when deciding if other situations are serious. Such instances could include medical events that may not be immediately life-threatening or result in death or hospitalization, but which may jeopardize the patient or may require intervention to prevent one of the outcomes listed in the definition above. Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias, or convulsions not resulting in hospitalization, or development of drug dependency or drug abuse.

The expedited reporting period for this study comprises the entire study period for each individual participant (from study enrolment until study completion or discontinuation from the study).

The study products for which expedited reporting are required are:

- VRC01, and
- Control.

The NIAID/DAIDS will report all unexpected SAEs related to the study products observed in this clinical trial to the FDA in accordance with 21 CFR 312.32 (IND Safety Reports). However, because safety is a primary study endpoint, the Sponsor Medical Officer will not be unblinded to study treatment assignment when there is an assessment of relatedness of the SAE with the study product(s); and the safety report will be sent to the FDA based on the blinded attribution assessment.

If the PSRT believes unblinding of the site PI to treatment assignment will assist with the clinical management of the SAE, the PSRT may consult the independent

NIAID DSMB for a recommendation. In the event the PSRT and/or the NIAID DSMB determines that unblinding is indicated, the unblinded statistician, DSMB Chair, or designee will inform the site physician of the participant's treatment assignment in such a manner as to maintain the study blind of the PSRT and study team. For additional impact and management of SAEs on the study, refer to Section 10.3.

# 10.2.4 Expedited reporting of AEs to pertinent national regulatory authorities

The study sponsor or designee(s) prepares and files expedited reports to appropriate regulatory authorities within the timelines required by pertinent national regulatory authorities.

Site IoRs/designees will submit AE information and any other relevant safety information to their ECs/IRBs in accordance with EC/IRB requirements.

#### 10.3 Safety pause and prompt PSRT AE review

When a trial is placed on safety pause, all enrollment and infusion with the product related to the event that triggered the pause will be held until further notice. The AEs that will lead to a safety pause or prompt HVTN 703/HPTN 081 PSRT AE review are summarized in Table 10-1. Infusions may be suspended for safety concerns other than those described in the table, or before pause rules are met, if, in the judgment of the HVTN 703/HPTN 081 PSRT, participant safety may be threatened. Criteria for an individual participant's departure from the schedule of infusions are listed in Section 5.3.

| Table 10-1 AE notification and | safety pause/AE review rules |
|--------------------------------|------------------------------|
|--------------------------------|------------------------------|

| Event and relationship to study products | Severity | CRS action <sup>a</sup> | HVTN Core <sup>b</sup> action |
|---|---|---|---|
| SAE, related | Grade 4 or 5 | Phone immediately, email and submit forms immediately | Immediate pause |
| SAE, not related | Grade 5 | Phone immediately, email and submit forms immediately | Immediate HVTN 703/HPTN 081 PSRT notification |
| SAE, related | Grade 3 | E-mail and submit forms immediately | Prompt HVTN 703/HPTN 081<br>PSRT AE review to consider<br>pause |
| AE <sup>c</sup> , related | Grade 4 or 3 | Email and submit forms immediately | Prompt HVTN 703/HPTN 081<br>PSRT AE review to consider<br>pause |

<sup>&</sup>lt;sup>a</sup>Phone numbers and email addresses are found on the Protocol home page on the HVTN Members' site (https://members.hvtn.org/protocols/hvtn703/HPTN081).

For all safety pauses, HVTN Core notifies the HVTN 703/HPTN 081 PSRT, HVTN Regulatory Affairs, DAIDS Pharmaceutical Affairs Branch (PAB), DAIDS Regulatory Affairs Branch (RAB), DAIDS Safety and Pharmacovigilance

<sup>&</sup>lt;sup>b</sup> HVTN CSS or HVTN Core designee

<sup>&</sup>lt;sup>c</sup> Does not include subjective reactogenicity symptoms (injection site pain, tenderness, fatigue/malaise, myalgia, arthralgia, chills, headache, nausea).

Team (SPT), and participating HVTN and HPTN CRSs. When an immediate safety pause is triggered, HVTN Core notifies the NIAID DSMB.

Once a trial is paused, the HVTN 703/HPTN 081 PSRT reviews safety data and decides whether the pause can be lifted or permanent discontinuation of infusions is appropriate, consulting the NIAID DSMB if necessary. HVTN Core notifies the participating HVTN and HPTN CRSs, HVTN Regulatory Affairs, DAIDS PAB, DAIDS RAB, and DAIDS SPT of the decision regarding resumption or discontinuation of study infusions. Based on the HVTN 703/HPTN 081 PSRT assessment, DAIDS RAB notifies the FDA as needed.

If an immediate HVTN 703/HPTN 081 PSRT notification or prompt HVTN 703/HPTN 081 PSRT AE review is triggered, HVTN Core notifies the HVTN 703/HPTN 081 PSRT as soon as possible during working hours (US Pacific Time)—or, if the information was received during off hours, by the morning of the next work day. If a prompt HVTN 703/HPTN 081 PSRT AE review cannot be completed within 72 hours of notification (excluding weekends and US federal holidays), an automatic safety pause occurs.

The HVTN and HPTN require that each CRS submit to its IRB/EC and an applicable RE protocol-related safety information (such as IND safety reports, notification of study product holds due to the pause rules, and notification of other unplanned safety pauses). CRSs must also follow all applicable RE reporting requirements.

In addition, all other AEs are reviewed routinely by the HVTN 703/HPTN 081 PSRT (see Section 10.4.2).

#### 10.4 Review of cumulative safety data

Routine safety review occurs at the start of enrollment and then throughout the study.

Reviews proceed from a standardized set of protocol-specific safety data reports. These reports are produced by the SDMC and include queries to the CRSs. Events are tracked by internal reports until resolution.

#### 10.4.1 Daily review

Blinded daily safety reviews are routinely conducted by HVTN Core for events requiring expedited reporting to DAIDS, and events that meet safety pause criteria or prompt HVTN 703/HPTN 081 PSRT AE review criteria.

#### 10.4.2 Twice monthly review

During the infusion phase of the trial, the HVTN 703/HPTN 081 PSRT reviews clinical safety reports twice each month and conducts calls to review the data as

appropriate. After the infusions and the final postinfusion safety visits are completed, less frequent reporting and safety reviews may be conducted at the discretion of the HVTN 703/HPTN 081 PSRT. The HVTN CSS or HVTN Core designee reviews reports of clinical and laboratory AEs. Events identified during the review that are considered questionable, inconsistent, or unexplained are referred to the CRS clinic coordinator for verification.

# 10.4.3 DSMB review of cumulative safety data

The DSMB will periodically review accumulating safety data. Prior to each such review, the SDMC will provide the DSMB with data as described in Section 4.7.1. Reports will be cumulative, generated from an up-to-date data file. Reports will show the data coded by treatment group; however, upon request of the DSMB, the SDMC will provide the Board with the actual treatment group.

# 10.5 Study termination

This study may be terminated early by NIAID upon recommendation by the DSMB, a pertinent national regulatory authority, Office for Human Research Protections (OHRP), or study product developer. In addition, the conduct of this study at an individual CRS may be terminated by the determination of the IRB/EC and any applicable RE.

# 10.6 Social impact reporting

It is possible that participants' involvement in the study could result in social impacts. For example, a participant's involvement in the study could become known to others, and a social harm may result (ie, because participants could be perceived as being HIV infected or at "high risk" for HIV infection). Participants could be treated unfairly, or could have problems being accepted by their families and/or communities. Alternatively, a social benefit may result (eg, a participant could feel good helping others).

Social harms are negative social impact events and social benefits are positive social impact events that a participant reports as affecting them as a result of being involved in a research study. It is not the researcher's opinion of how they perceive an event has affected a participant. Social impacts will be collected and reported on CRFs during scheduled visits (see Appendix J through Appendix M). A social harm that is reported by the participant and judged by the IoR/designee to be serious or unexpected will be reported to the responsible site's IRB at least annually, or according to their individual requirements. In the event that a participant reports a social harm, every effort will be made by study staff to provide appropriate care and counseling to the participant as necessary, and/or referral to appropriate resources for the safety of the participant. While maintaining participant confidentiality, study sites may engage their Community

#### HVTN 703/HPTN 081 Version 4.0 / December 14, 2017

Advisory Board (CAB) in exploring the social context surrounding instances of social harms to minimize the potential occurrence of such an impact.

# 11 Protocol conduct

This protocol and all actions and activities connected with it will be conducted in compliance with Good Clinical Practice (GCP) (ICHe6), the HVTN and HPTN network-specific *Manuals of Operations*, and DAIDS Clinical Research Policies and Standard Procedures Documents, including procedures for the following:

- Protocol registration, activation, and implementation;
- Informed consent, screening, and enrollment;
- Study participant reimbursement;
- Clinical and safety assessments;
- Safety monitoring and reporting;
- Data collection, documentation, transfer, and storage;
- Participant confidentiality;
- Study follow-up and close-out;
- Unblinding of staff and participants;
- Quality control;
- Protocol monitoring and compliance;
- Advocacy and assistance to participants regarding negative social impacts associated with the trial;
- Risk reduction counseling;
- Specimen collection, processing, and analysis;
- Ancillary studies, and
- Destruction of specimens.

Any policies or procedures that vary from DAIDS, HVTN, or HPTN standards or require additional instructions (eg, instructions for randomization specific to this study) will be described in the SSP.

# 11.1 Emergency communication with study participants

As in all clinical research, this study may generate a need to reach participants quickly to avoid imminent harm, or to report study findings that may otherwise concern their health or welfare.

When such communication is needed, the CRS will request that its IRB/EC and any applicable RE expedite review of the message. If this review cannot be completed in a timeframe consistent with the urgency of the required communication, the site should contact the participant first, and then notify the IRB/EC and any applicable RE of the matter as soon as possible.

# 12 Ethical considerations

It is critical that universally accepted ethical guidelines are followed at all sites involved in the conduct of clinical trials. The HVTN and HPTN (hereafter, referred to as the "Networks") have addressed ethical concerns in the following ways:

- Network trials are designed and conducted to enhance the knowledge base necessary to find new methods for preventing HIV infection, using methods that are scientifically rigorous and valid, and in accordance with GCP guidelines.
- Network scientists and operational staff incorporate the philosophies underlying major codes [136-138], declarations, and other guidance documents relevant to human subjects research into the design and conduct of HIV prevention clinical trials.
- Network scientists and operational staff are committed to substantive community input—into the planning, conduct, and follow-up of its research—to help ensure that locally appropriate cultural and linguistic needs of study populations are met. CABs are required by DAIDS and supported at all Network research sites to ensure community input, in accordance with Good Participatory Practices (GPP) and all local and national guidelines [139].
- Network clinical trial staff counsel study participants routinely on how to reduce HIV risk. Participants who become HIV infected during the trial are provided counseling on notifying their partners and about HIV infection according to local guidelines. Staff members will also counsel them about reducing their risk of transmitting HIV to others.
- The Networks require that all international Network sites lacking national plans for providing ART develop plans for the care and treatment of participants who acquire HIV infection during a trial. Each plan is developed in consultation with representatives of host countries, communities from which potential trial participants will be drawn, sponsors, and the Networks. Participants will be referred to programs for ART provision when the appropriate criteria for starting ART are met. If a program is not available at a site and ART is needed, a privately established fund will be used to pay for access to treatment to the fullest extent possible.
- The Networks agree that appropriate referrals for access to PrEP and PEP should be provided according to national and/or local guidelines.
- The Networks provide training so that all participating sites similarly ensure fair participant selection, protect the privacy of research participants, and obtain meaningful informed consent. During the study, participants will have

their wellbeing monitored, and to the fullest extent possible, their privacy protected. Participants may withdraw from the study at any time.

- Prior to implementation, Network trials are rigorously reviewed by scientists who are not involved in the conduct of the trials under consideration.
- Network trials are reviewed by local and national regulatory bodies and are conducted in compliance with all applicable national and local regulations.
- The Networks design their research to minimize risk and maximize benefit to both study participants and their local communities. For example, Network protocols provide enhancement of participants' knowledge of HIV and HIV prevention, as well as counseling, guidance, and assistance with any social impacts that may result from research participation. Network protocols also include careful medical review of each research participant's health conditions and reactions to study products while in the study.
- Network research aims to benefit local communities by directly addressing the health and HIV prevention needs of those communities and by strengthening the capacity of the communities through training, support, shared knowledge, and equipment. Researchers involved in Network trials are able to conduct other critical research in their local research settings.
- The Networks recognize the importance of institutional review and values the role of in country IRBs, ECs, and any applicable REs as custodians responsible for ensuring the ethical conduct of research in each setting.

#### 13 IRB/EC/RE review considerations

US Food and Drug Administration (FDA) and other US federal regulations require IRBs/ECs to ensure that certain requirements are satisfied on initial and continuing review of research (Title 45, Code of Federal Regulations (CFR), Part 46.111(a) 1-7; 21 CFR 56.111(a) 1-7). The following section highlights how this protocol addresses each of these research requirements. Each Network Investigator welcomes IRB/EC and any applicable RE questions or concerns regarding these research requirements.

This trial is being conducted in Africa, with funding from the US NIH. Due to this, the trial is subject to both US and local regulations and guidelines on the protection of human research subjects and ethical research conduct. Where there is a conflict in regulations or guidelines, the regulation or guideline providing the maximum protection of human research subjects will be followed.

In compliance with international and local (as appropriate) GCP, each research location has a locally based Principal Investigator (PI) who is qualified to conduct (and supervise the conduct of) the research; and the research addresses an important local health need for an HIV prevention method. In addition, the investigators take responsibility for the conduct of the study and the control of the study products, including obtaining all appropriate regulatory and ethical reviews of the research. Each participating site has a standard operating procedure for ensuring that participants have the necessary information to make a decision whether or not to consent to the research.

The sections below address each of the review concerns by IRBs/ECs and any applicable REs regarding how the research will be conducted.

#### 13.1 Minimized risks to participants

# 45 CFR 46.111 (a) 1 and 21 CFR 56.111 (a) 1: Risks to subjects are minimized.

This protocol minimizes risks to participants by (a) correctly and promptly informing participants about risks so that they can join in partnership with the researcher in recognizing and reporting harms; (b) respecting local/national blood draw limits; (c) performing direct observation of participants following study product administration and collecting information regarding side effects for several days following study product administration; (d) having staff properly trained in administering study procedures that may cause physical harm or psychological distress, such as blood draws, study product infusions, HIV testing and counseling and HIV risk reduction counseling; (e) providing HIV risk reduction counseling and checking on contraception use; and (f) providing safety monitoring.

#### 13.2 Reasonable risk/benefit balance

45 CFR 46.111(a) 2 and 21 CFR 56.111(a) 2: Risks to subjects are reasonable in relation to anticipated benefits, if any, to subjects, and the importance of the knowledge that may reasonably be expected to result.

In all public health research, the risk-benefit ratio may be difficult to assess because the benefits to a healthy participant are not as apparent as they would be in treatment protocols, where a study participant may be ill and may have exhausted all conventional treatment options. However, this protocol is designed to minimize the risks to participants while maximizing the potential value of the knowledge it is designed to generate.

#### 13.3 Equitable subject selection

# 45 CFR 46.111 (a) 3 and 21 CFR 56.111 (a) 3: Subject selection is equitable

This protocol has specific inclusion and exclusion criteria for investigators to follow in admitting participants into the protocol. Participants are selected because of these criteria and not because of positions of vulnerability or privilege. Investigators are required to maintain screening and enrollment logs to document volunteers who screened into and out of the protocol and for what reasons.

#### 13.4 Appropriate informed consent

45 CFR 46.111 (a) 4 & 5 and 21 CFR 56.111 (a) 4 & 5: Informed consent is sought from each prospective subject or the subject's legally authorized representative as required by 45 CFR 46.116 and 21 CFR Part 50; informed consent is appropriately documented as required by 45 CFR 46.117 and 21 CFR 50.27

The protocol specifies that informed consent must be obtained before any study procedures are initiated and assessed throughout the trial (see Section 7.1). Each site is provided training in informed consent by the Networks as part of its entering the respective Network. The Networks require a signed consent document for documentation, in addition to chart notes or a consent checklist.

#### 13.5 Adequate safety monitoring

45 CFR 46.111 (a) 6 and 21 CFR 56.111 (a) 6: There is adequate provision for monitoring the data collected to ensure the safety of subjects.

This protocol has extensive safety monitoring in place (Section 10). Safety is monitored daily by the HVTN CSS or HVTN Core designee and routinely by the HVTN 703/HPTN 081 PSRT. In addition, a DSMB periodically reviews study data.

#### 13.6 Protect privacy/confidentiality

45 CFR 46.111 (a) 7 and 21 CFR 56.111 (a) 7: There are adequate provisions to protect the privacy of subjects and maintain the confidentiality of data.

Privacy refers to an individual's right to be free from unauthorized or unreasonable intrusion into his/her private life and the right to control access to individually identifiable information about him/her. The term "privacy" concerns research participants or potential research participants as individuals whereas the term "confidentiality" is used to refer to the treatment of information about those individuals. This protocol respects the privacy of participants by informing them about who will have access to their personal information and study data (see Appendix A). The privacy of participants is protected by assigning unique identifiers in place of the participant's name on study data and specimens. In addition, each staff member at each study site in this protocol signs an Agreement on Confidentiality and Use of Data/Specimens with the Networks and each study site participating in the protocol is required to have a standard operating procedure on how the staff members will protect the confidentiality of study participants.

# 14 Version history

The Protocol Team may modify the original version of the protocol. Modifications are made to Network protocols via clarification memos, letters of amendment, or full protocol amendments.

The version history of, and modifications to, Protocol HVTN 703/HPTN 081 are described below.

**Protocol history and modifications** 

#### Date: December 14, 2017

Protocol version: Version 4.0

Protocol modification: Full Protocol Amendment 3

- Item 1 Sample size increased from 1500 to 1900
- Item 2 Added in Appendices A and C: Broad regulatory agency access to participant study records

#### **Date: August 25, 2017**

Protocol version: Version 3.0

Protocol modification: Full Protocol Amendment 2

- Item 1 Revised: Study duration and participant follow-up
- Item 2 Updated in Section 1.1: Protocol team membership
- Item 3 Revised in Section 2.4.5, *Trial monitoring*: Feasibility assessment
- Item 4 Updated in Sections 2.9, 2.9.3, 2.9.4, 2.10, and Appendix A: VRC01 clinical experience in HVTN 104
- Item 5 Updated in Section 2.9.5, *Particle formation*, and Section 6.2, *Study product formulation*: Product description and formulation/preparation instructions
- Item 6 Revised in Section 4.7.3: Monitoring for futility to assess PE
- Item 7 Clarified in Section 5: Eligibility determination
- Item 8 Clarified in Section 5.2, *Exclusion criteria*: Tissue or organ transplantation exclusion criterion
- Item 9 Clarified in Section 6.4, *Administration*: IV bag label weight and IV tubing flushing
- Item 10 Clarified in Section 7.3, *Enrollment and infusion visits*: Timing of HIV infection assessment and HIV testing
- Item 11 Updated in Section 7.10, Assessments of reactogenicity, Section 10.2.2, AE reporting, and Section 15, Document references (other than literature citations): DAIDS AE grading table version and exceptions
- Item 12 Updated in Sections 10.2: URLs for referenced documents

- Item 13 Updated in Section 10.2.3: Expedited reporting of adverse events to DAIDS
- Item 14 Updated in Section 14: Version history
- Item 15 Updated in Section 15, *Document references (other than literature citations)*: Documents and URLs
- Item 16 Updated in Section 16: Acronyms and abbreviations
- Item 17 Updated in Appendix A, Sample informed consent form: Minimum infusion time
- Item 18 Corrected in Appendix A, Sample informed consent form: Blood draw volumes
- Item 19 Clarified in Appendix A, Sample informed consent form: Early termination
- Item 20 Revised in Appendix B, *Approved birth control methods (for sample informed consent form)*: Approved contraception methods
- Item 21 Corrected in Appendix D, *Tables of procedures (for sample informed consent form)*: Procedure timepoint
- Item 22 Clarified in Appendix F: DBS allowance applies to Visit and 56-day blood draw totals
- Item 23 Updated in Appendices F through I: Assay locations and HVTN laboratory listings
- Item 24 Revised in Appendices G, H, K, and L: Table format and Schedule 3 blood draws at Visit #.X
- Item 25 Clarified in Appendices J and M: Provision of HIV test results
- Item 26 Added as Appendix N: Protocol signature page
- Item 27 Updated in Sections 6.2 through 6.4 per Clarification Memo 1 to protocol Version 2.0: Study product description, storage, and administration instructions
- Item 28 Corrected: Minor typographical, grammatical, and formatting errors

#### **Date: March 8, 2017**

Protocol version: Version 2.0

Protocol modification: Clarification Memo 1

- Item 1 Updated in Section 6.2, *Study product formulation*: VRC01 description and storage temperature
- Item 2 Revised in Sections 6.3 and 6.4: Holding times for study products after preparation
- Item 3 Updated in Section 6.4, Administration: Minimum infusion time period
- Item 4 Added in Section 6.4, *Administration*: In-line filter set requirement
- Item 5 Clarified in Sections 6.3.1 and 6.3.2: VRC01 vials with visible particles not to be used

#### Date: June 24, 2016


Protocol modification: Full Protocol Amendment 1

- Item 1 Study population limited to women in sub-Saharan Africa at risk of acquiring HIV through sexual transmission
- Item 2 Added in Section 1, Overview: Note regarding enrollment numbers
- Item 3 Revised in Section 1, *Overview*, and Section 5.1, *Inclusion criteria*: Participant age range
- Item 4 Updated in Section 1.1, Protocol Team: Membership and affiliations
- Item 5 Clarified in Section 2.1, *Rationale for trial concept*: Worldwide HIV infections and licensure status of VRC01
- Item 6 Updated: Section 2.4.5, Trial monitoring
- Item 7 Updated: Section 2.6, Plans for future product development and testing
- Item 8 Added in Section 2.8.1, *Protection against* challenge *in NHP models*: Non-neutralizing mechanisms of bnAb protection in NHP challenge studies
- Item 9 Added in Section 2.9.2, *VRC 602*: Information on serum neutralizing activity and anti-VRC01 antibodies
- Item 10 Updated in Sections 2.9.3 and 2.9.4: Phase 1 clinical trial experience and VRC01 safety summary
- Item 11 Added in Section 2.9.3: VRC01 pharmacokinetics in HVTN 104
- Item 12 Revised in Sections 3.3, 4.8, and 9.6 and Appendix F: PrEP use monitoring
- Item 13 Revised: Section 4, Statistical considerations
- Item 14 Clarified in Section 5.1, *Inclusion criteria*: Urine protein measures
- Item 15 Revisions in Section 5.2: Exclusion criteria
- Item 16 Clarified in Section 5.3.3, *Discontinuing infusions for a participant*:

  Participants for whom infusions are stopped for reasons other than HIV infection
- Item 17 Updated in Section 6, *Study product preparation and administration*: Study product regimen, formulation, storage, preparation, and administration instructions
- Item 18 Removed in Section 7.2, *Pre-enrollment procedures*: Required recording of generic names for concomitant medications
- Item 19 Clarified in Section 7.3, *Enrollment and infusion visits*: Urine dipstick and instructions for infusion observation and reactogenicity assessment
- Item 20 Corrected in Section 7.4: Post-infusion visits for HIV-uninfected study participants
- Item 21 Corrected in Section 7.5, *HIV counseling and testing*: PrEP information source

- Item 22 Clarified in Section 7.5.1, *Study product-related seroreactivity*: Serum concentrations tested and reference to HIV testing only
- Item 23 Added as (new) Section 7.6: Follow-up visits for HIV-infected participants
- Item 24 Added as (new) Section 7.7 and Appendices I and M: Follow-up for study participants for whom infusions have been stopped for reasons other than HIV infection
- Item 25 Corrected in Section 7.8, *Contraception status*: Where to find details regarding contraception requirements
- Item 26 Clarified in Section 7.9 and Appendices F, I, J, and M: Urine testing
- Item 27 Clarified in Sections 7.10, *Assessments of reactogenicity*: Systemic and local signs and symptoms and infusion sites reactions
- Item 28 Revised in Section 7.11, *Visit windows and* missed *visits*: Visits for performance of safety assessments and local safety labs
- Item 29 Corrected in Section 8.5, *HIV infection during* the *study*: Visit schedules for HIV-infected study participants
- Item 30 Revised in Section 9.5.1, Anti-VRC01 antibody assay: Assay description
- Item 31 Clarified in Section 9.5.2, *Neutralizing antibody* assay: Range of applicability
- Item 32 Clarified in Section 10.1.1, *HVTN 703/HPTN* 081 *PSRT*: Protocol safety review team membership
- Item 33 Removed in Section 10.1.3, *Roles and responsibilities in safety monitoring*: Reference to planned holds
- Item 34 Added in Section 10.2.2, *AE reporting*: Uterine bleeding secondary to contraception
- Item 35 Added in Section 10.2.2, AE reporting: African working hours
- Item 36 Updated in Section 10.2.3, Expedited reporting of adverse events to DAIDS: DAERS support email address
- Item 37 Corrected in Section 10.4.2: PSRT review timing
- Item 38 Clarified in Section 10.4.3: Cumulative safety data reports to DSMB
- Item 39 Removed in Section 10.6, *Social impact reporting*: Reference to Study Specific Procedures (SSP)
- Item 40 Updated in Section 15: URL for DAIDS source documentation requirements
- Item 41 Updated and clarified: Appendix A, Sample informed consent form
- Item 42 Added in Appendix A and (optional) Appendix E: Consent for HIV-infected study participants
- Item 43 Clarified in Appendix A and C consent forms: Potential genetic testing
- Item 44 Added in Appendix A, C, and E consent forms: MCC contact information

- Item 45 Added in Appendix B, *Approved birth control methods*: Injectable contraceptives
- Item 46 Added in Appendix D: Procedure tables for HIV-infected participants and for participants whose infusions have been stopped for reasons other than HIV infection
- Item 47 Clarified in footnotes to Appendix F and J: Pregnancy testing
- Item 48 Clarified in Appendices F, G, and I: HVTN and non-HVTN endpoint laboratories
- Item 49 Added in Appendix F: VRC lab for anti-VRC01 antibody levels
- Item 50 Corrected in Appendices G, H, K, and L: Appendix titles, visit schedules, visit numbering, and procedures
- Item 51 Added in Appendices G and H: Whole blood samples for confirmatory HIV testing
- Item 52 Clarified in Appendix J, Schedule 1—Procedures at CRS for HIV-uninfected participants: No participant questionnaire at Visit 0 (screening visit)
- Item 53 Added to Appendices K and L: Local lab assessments
- Item 54 Updated and corrected throughout the protocol document: Acronyms, abbreviations, numbering of figures, tables, and appendices, cross-references, and grammatical errors

## Date: April 15, 2016

Protocol version: Version 1.0

Protocol modification: Clarification Memo 2

Item 1 Clarified in Appendix I, Schedule 1—Procedures at CRS for HIV-uninfected participants: No participant questionnaire during screening

#### Date: February 22, 2016


Protocol modification: Clarification Memo 1

Item 1 Corrected in Appendices G, H, J, and K: Visit numbering

[Note: Clarification Memo 1 dated February 22, 2016 replaces Clarification Memo 1 dated September 4, 2015 and Letter of Amendment 1 dated September 28, 2015.]

## Date: September 28, 2015


Protocol modification: Letter of Amendment 1

- Item 1 Corrected in Appendices G, H, J, and K: Visit schedules
- Item 2 Clarified in Appendices J and K: Assessment of HIV/AIDS-related conditions applies to both complete and abbreviated physical exams

# Item 3 Removed in Appendices J and K: Social impact assessment questionnaire

# Date: September 4, 2015


Protocol modification: Clarification Memo 1

Item 1 Corrected in Appendices G, H, J, and K: Visit numbering

Item 2 Corrected: Titles of Appendices J and K

# **Date: August 11, 2015**

Protocol version: 1.0

Protocol modification: NA

# 15 Document references (other than literature citations)

Other documents referred to in this protocol, and containing information relevant to the conduct of this study, include:

- Assessment of Understanding. Accessible through the HVTN protocolspecific website.
- Current CDC Guidelines. Revised Recommendations for HIV Testing of Adults, Adolescents, and Pregnant Women in Health-Care Settings. Available at http://www.cdc.gov/mmwr/PDF/rr/rr5514.pdf
- Division of AIDS (DAIDS) Clinical Research Policies and Standard Procedures Documents. Available at https://www.niaid.nih.gov/research/daids-clinical-research-policies-standard-procedures
- Division of AIDS Protocol Registration Manual. Available at https://www.niaid.nih.gov/sites/default/files/prmanual.pdf
- Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events. Version 2.1, dated July 2017. Available at http://rsc.techres.com/clinical-research-sites/safety-reporting/daids-grading-tables
- The Manual for Expedited Reporting of Adverse Events to DAIDS. Version 2.0, January 2010. Available at http://rsc.tech-res.com/clinical-research-sites/safety-reporting/manual
- HVTN Certificate of Confidentiality. Accessible through the HVTN website.
- HVTN 703/HPTN 081 Special Instructions. Accessible through the HVTN protocol-specific website.
- HVTN 703/HPTN 081 Study Specific Procedures. Accessible through the HVTN protocol-specific website.
- HVTN Manual of Operations. Accessible through the HVTN website.
- Dangerous Goods Regulations (updated annually), International Air Transport Association. Available for purchase at http://www.iata.org/publications/dgr/Pages/index.aspx
- HVTN Lab Assay Algorithm (available upon request)
- International Conference on Harmonisation (ICH) E6 (R1), Guideline for Good Clinical Practice: Section 4.8, Informed consent of trial subjects.

Available at http://www.ich.org/products/guidelines/efficacy/article/efficacy-guidelines.html

- HVTN 703/HPTN 081 Participants' Bill of Rights and Responsibilities. Accessible through the HVTN website.
- NIH Policy on Reporting Race and Ethnicity Data: Subjects in Clinical Research. Available at http://grants1.nih.gov/grants/guide/notice-files/NOT-OD-01-053.html
- Pharmacy Guidelines and Instructions for DAIDS Clinical Trials Networks, July 2008.
- Requirements for Source Documentation in DAIDS Funded and/or Sponsored Clinical Trials. Available at https://www.niaid.nih.gov/labsandresources/resources/daidsclinrsrch/Pages/ClinicalSite.aspx
- Title 21, Code of Federal Regulations, Part 50. Available at http://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfcfr/CFRSearch.cfm?CFR Part=50
- Title 45, Code of Federal Regulations, Part 46. Available at http://www.hhs.gov/ohrp/humansubjects/guidance/45cfr46.html

See Section 17 for literature cited in the background and statistics sections of this protocol.

# 16 Acronyms and abbreviations

ACASI audio computer assisted self-interview
ADCC antibody-dependent cellular cytotoxicity
ADCP antibody-dependent cellular phagocytosis
ADCVI antibody-dependent cellular viral inhibition

AIA anti-idiotypic antibody ALP alkaline phosphatase ALT alanine aminotransferase

aPTT activated partial thromboplastin time

ART antiretroviral therapy ARV antiretroviral (drug)

AST aspartate aminotransferase bnAb broadly neutralizing antibody CAB Community Advisory Board

CBC complete blood count

CDC US Centers for Disease Control and Prevention

CFR Code of Federal Regulations

CHO Chinese hamster ovary
CI confidence intervals
CRF case report form

CRPMC (NIAID) Clinical Research Products Management Center

CRS\* clinical research site

DAERS DAIDS Adverse Experience Reporting System

DAIDS Division of AIDS (US NIH)

DHHS US Department of Health and Human Services
DSMB (NIAID) Data and Safety Monitoring Board

EAE adverse events requiring expedited reporting to DAIDS

EC Ethics Committee
EIA enzyme immunoassay

ELISA enzyme-linked immunosorbent assay

FcRn neonatal Fc receptor

FDA US Food and Drug Administration

FHCRC Fred Hutchinson Cancer Research Center

FTC emtricitabine GC gonorrhea

GCP Good Clinical PracticeGLP Good Laboratory PracticeGMP Good Manufacturing Practice

Hgb hemoglobin

#### HVTN 703/HPTN 081 Version 4.0 / December 14, 2017

HIPAA Health Insurance Portability and Accountability Act

HPTN HIV Prevention Trials Network HVTN HIV Vaccine Trials Network

IB Investigator's Brochure

IC<sub>50</sub> inhibitory concentration (50%)

ICF informed consent form

ICH International Conference on Harmonisation

IgG immunoglobulin G

IND Investigational New Drug (application)

IRB Institutional Review Board

IV intravenous

LANL Los Alamos National Laboratory

LC Laboratory Center

LOC Leadership and Operations Center

mAb monoclonal antibody
MITT modified intent-to-treat
MSM men who have sex with men

NDOH (South Africa) National Department of Health

NHP nonhuman primate

NIAID National Institute of Allergy and Infectious Diseases (US NIH)

NICD National Institute for Communicable Diseases (Johannesburg, South

Africa)

NIH US National Institutes of Health

NVITAL NIAID Vaccine Immune T-Cell Antibody Laboratory

OC Oversight Committee

PBMC peripheral blood mononuclear cell

PE prevention efficacy

PEP postexposure prophylaxis
PI Principal Investigator

PK pharmacokinetic

PMTCT prevention of mother-to-child (HIV) transmission

PrEP pre-exposure prophylaxis
PSRT Protocol Safety Review Team

PYR person year

RAB DAIDS Regulatory Affairs Branch

RE regulatory entity

RSC (DAIDS) Regulatory Support Center

RSV respiratory syncytial virus SAE serious adverse event

#### HVTN 703/HPTN 081 Version 4.0 / December 14, 2017

SC subcutaneous

SCHARP Statistical Center for HIV/AIDS Research and Prevention

SDMC statistical and data management center SHIV simian-human immunodeficiency virus

SPT DAIDS Safety and Pharmacovigilance Team

SSP study specific procedures
STI sexually transmitted infection

TasP treatment as prevention

TCID<sub>50</sub> tissue culture infectious dose (50%)

TDF tenofovir disoproxil fumarate

TFV tenofovir TG transgender

tMLE targeted maximum likelihood estimation

USP United States Pharmacopeia

UW-VSL University of Washington Virology Specialty Laboratory

VRC Vaccine Research Center (NIAID)

VRP Vaccine Research Program WHO World Health Organization

<sup>\*</sup> CRSs were formerly referred to as HIV Vaccine Trial Units (HVTUs). Conversion to use of the term CRS is in process, and some HVTN documents may still refer to HVTUs.

## 17 Literature cited

- UNAIDS. Report on the Global AIDS Epidemic, 2012 country progress reports. http://www.unaids.org/en/dataanalysis/knowyourresponse/countryprogressreports/2012 countries/. 2013. Last accessed: 2-20-2013
- 2. UNAIDS. Global Report: Report on the global AIDS epidemic 2013. **2013**;UNAIDS / JC2502/1/E.
- 3. WHO in partnership with UNICEF and UNAIDS. Global Report on HIV Treatment 2013: Results, Impact and Opportunities. **2014**.
- 4. UNAIDS. Local Epidemics Issues Brief. 2014.
- 5. HIV/AIDS Fact Sheet.11-2015. <a href="http://www.who.int/mediacentre/factsheets/fs360/en/">http://www.who.int/mediacentre/factsheets/fs360/en/</a>, accessed February 8, 2016.
- 6. Cohen MS, Chen YQ, McCauley M, Gamble T, Hosseinipour MC, Kumarasamy N, Hakim JG, Kumwenda J, Grinsztejn B, Pilotto JH, Godbole SV, Mehendale S, Chariyalertsak S, Santos BR, Mayer KH, Hoffman IF, Eshleman SH, Piwowar-Manning E, Wang L, Makhema J, Mills LA, de BG, Sanne I, Eron J, Gallant J, Havlir D, Swindells S, Ribaudo H, Elharrar V, Burns D, Taha TE, Nielsen-Saines K, Celentano D, Essex M, Fleming TR. Prevention of HIV-1 infection with early antiretroviral therapy. N Engl J Med 2011;365:493-505.
- 7. Grant RM, Lama JR, Anderson PL, McMahan V, Liu AY, Vargas L, Goicochea P, Casapia M, Guanira-Carranza JV, Ramirez-Cardich ME, Montoya-Herrera O, Fernandez T, Veloso VG, Buchbinder SP, Chariyalertsak S, Schechter M, Bekker LG, Mayer KH, Kallas EG, Amico KR, Mulligan K, Bushman LR, Hance RJ, Ganoza C, Defechereux P, Postle B, Wang F, McConnell JJ, Zheng JH, Lee J, Rooney JF, Jaffe HS, Martinez AI, Burns DN, Glidden DV. Preexposure chemoprophylaxis for HIV prevention in men who have sex with men. N Engl J Med 2010;363:2587-99.
- 8. Guidelines for the Use of Antiretroviral Agents in HIV-1-Infected Adults and Adolescents: Limitations to Treatment Safety and Efficacy: Adverse Effects of Antiretroviral Agents. http://aidsinfo.nih.gov/guidelines. 5-1-2014. Last accessed: 2-17-2015
- 9. van der Straten A, Van Damme L, Haberer JE, Bangsberg DR. Unraveling the divergent results of pre-exposure prophylaxis trials for HIV prevention. AIDS **2012**;26:F13-F19.
- 10. Winokur PL, Stapleton JT. Immunoglobulin prophylaxis for hepatitis A. Clin Infect Dis **1992**;14:580-6.
- 11. Fiore AE, Wasley A, Bell BP. Prevention of hepatitis A through active or passive immunization: recommendations of the Advisory Committee on Immunization Practices (ACIP). MMWR Recomm Rep **2006**;55:1-23.
- 12. Graham BS, Ambrosino DM. History of passive antibody administration for prevention and treatment of infectious diseases. Curr Opin HIV AIDS **2015**;10:129-34.

- 13. Palivizumab, a Humanized Respiratory Syncytial Virus Monoclonal Antibody, Reduces Hospitalization From Respiratory Syncytial Virus Infection in High-risk Infants. Pediatrics **1998**;102:531-7.
- 14. Carbonell-Estrany X, Simoes EA, Dagan R, Hall CB, Harris B, Hultquist M, Connor EM, Losonsky GA. Motavizumab for prophylaxis of respiratory syncytial virus in high-risk children: a noninferiority trial. Pediatrics **2010**;125:e35-e51.
- 15. Homaira N, Rawlinson W, Snelling TL, Jaffe A. Effectiveness of Palivizumab in Preventing RSV Hospitalization in High Risk Children: A Real-World Perspective. Int J Pediatr **2014**;2014:571609.
- 16. Li Y, Migueles SA, Welcher B, Svehla K, Phogat A, Louder MK, Wu X, Shaw GM, Connors M, Wyatt RT, Mascola JR. Broad HIV-1 neutralization mediated by CD4-binding site antibodies. Nat Med **2007**;13:1032-4.
- 17. Simek MD, Rida W, Priddy FH, Pung P, Carrow E, Laufer DS, Lehrman JK, Boaz M, Tarragona-Fiol T, Miiro G, Birungi J, Pozniak A, McPhee DA, Manigart O, Karita E, Inwoley A, Jaoko W, Dehovitz J, Bekker LG, Pitisuttithum P, Paris R, Walker LM, Poignard P, Wrin T, Fast PE, Burton DR, Koff WC. Human immunodeficiency virus type 1 elite neutralizers: individuals with broad and potent neutralizing activity identified by using a high-throughput neutralization assay together with an analytical selection algorithm. J Virol 2009;83:7337-48.
- 18. Wu X, Yang ZY, Li Y, Hogerkorp CM, Schief WR, Seaman MS, Zhou T, Schmidt SD, Wu L, Xu L, Longo NS, McKee K, O'Dell S, Louder MK, Wycuff DL, Feng Y, Nason M, Doria-Rose N, Connors M, Kwong PD, Roederer M, Wyatt RT, Nabel GJ, Mascola JR. Rational design of envelope identifies broadly neutralizing human monoclonal antibodies to HIV-1. Science **2010**;329:856-61.
- 19. Zhou T, Georgiev I, Wu X, Yang ZY, Dai K, Finzi A, Kwon YD, Scheid JF, Shi W, Xu L, Yang Y, Zhu J, Nussenzweig MC, Sodroski J, Shapiro L, Nabel GJ, Mascola JR, Kwong PD. Structural basis for broad and potent neutralization of HIV-1 by antibody VRC01. Science **2010**;329:811-7.
- 20. Gray ES, Taylor N, Wycuff D, Moore PL, Tomaras GD, Wibmer CK, Puren A, DeCamp A, Gilbert PB, Wood B, Montefiori DC, Binley JM, Shaw GM, Haynes BF, Mascola JR, Morris L. Antibody specificities associated with neutralization breadth in plasma from human immunodeficiency virus type 1 subtype C-infected blood donors. J Virol 2009:83:8925-37.
- 21. Gray ES, Madiga MC, Hermanus T, Moore PL, Wibmer CK, Tumba NL, Werner L, Mlisana K, Sibeko S, Williamson C, Abdool Karim SS, Morris L. The neutralization breadth of HIV-1 develops incrementally over four years and is associated with CD4+ T cell decline and high viral load during acute infection. J Virol **2011**;85:4828-40.
- 22. Corti D, Langedijk JP, Hinz A, Seaman MS, Vanzetta F, Fernandez-Rodriguez BM, Silacci C, Pinna D, Jarrossay D, Balla-Jhagjhoorsingh S, Willems B, Zekveld MJ, Dreja H, O'Sullivan E, Pade C, Orkin C, Jeffs SA, Montefiori DC, Davis D, Weissenhorn W, McKnight A, Heeney JL, Sallusto F, Sattentau QJ, Weiss RA, Lanzavecchia A. Analysis of memory B cell responses and isolation of novel monoclonal antibodies with neutralizing breadth from HIV-1-infected individuals. PLoS ONE **2010**;5:e8805.

- 23. Walker LM, Huber M, Doores KJ, Falkowska E, Pejchal R, Julien JP, Wang SK, Ramos A, Chan-Hui PY, Moyle M, Mitcham JL, Hammond PW, Olsen OA, Phung P, Fling S, Wong CH, Phogat S, Wrin T, Simek MD, Koff WC, Wilson IA, Burton DR, Poignard P. Broad neutralization coverage of HIV by multiple highly potent antibodies. Nature **2011**;477:466-70.
- 24. Scheid JF, Mouquet H, Ueberheide B, Diskin R, Klein F, Oliveira TY, Pietzsch J, Fenyo D, Abadir A, Velinzon K, Hurley A, Myung S, Boulad F, Poignard P, Burton DR, Pereyra F, Ho DD, Walker BD, Seaman MS, Bjorkman PJ, Chait BT, Nussenzweig MC. Sequence and structural convergence of broad and potent HIV antibodies that mimic CD4 binding. Science 2011;333:1633-7.
- 25. Binley JM, Lybarger EA, Crooks ET, Seaman MS, Gray E, Davis KL, Decker JM, Wycuff D, Harris L, Hawkins N, Wood B, Nathe C, Richman D, Tomaras GD, Bibollet-Ruche F, Robinson JE, Morris L, Shaw GM, Montefiori DC, Mascola JR. Profiling the specificity of neutralizing antibodies in a large panel of plasmas from patients chronically infected with human immunodeficiency virus type 1 subtypes B and C. J Virol 2008;82:11651-68.
- 26. Sather DN, Armann J, Ching LK, Mavrantoni A, Sellhorn G, Caldwell Z, Yu X, Wood B, Self S, Kalams S, Stamatatos L. Factors associated with the development of cross-reactive neutralizing antibodies during human immunodeficiency virus type 1 infection. J Virol 2009;83:757-69.
- 27. Falkowska E, Ramos A, Feng Y, Zhou T, Moquin S, Walker LM, Wu X, Seaman MS, Wrin T, Kwong PD, Wyatt RT, Mascola JR, Poignard P, Burton DR. PGV04, an HIV-1 gp120 CD4 binding site antibody, is broad and potent in neutralization but does not induce conformational changes characteristic of CD4. J Virol 2012;86:4394-403.
- 28. Walker LM, Phogat SK, Chan-Hui PY, Wagner D, Phung P, Goss JL, Wrin T, Simek MD, Fling S, Mitcham JL, Lehrman JK, Priddy FH, Olsen OA, Frey SM, Hammond PW, Kaminsky S, Zamb T, Moyle M, Koff WC, Poignard P, Burton DR. Broad and potent neutralizing antibodies from an African donor reveal a new HIV-1 vaccine target. Science 2009;326:285-9.
- 29. Walker LM, Simek MD, Priddy F, Gach JS, Wagner D, Zwick MB, Phogat SK, Poignard P, Burton DR. A limited number of antibody specificities mediate broad and potent serum neutralization in selected HIV-1 infected individuals. PLoS Pathog **2010**;6:e1001028.
- 30. McLellan JS, Pancera M, Carrico C, Gorman J, Julien JP, Khayat R, Louder R, Pejchal R, Sastry M, Dai K, O'Dell S, Patel N, Shahzad-ul-Hussan S, Yang Y, Zhang B, Zhou T, Zhu J, Boyington JC, Chuang GY, Diwanji D, Georgiev I, Kwon YD, Lee D, Louder MK, Moquin S, Schmidt SD, Yang ZY, Bonsignori M, Crump JA, Kapiga SH, Sam NE, Haynes BF, Burton DR, Koff WC, Walker LM, Phogat S, Wyatt R, Orwenyo J, Wang LX, Arthos J, Bewley CA, Mascola JR, Nabel GJ, Schief WR, Ward AB, Wilson IA, Kwong PD. Structure of HIV-1 gp120 V1/V2 domain with broadly neutralizing antibody PG9. Nature 2011;480:336-43.
- 31. Kong L, Lee JH, Doores KJ, Murin CD, Julien JP, McBride R, Liu Y, Marozsan A, Cupo A, Klasse PJ, Hoffenberg S, Caulfield M, King CR, Hua Y, Le KM, Khayat R, Deller MC, Clayton T, Tien H, Feizi T, Sanders RW, Paulson JC, Moore JP, Stanfield RL,

- Burton DR, Ward AB, Wilson IA. Supersite of immune vulnerability on the glycosylated face of HIV-1 envelope glycoprotein gp120. Nat Struct Mol Biol **2013**;20:796-803.
- 32. Huang J, Ofek G, Laub L, Louder MK, Doria-Rose NA, Longo NS, Imamichi H, Bailer RT, Chakrabarti B, Sharma SK, Alam SM, Wang T, Yang Y, Zhang B, Migueles SA, Wyatt R, Haynes BF, Kwong PD, Mascola JR, Connors M. Broad and potent neutralization of HIV-1 by a gp41-specific human antibody. Nature **2012**;491:406-12.
- 33. Stamatatos L, Morris L, Burton DR, Mascola JR. Neutralizing antibodies generated during natural HIV-1 infection: good news for an HIV-1 vaccine? Nat Med **2009**;15:866-70.
- 34. Walker LM, Burton DR. Rational antibody-based HIV-1 vaccine design: current approaches and future directions. Curr Opin Immunol **2010**;22:358-66.
- 35. Burton DR, Ahmed R, Barouch DH, Butera ST, Crotty S, Godzik A, Kaufmann DE, McElrath MJ, Nussenzweig MC, Pulendran B, Scanlan CN, Schief WR, Silvestri G, Streeck H, Walker BD, Walker LM, Ward AB, Wilson IA, Wyatt R. A Blueprint for HIV Vaccine Discovery. Cell Host Microbe 2012;12:396-407.
- 36. Burton DR, Stanfield RL, Wilson IA. Antibody vs. HIV in a clash of evolutionary titans. Proc Natl Acad Sci U S A **2005**;102:14943-8.
- 37. Kwong PD, Mascola JR. Human antibodies that neutralize HIV-1: identification, structures, and B cell ontogenies. Immunity **2012**;37:412-25.
- 38. Georgiev IS, Gordon JM, Zhou T, Kwong PD. Elicitation of HIV-1-neutralizing antibodies against the CD4-binding site. Curr Opin HIV AIDS **2013**;8:382-92.
- 39. Wu X, Wang C, O'Dell S, Li Y, Keele BF, Yang Z, Imamichi H, Doria-Rose N, Hoxie JA, Connors M, Shaw GM, Wyatt RT, Mascola JR. Selection pressure on HIV-1 envelope by broadly neutralizing antibodies to the conserved CD4-binding site. J Virol **2012**;86:5844-56.
- 40. Shibata R, Igarashi T, Haigwood N, Buckler-White A, Ogert R, Ross W, Willey R, Cho MW, Martin MA. Neutralizing antibody directed against the HIV-1 envelope glycoprotein can completely block HIV-1/SIV chimeric virus infections of macaque monkeys. Nat Med 1999;5:204-10.
- 41. Baba TW, Liska V, Hofmann-Lehmann R, Vlasak J, Xu W, Ayehunie S, Cavacini LA, Posner MR, Katinger H, Stiegler G, Bernacky BJ, Rizvi TA, Schmidt R, Hill LR, Keeling ME, Lu Y, Wright JE, Chou TC, Ruprecht RM. Human neutralizing monoclonal antibodies of the IgG1 subtype protect against mucosal simian-human immunodeficiency virus infection. Nat Med **2000**;6:200-6.
- 42. Hofmann-Lehmann R, Vlasak J, Rasmussen RA, Jiang S, Li PL, Baba TW, Montefiori DC, Bernacky BJ, Rizvi TA, Schmidt R, Hill LR, Keeling ME, Katinger H, Stiegler G, Cavacini LA, Posner MR, Ruprecht RM. Postnatal pre- and postexposure passive immunization strategies: protection of neonatal macaques against oral simian-human immunodeficiency virus challenge. J Med Primatol **2002**;31:109-19.

- 43. Nishimura Y, Igarashi T, Haigwood N, Sadjadpour R, Plishka RJ, Buckler-White A, Shibata R, Martin MA. Determination of a statistically valid neutralization titer in plasma that confers protection against simian-human immunodeficiency virus challenge following passive transfer of high-titered neutralizing antibodies. J Virol 2002;76:2123-30.
- 44. Hessell AJ, Rakasz EG, Poignard P, Hangartner L, Landucci G, Forthal DN, Koff WC, Watkins DI, Burton DR. Broadly neutralizing human anti-HIV antibody 2G12 is effective in protection against mucosal SHIV challenge even at low serum neutralizing titers. PLoS Pathog 2009;5:e1000433.
- 45. Hessell AJ, Poignard P, Hunter M, Hangartner L, Tehrani DM, Bleeker WK, Parren PW, Marx PA, Burton DR. Effective, low-titer antibody protection against low-dose repeated mucosal SHIV challenge in macaques. Nat Med **2009**;15:951-4.
- 46. Moldt B, Rakasz EG, Schultz N, Chan-Hui PY, Swiderek K, Weisgrau KL, Piaskowski SM, Bergman Z, Watkins DI, Poignard P, Burton DR. Highly potent HIV-specific antibody neutralization in vitro translates into effective protection against mucosal SHIV challenge in vivo. Proc Natl Acad Sci U S A **2012**;109:18921-5.
- 47. Pegu A, Yang ZY, Boyington JC, Wu L, Ko SY, Schmidt SD, McKee K, Kong WP, Shi W, Chen X, Todd JP, Letvin NL, Huang J, Nason MC, Hoxie JA, Kwong PD, Connors M, Rao SS, Mascola JR, Nabel GJ. Neutralizing antibodies to HIV-1 envelope protect more effectively in vivo than those to the CD4 receptor. Sci Transl Med 2014;6:243ra88.
- 48. Ko SY, Pegu A, Rudicell RS, Yang ZY, Joyce MG, Chen X, Wang K, Bao S, Kraemer TD, Rath T, Zeng M, Schmidt SD, Todd JP, Penzak SR, Saunders KO, Nason MC, Haase AT, Rao SS, Blumberg RS, Mascola JR, Nabel GJ. Enhanced neonatal Fc receptor function improves protection against primate SHIV infection. Nature **2014**;514:642-5.
- 49. Rudicell RS, Kwon YD, Ko SY, Pegu A, Louder MK, Georgiev IS, Wu X, Zhu J, Boyington JC, Chen X, Shi W, Yang ZY, Doria-Rose NA, McKee K, O'Dell S, Schmidt SD, Chuang GY, Druz A, Soto C, Yang Y, Zhang B, Zhou T, Todd JP, Lloyd KE, Eudailey J, Roberts KE, Donald BR, Bailer RT, Ledgerwood J, Mullikin JC, Shapiro L, Koup RA, Graham BS, Nason MC, Connors M, Haynes BF, Rao SS, Roederer M, Kwong PD, Mascola JR, Nabel GJ. Enhanced potency of a broadly neutralizing HIV-1 antibody in vitro improves protection against lentiviral infection in vivo. J Virol 2014;88:12669-82.
- 50. Florese RH, Demberg T, Xiao P, Kuller L, Larsen K, Summers LE, Venzon D, Cafaro A, Ensoli B, Robert-Guroff M. Contribution of nonneutralizing vaccine-elicited antibody activities to improved protective efficacy in rhesus macaques immunized with Tat/Env compared with multigenic vaccines. J Immunol 2009;182:3718-27.
- 51. Forthal DN, Landucci G, Phan TB, Becerra J. Interactions between natural killer cells and antibody Fc result in enhanced antibody neutralization of human immunodeficiency virus type 1. J Virol **2005**;79:2042-9.
- 52. Asmal M, Sun Y, Lane S, Yeh W, Schmidt SD, Mascola JR, Letvin NL. Antibodydependent cell-mediated viral inhibition emerges after simian immunodeficiency virus

- SIVmac251 infection of rhesus monkeys coincident with gp140-binding antibodies and is effective against neutralization-resistant viruses. J Virol **2011**;85:5465-75.
- 53. Tudor D, Derrien M, Diomede L, Drillet AS, Houimel M, Moog C, Reynes JM, Lopalco L, Bomsel M. HIV-1 gp41-specific monoclonal mucosal IgAs derived from highly exposed but IgG-seronegative individuals block HIV-1 epithelial transcytosis and neutralize CD4(+) cell infection: an IgA gene and functional analysis. Mucosal Immunol 2009;2:412-26.
- 54. Doria-Rose NA, Schramm CA, Gorman J, Moore PL, Bhiman JN, DeKosky BJ, Ernandes MJ, Georgiev IS, Kim HJ, Pancera M, Staupe RP, Altae-Tran HR, Bailer RT, Crooks ET, Cupo A, Druz A, Garrett NJ, Hoi KH, Kong R, Louder MK, Longo NS, McKee K, Nonyane M, O'Dell S, Roark RS, Rudicell RS, Schmidt SD, Sheward DJ, Soto C, Wibmer CK, Yang Y, Zhang Z, Mullikin JC, Binley JM, Sanders RW, Wilson IA, Moore JP, Ward AB, Georgiou G, Williamson C, Abdool Karim SS, Morris L, Kwong PD, Shapiro L, Mascola JR. Developmental pathway for potent V1V2-directed HIV-neutralizing antibodies. Nature 2014;509:55-62.
- 55. Pancera M, Shahzad-ul-Hussan S, Doria-Rose NA, McLellan JS, Bailer RT, Dai K, Loesgen S, Louder MK, Staupe RP, Yang Y, Zhang B, Parks R, Eudailey J, Lloyd KE, Blinn J, Alam SM, Haynes BF, Amin MN, Wang LX, Burton DR, Koff WC, Nabel GJ, Mascola JR, Bewley CA, Kwong PD. Structural basis for diverse N-glycan recognition by HIV-1-neutralizing V1-V2-directed antibody PG16. Nat Struct Mol Biol 2013;20:804-13.
- 56. Zhou T, Lynch RM, Chen L, Acharya P, Wu X, Doria-Rose NA, Joyce MG, Lingwood D, Soto C, Bailer RT, Ernandes MJ, Kong R, Longo NS, Louder MK, McKee K, O'Dell S, Schmidt SD, Tran L, Yang Z, Druz A, Luongo TS, Moquin S, Srivatsan S, Yang Y, Zhang B, Zheng A, Pancera M, Kirys T, Georgiev IS, Gindin T, Peng HP, Yang AS, Mullikin JC, Gray MD, Stamatatos L, Burton DR, Koff WC, Cohen MS, Haynes BF, Casazza JP, Connors M, Corti D, Lanzavecchia A, Sattentau QJ, Weiss RA, West AP, Jr., Bjorkman PJ, Scheid JF, Nussenzweig MC, Shapiro L, Mascola JR, Kwong PD. Structural Repertoire of HIV-1-Neutralizing Antibodies Targeting the CD4 Supersite in 14 Donors. Cell 2015;161:1280-92.
- 57. Chuang GY, Acharya P, Schmidt SD, Yang Y, Louder MK, Zhou T, Kwon YD, Pancera M, Bailer RT, Doria-Rose NA, Nussenzweig MC, Mascola JR, Kwong PD, Georgiev IS. Residue-level prediction of HIV-1 antibody epitopes based on neutralization of diverse viral strains. J Virol 2013;87:10047-58.
- 58. Derdeyn CA, Decker JM, Bibollet-Ruche F, Mokili JL, Muldoon M, Denham SA, Heil ML, Kasolo F, Musonda R, Hahn BH, Shaw GM, Korber BT, Allen S, Hunter E. Envelope-constrained neutralization-sensitive HIV-1 after heterosexual transmission. Science **2004**;303:2019-22.
- 59. Wilen CB, Parrish NF, Pfaff JM, Decker JM, Henning EA, Haim H, Petersen JE, Wojcechowskyj JA, Sodroski J, Haynes BF, Montefiori DC, Tilton JC, Shaw GM, Hahn BH, Doms RW. Phenotypic and immunologic comparison of clade B transmitted/founder and chronic HIV-1 envelope glycoproteins. J Virol 2011;85:8514-27.
- 60. UNAIDS. The GAP Report. 2014.

- 61. Padian NS, van der SA, Ramjee G, Chipato T, de Bruyn G, Blanchard K, Shiboski S, Montgomery ET, Fancher H, Cheng H, Rosenblum M, van der LM, Jewell N, Mcintyre J. Diaphragm and lubricant gel for prevention of HIV acquisition in southern African women: a randomised controlled trial. Lancet **2007**;370:251-61.
- 62. Celum C, Wald A, Hughes J, Sanchez J, reid S, Delany-Moretlwe S, Cowan F, Casapia M, Ortiz A, Fuchs J, Buchbinder S, Koblin B, Zwerski S, Rose S, Wang J, Corey L. Effect of aciclovir on HIV-1 acquisition in herpes simplex virus 2 seropositive women and men who have sex with men: a randomised, double-blind, placebo-controlled trial. Lancet 2008;371:2109-19.
- 63. Gray GE, Allen M, Moodie Z, Churchyard G, Bekker LG, Nchabeleng M, Mlisana K, Metch B, de BG, Latka MH, Roux S, Mathebula M, Naicker N, Ducar C, Carter DK, Puren A, Eaton N, McElrath MJ, Robertson M, Corey L, Kublin JG. Safety and efficacy of the HVTN 503/Phambili study of a clade-B-based HIV-1 vaccine in South Africa: a double-blind, randomised, placebo-controlled test-of-concept phase 2b study. Lancet Infect Dis 2011;11:507-15.
- 64. Gray GE, Moodie Z, Metch B, Gilbert PB, Bekker LG, Churchyard G, Nchabeleng M, Mlisana K, Laher F, Roux S, Mngadi K, Innes C, Mathebula M, Allen M, McElrath MJ, Robertson M, Kublin J, Corey L. Recombinant adenovirus type 5 HIV gag/pol/nef vaccine in South Africa: unblinded, long-term follow-up of the phase 2b HVTN 503/Phambili study. Lancet Infect Dis **2014**;14:388-96.
- 65. Abdool KQ, Abdool Karim SS, Frohlich JA, Grobler AC, Baxter C, Mansoor LE, Kharsany AB, Sibeko S, Mlisana KP, Omar Z, Gengiah TN, Maarschalk S, Arulappan N, Mlotshwa M, Morris L, Taylor D. Effectiveness and safety of tenofovir gel, an antiretroviral microbicide, for the prevention of HIV infection in women. Science 2010;329:1168-74.
- 66. Van Damme L, Corneli A, Ahmed K, Agot K, Lombaard J, Kapiga S, Malahleha M, Owino F, Manongi R, Onyango J, Temu L, Monedi MC, Mak'Oketch P, Makanda M, Reblin I, Makatu SE, Saylor L, Kiernan H, Kirkendale S, Wong C, Grant R, Kashuba A, Nanda K, Mandala J, Fransen K, Deese J, Crucitti T, Mastro TD, Taylor D. Preexposure prophylaxis for HIV infection among African women. N Engl J Med 2012;367:411-22.
- 67. NIAID. Daily-Use HIV Prevention Approaches Prove Ineffective Among Women in NIH Study. <a href="http://www.niaid.nih.gov/news/newsreleases/2013/Pages/VOICEwomen.aspx.3-4-2013">http://www.niaid.nih.gov/news/newsreleases/2013/Pages/VOICEwomen.aspx.3-4-2013</a>
- 68. World Medical Association. Ethical Principles for Medical Research Involving Human Subjects, Note of Clarification on Paragraph 29. **2002**.
- 69. Emanuel EJ, Wendler D, Grady C. What makes clinical research ethical? JAMA **2000**;283:2701-11.
- 70. Emanuel EJ, Miller FG. The ethics of placebo-controlled trials--a middle ground. N Engl J Med **2001**;345:915-9.
- 71. Ng CT, Jaworski JP, Jayaraman P, Sutton WF, Delio P, Kuller L, Anderson D, Landucci G, Richardson BA, Burton DR, Forthal DN, Haigwood NL. Passive neutralizing antibody

- controls SHIV viremia and enhances B cell responses in infant macaques. Nat Med **2010**;16:1117-9.
- 72. Lynch RM, Wong P, Tran L, O'Dell S, Nason MC, Li Y, Wu X, Mascola JR. HIV-1 fitness cost associated with escape from the VRC01 class of CD4 binding site neutralizing antibodies. J Virol **2015**;89:4201-13.
- 73. Gilbert PB, Grove D, Gabriel E, Huang Y, Gray G, Hammer SM, Buchbinder SP, Kublin J, Corey L, Self SG. A Sequential Phase 2b Trial Design for Evaluating Vaccine Efficacy and Immune Correlates for Multiple HIV Vaccine Regimens. Stat Commun Infect Dis **2011**;3.
- 74. Kamb ML, Fishbein M, Douglas JM, Jr., Rhodes F, Rogers J, Bolan G, Zenilman J, Hoxworth T, Malotte CK, Iatesta M, Kent C, Lentz A, Graziano S, Byers RH, Peterman TA. Efficacy of risk-reduction counseling to prevent human immunodeficiency virus and sexually transmitted diseases: a randomized controlled trial. Project RESPECT Study Group. JAMA 1998;280:1161-7.
- 75. Grant RM, Anderson PL, McMahan V, Liu A, Amico KR, Mehrotra M, Hosek S, Mosquera C, Casapia M, Montoya O, Buchbinder S, Veloso VG, Mayer K, Chariyalertsak S, Bekker LG, Kallas EG, Schechter M, Guanira J, Bushman L, Burns DN, Rooney JF, Glidden DV. Uptake of pre-exposure prophylaxis, sexual practices, and HIV incidence in men and transgender women who have sex with men: a cohort study. Lancet Infect Dis 2014;14:820-9.
- 76. McCormack S, Dunn DT, Desai M, Dolling DI, Gafos M, Gilson R, Sullivan AK, Clarke A, Reeves I, Schembri G, Mackie N, Bowman C, Lacey CJ, Apea V, Brady M, Fox J, Taylor S, Antonucci S, Khoo SH, Rooney J, Nardone A, Fisher M, McOwan A, Phillips AN, Johnson AM, Gazzard B, Gill ON. Pre-exposure prophylaxis to prevent the acquisition of HIV-1 infection (PROUD): effectiveness results from the pilot phase of a pragmatic open-label randomised trial. Lancet **2015**.
- 77. McCormack S, Dunn D. Pragmatic open-label randomized trial of preexposure prophylaxis: The PROUD study (Abstract 22LB). Conference on Retroviruses and Opportunistic Infections, Seattle, Washington (USA), February 23-26, **2015**
- 78. Molina J-M, Capitant C, Charreau I, Meyer L, Spire B, Pialoux G, Chidiac C, Delfraissy J-F, Tremblay C. On demand PrEP with Oral TDF-FTC in MSM: Results of the ANRS Ipergay trial (Abstract 23LB). Conference on Retroviruses and Opportunistic Infections, Seattle, Washington (USA), February 23-26, **2015**
- 79. Molina JM, Capitant C, Spire B, Pialoux G, Cotte L, Charreau I, Tremblay C, Le Gall JM, Cua E, Pasquet A, Raffi F, Pintado C, Chidiac C, Chas J, Charbonneau P, Delaugerre C, Suzan-Monti M, Loze B, Fonsart J, Peytavin G, Cheret A, Timsit J, Girard G, Lorente N, Preau M, Rooney JF, Wainberg MA, Thompson D, Rozenbaum W, Dore V, Marchand L, Simon MC, Etien N, Aboulker JP, Meyer L, Delfraissy JF. On-Demand Preexposure Prophylaxis in Men at High Risk for HIV-1 Infection. N Engl J Med 2015;373:2237-46.
- 80. Baeten JM, Donnell D, Ndase P, Mugo NR, Campbell JD, Wangisi J, Tappero JW, Bukusi EA, Cohen CR, Katabira E, Ronald A, Tumwesigye E, Were E, Fife KH, Kiarie J, Farquhar C, John-Stewart G, Kakia A, Odoyo J, Mucunguzi A, Nakku-Joloba E,

- Twesigye R, Ngure K, Apaka C, Tamooh H, Gabona F, Mujugira A, Panteleeff D, Thomas KK, Kidoguchi L, Krows M, Revall J, Morrison S, Haugen H, Emmanuel-Ogier M, Ondrejcek L, Coombs RW, Frenkel L, Hendrix C, Bumpus NN, Bangsberg D, Haberer JE, Stevens WS, Lingappa JR, Celum C. Antiretroviral prophylaxis for HIV prevention in heterosexual men and women. N Engl J Med **2012**;367:399-410.
- 81. Rees, H, Delany-Moretlwa, S, Baron, D, Lombard, C, Gray, G, Myers, L, Panchia, R, Schwartz, J, and Doncel, G. FACTS 001 Phase III trial of pericoital Tenofovir 1% gel for HIV prevention in women (Abstract 26LB).

  <a href="http://www.croiconference.org/sessions/facts-001-phase-iii-trial-pericoital-tenofovir-1-gel-hiv-prevention-women">http://www.croiconference.org/sessions/facts-001-phase-iii-trial-pericoital-tenofovir-1-gel-hiv-prevention-women</a>. 2015. Last accessed: 6-15-2015
- 82. Marrazzo JM, Ramjee G, Richardson BA, Gomez K, Mgodi N, Nair G, Palanee T, Nakabiito C, van der Straten A, Noguchi L, Hendrix CW, Dai JY, Ganesh S, Mkhize B, Taljaard M, Parikh UM, Piper J, Masse B, Grossman C, Rooney J, Schwartz JL, Watts H, Marzinke MA, Hillier SL, McGowan IM, Chirenje ZM. Tenofovir-based preexposure prophylaxis for HIV infection among African women. N Engl J Med 2015;372:509-18.
- 83. Hanscom B, Janes H, Guarino P, Huang Y, Brown E, Ying Q, Hammer S, Gilbert P, Donnell D. Is oral PrEP effective in preventing HIV in women? **2015**.
- 84. Patterson KB, Prince HA, Kraft E, Jenkins AJ, Shaheen NJ, Rooney JF, Cohen MS, Kashuba AD. Penetration of tenofovir and emtricitabine in mucosal tissues: implications for prevention of HIV-1 transmission. Sci Transl Med **2011**;3:112re4.
- 85. Cottrell ML, Yang KH, Prince HM, Sykes C, White N, Malone S, Dellon ES, Madanick RD, Shaheen NJ, Hudgens MG, Wulff J, Patterson KB, Nelson JA, Kashuba AD. A Translational Pharmacology Approach to Predicting HIV Pre-Exposure Prophylaxis Outcomes in Men and Women Using Tenofovir Disoproxil Fumarate+/-Emtricitabine. J Infect Dis 2016.
- 86. Centers for Disease Control and Prevention. Interim Guidance: Prexposure Prophylaxis for the Prevention of HIV Infection in Men Who Have Sex With Men.

  <a href="http://www.cdc.gov/mmwr/preview/mmwrhtml/mm6003a1.htm">http://www.cdc.gov/mmwr/preview/mmwrhtml/mm6003a1.htm</a>. 1-28-2011. Last accessed: 4-10-2015</a>
- 87. World Health Organization. Guidance on oral pre-exposure prophylaxis (PrEP) for serodiscordant couples, men and transgender women who have sex with men at high risk of HIV. July 2012. **2012**.
- 88. US Public Health Service. Preexposure Prophylaxis for the Prevention of HIV Infection in the United States 2014: A Clinical Practice Guideline. **2014**.
- 89. US Public Health Service. Preexposure Prophylaxis for the Preventon of HIV Infection in the United States 2014: Clinical Providers' Supplement. 2014. US Centers for Disease Control and Prevention.
- 90. WHO. Consolidated guidelines on the use of antiretroviral drugs for treating and preventing HIV infection. Recommendations for a public health approach.

  <a href="http://www.who.int/hiv/pub/guidelines/arv2013/download/en/">http://www.who.int/hiv/pub/guidelines/arv2013/download/en/</a>. 6-30-2013. Last accessed: 2-2-2015</a>

- 91. World Health Organization. Guideline on when to start antiretroviral therapy and on preexposure prophylaxis for HIV. **2015**.
- 92. Ponce R, Abad L, Amaravadi L, Gelzleichter T, Gore E, Green J, Gupta S, Herzyk D, Hurst C, Ivens IA, Kawabata T, Maier C, Mounho B, Rup B, Shankar G, Smith H, Thomas P, Wierda D. Immunogenicity of biologically-derived therapeutics: assessment and interpretation of nonclinical safety studies. Regul Toxicol Pharmacol **2009**;54:164-82.
- 93. Lobo ED, Hansen RJ, Balthasar JP. Antibody pharmacokinetics and pharmacodynamics. J Pharm Sci **2004**;93:2645-68.
- 94. Li Y, O'Dell S, Walker LM, Wu X, Guenaga J, Feng Y, Schmidt SD, McKee K, Louder MK, Ledgerwood JE, Graham BS, Haynes BF, Burton DR, Wyatt RT, Mascola JR. Mechanism of neutralization by the broadly neutralizing HIV-1 monoclonal antibody VRC01. J Virol 2011;85:8954-67.
- 95. Haynes BF, Fleming J, St Clair EW, Katinger H, Stiegler G, Kunert R, Robinson J, Scearce RM, Plonk K, Staats HF, Ortel TL, Liao HX, Alam SM. Cardiolipin polyspecific autoreactivity in two broadly neutralizing HIV-1 antibodies. Science **2005**;308:1906-8.
- 96. Mascola JR, Lewis MG, Stiegler G, Harris D, VanCott TC, Hayes D, Louder MK, Brown CR, Sapan CV, Frankel SS, Lu Y, Robb ML, Katinger H, Birx DL. Protection of Macaques against pathogenic simian/human immunodeficiency virus 89.6PD by passive transfer of neutralizing antibodies. J Virol **1999**;73:4009-18.
- 97. Mascola JR, Stiegler G, VanCott TC, Katinger H, Carpenter CB, Hanson CE, Beary H, Hayes D, Frankel SS, Birx DL, Lewis MG. Protection of macaques against vaginal transmission of a pathogenic HIV-1/SIV chimeric virus by passive infusion of neutralizing antibodies. Nat Med **2000**;6:207-10.
- 98. Mascola JR. Defining the protective antibody response for HIV-1. Curr Mol Med **2003**;3:209-16.
- 99. Nishimura Y, Igarashi T, Haigwood N, Sadjadpour R, Plishka RJ, Buckler-White A, Shibata R, Martin MA. Determination of a statistically valid neutralization titer in plasma that confers protection against simian-human immunodeficiency virus challenge following passive transfer of high-titered neutralizing antibodies. J Virol **2002**;76:2123-30.
- 100. Parren PW, Marx PA, Hessell AJ, Luckay A, Harouse J, Cheng-Mayer C, Moore JP, Burton DR. Antibody protects macaques against vaginal challenge with a pathogenic R5 simian/human immunodeficiency virus at serum levels giving complete neutralization in vitro. J Virol **2001**;75:8340-7.
- 101. Sadjadpour R, Donau OK, Shingai M, Buckler-White A, Kao S, Strebel K, Nishimura Y, Martin MA. Emergence of gp120 V3 variants confers neutralization resistance in an R5 simian-human immunodeficiency virus-infected macaque elite neutralizer that targets the N332 glycan of the human immunodeficiency virus type 1 envelope glycoprotein. J Virol 2013;87:8798-804.
- 102. Gautam R, Nishimura Y, Lee WR, Donau O, Buckler-White A, Shingai M, Sadjadpour R, Schmidt SD, LaBranche CC, Keele BF, Montefiori D, Mascola JR, Martin MA.

- Pathogenicity and mucosal transmissibility of the R5-tropic simian/human immunodeficiency virus SHIV(AD8) in rhesus macaques: implications for use in vaccine studies. J Virol **2012**;86:8516-26.
- 103. Shingai M, Donau OK, Plishka RJ, Buckler-White A, Mascola JR, Nabel GJ, Nason MC, Montefiori D, Moldt B, Poignard P, Diskin R, Bjorkman PJ, Eckhaus MA, Klein F, Mouquet H, Cetrulo Lorenzi JC, Gazumyan A, Burton DR, Nussenzweig MC, Martin MA, Nishimura Y. Passive transfer of modest titers of potent and broadly neutralizing anti-HIV monoclonal antibodies block SHIV infection in macaques. J Exp Med 2014;211:2061-74.
- 104. Hessell AJ, Hangartner L, Hunter M, Havenith CE, Beurskens FJ, Bakker JM, Lanigan CM, Landucci G, Forthal DN, Parren PW, Marx PA, Burton DR. Fc receptor but not complement binding is important in antibody protection against HIV. Nature **2007**;449:101-4.
- 105. Saunders KO, Pegu A, Georgiev IS, Zeng M, Joyce MG, Yang ZY, Ko SY, Chen X, Schmidt SD, Haase AT, Todd JP, Bao S, Kwong PD, Rao SS, Mascola JR, Nabel GJ. Sustained Delivery of a Broadly Neutralizing Antibody in Nonhuman Primates Confers Long-Term Protection against Simian/Human Immunodeficiency Virus Infection. J Virol 2015;89:5895-903.
- 106. Lynch RM, Boritz E, Coates EE, DeZure A, Madden P, Costner P, Enama ME, Plummer S, Holman L, Hendel CS, Gordon I, Casazza J, Conan-Cibotti M, Migueles SA, Tressler R, Bailer RT, McDermott A, Narpala S, O'Dell S, Wolf G, Lifson JD, Freemire BA, Gorelick RJ, Pandey JP, Mohan S, Chomont N, Fromentin R, Chun TW, Fauci AS, Schwartz RM, Koup RA, Douek DC, Hu Z, Capparelli E, Graham BS, Mascola JR, Ledgerwood JE. Virologic effects of broadly neutralizing antibody VRC01 administration during chronic HIV-1 infection. Sci Transl Med 2015;7:319ra206.
- 107. Ledgerwood JE, Coates EE, Yamshchikov G, Saunders JG, Holman L, Enama ME, DeZure A, Lynch RM, Gordon I, Plummer S, Hendel CS, Pegu A, Conan-Cibotti M, Sitar S, Bailer RT, Narpala S, McDermott A, Louder M, O'Dell S, Mohan S, Pandey JP, Schwartz RM, Hu Z, Koup RA, Capparelli E, Mascola JR, Graham BS. Safety, pharmacokinetics and neutralization of the broadly neutralizing HIV-1 human monoclonal antibody VRC01 in healthy adults. Clin Exp Immunol 2015;182:289-301.
- 108. Hansel TT, Kropshofer H, Singer T, Mitchell JA, George AJ. The safety and side effects of monoclonal antibodies. Nat Rev Drug Discov **2010**;9:325-38.
- Bugelski PJ, Achuthanandam R, Capocasale RJ, Treacy G, Bouman-Thio E. Monoclonal antibody-induced cytokine-release syndrome. Expert Rev Clin Immunol 2009;5:499-521.
- 110. Vogel WH. Infusion reactions: diagnosis, assessment, and management. Clin J Oncol Nurs **2010**;14:E10-E21.
- 111. Rosenbaum P. The consequences of adjustment for a concomitant variable that has been affected by the treatment. Journal of the Royal Statistical Society, Series A (General) **1984**;147:656-66.
- 112. Joffe MM, Greene T. Related causal frameworks for surrogate outcomes. Biometrics **2009**;65:530-8.
- 113. Follmann D. Augmented designs to assess immune response in vaccine trials. Biometrics **2006**;62:1161-9.
- 114. Gilbert PB, Hudgens MG. Evaluating candidate principal surrogate endpoints. Biometrics **2008**;64:1146-54.
- 115. Huang Y, Gilbert PB, Wolfson J. Design and estimation for evaluating principal surrogate markers in vaccine trials. Biometrics **2013**;69:301-9.
- 116. Rida W, Fast P, Hoff R, Fleming T. Intermediate-size trials for the evaluation of HIV vaccine candidates: a workshop summary. J Acquir Immune Defic Syndr Hum Retrovirol 1997;16:195-203.
- 117. Juraska, M, Grove, D, Yu, X, and Gilbert, PG. seqDesign: Simulation and Group Sequential Monitoring of Randomized Two-Stage Treatment Efficacy Trials with Time-to-Event Endpoints. R package version 1.1. <a href="http://CRAN.R-project.org?package=seqDesign">http://CRAN.R-project.org?package=seqDesign</a>. 4-27-2015. Last accessed: 5-15-2015
- 118. Thigpen MC, Kebaabetswe PM, Paxton LA, Smith DK, Rose CE, Segolodi TM, Henderson FL, Pathak SR, Soud FA, Chillag KL, Mutanhaurwa R, Chirwa LI, Kasonde M, Abebe D, Buliva E, Gvetadze RJ, Johnson S, Sukalac T, Thomas VT, Hart C, Johnson JA, Malotte CK, Hendrix CW, Brooks JT. Antiretroviral preexposure prophylaxis for heterosexual HIV transmission in Botswana. N Engl J Med 2012;367:423-34.
- 119. Miettinen O, Nurminen M. Comparative analysis of two rates. Stat Med 1985;4:213-26.
- 120. Freidlin B, Korn EL, Gray R. A general inefficacy interim monitoring rule for randomized clinical trials. Clin Trials **2010**;7:197-208.
- 121. Hammer SM, Sobieszczyk ME, Janes H, Karuna ST, Mulligan MJ, Grove D, Koblin BA, Buchbinder SP, Keefer MC, Tomaras GD, Frahm N, Hural J, Anude C, Graham BS, Enama ME, Adams E, DeJesus E, Novak RM, Frank I, Bentley C, Ramirez S, Fu R, Koup RA, Mascola JR, Nabel GJ, Montefiori DC, Kublin J, McElrath MJ, Corey L, Gilbert PB. Efficacy trial of a DNA/rAd5 HIV-1 preventive vaccine. N Engl J Med 2013;369:2083-92.
- 122. Schoenfeld DA. Sample-size formula for the proportional-hazards regression model. Biometrics **1983**;39:499-503.
- 123. Kalbfleisch J, Prentice R. The Statistical Analysis of Failure Time Data (Second Edition). John Wiley & Sons, Inc., **2002**.
- 124. Moore K, van der Laan M. Application of time-to-event methods in the assessment of safety in clinical trials. U. C. Berkeley Division of Biostatistics Working Paper Series, Paper 248. 2009.
- 125. van der Laan M, Rose S. Targeted Learning: Causal Inference for Observational and Experimental Data. Springer, **2011**.

- 126. Gilbert PB, Wei LJ, Kosorok MR, Clemens JD. Simultaneous inferences on the contrast of two hazard functions with censored observations. Biometrics **2002**;58:773-80.
- 127. Edlefsen P, Magaret C, Poon A, Matsen I, Eller L, Tovanabutra S, Chopera D, Labuschagne P, Warth C, Holzman T, Rossenkahm R, Abrahams M-R, Logan M, Anthony C, Botha G, Matten D, Nitayaphan S, Rono K, Sekiziyivu A, Ndabambi N, Travers S, Michael N, Williamson C, Robb N, Gilbert P. Systematic evaluation of HIV infection time and founder inferences using SGA and Illumina sequences . Keystone Symposia on Molecular and Cellular Biology, HIV Vaccines (X8), Olympic Valley, California, USA, March 20-24, 2016, **2016**
- 128. Gilbert P, Wang M, Wrin T, Petropoulos C, Gurwith M, Sinangil F, D'Souza P, Rodriguez-Chavez IR, DeCamp A, Giganti M, Berman PW, Self SG, Montefiori DC. Magnitude and breadth of a nonprotective neutralizing antibody response in an efficacy trial of a candidate HIV-1 gp120 vaccine. J Infect Dis **2010**;202:595-605.
- 129. Montefiori DC. Measuring HIV neutralization in a luciferase reporter gene assay. Methods Mol Biol **2009**;485:395-405.
- 130. Todd CA, Greene KM, Yu X, Ozaki DA, Gao H, Huang Y, Wang M, Li G, Brown R, Wood B, D'Souza MP, Gilbert P, Montefiori DC, Sarzotti-Kelsoe M. Development and implementation of an international proficiency testing program for a neutralizing antibody assay for HIV-1 in TZM-bl cells. J Immunol Methods **2012**;375:57-67.
- 131. Ozaki DA, Gao H, Todd CA, Greene KM, Montefiori DC, Sarzotti-Kelsoe M. International technology transfer of a GCLP-compliant HIV-1 neutralizing antibody assay for human clinical trials. PLoS ONE **2012**;7:e30963.
- 132. Fogel JM, Wang L, Parsons TL, Ou SS, Piwowar-Manning E, Chen Y, Mudhune VO, Hosseinipour MC, Kumwenda J, Hakim JG, Chariyalertsak S, Panchia R, Sanne I, Kumarasamy N, Grinsztejn B, Makhema J, Pilotto J, Santos BR, Mayer KH, McCauley M, Gamble T, Bumpus NN, Hendrix CW, Cohen MS, Eshleman SH. Undisclosed antiretroviral drug use in a multinational clinical trial (HIV Prevention Trials Network 052). J Infect Dis 2013;208:1624-8.
- 133. Marzinke MA, Clarke W, Wang L, Cummings V, Liu TY, Piwowar-Manning E, Breaud A, Griffith S, Buchbinder S, Shoptaw S, Del RC, Magnus M, Mannheimer S, Fields SD, Mayer KH, Wheeler DP, Koblin BA, Eshleman SH, Fogel JM. Nondisclosure of HIV status in a clinical trial setting: antiretroviral drug screening can help distinguish between newly diagnosed and previously diagnosed HIV infection. Clin Infect Dis 2014;58:117-20.
- 134. Castillo-Mancilla JR, Zheng JH, Rower JE, Meditz A, Gardner EM, Predhomme J, Fernandez C, Langness J, Kiser JJ, Bushman LR, Anderson PL. Tenofovir, emtricitabine, and tenofovir diphosphate in dried blood spots for determining recent and cumulative drug exposure. AIDS Res Hum Retroviruses **2013**;29:384-90.
- 135. Bushman LR, Kiser JJ, Rower JE, Klein B, Zheng JH, Ray ML, Anderson PL. Determination of nucleoside analog mono-, di-, and tri-phosphates in cellular matrix by solid phase extraction and ultra-sensitive LC-MS/MS detection. J Pharm Biomed Anal **2011**;56:390-401.

- 136. UNAIDS. Ethical considerations in biomedical HIV prevention trials. 2007.
- 137. The National Commission for the Protection of Human Subjects of Biomedical and Behavioral Research. The Belmont Report: Ethical Principles and Guidelines for the Protection of Human Subjects of Research. 1979.
- 138. Council for International Organizations of Medical Sciences (CIOMS). International ethical guidelines for biomedical research involving human subjects. Bull Med Ethics **2002**;17-23.
- 139. UNAIDS/JC1853E (Second edition J2. Good participatory practice: Guidelines for biomedical HIV prevention trials. 2011.

### Appendix A Sample informed consent form

Title: A phase 2b study to evaluate the safety and efficacy of VRC01 broadly neutralizing monoclonal antibody in reducing acquisition of HIV-1 infection in women in sub-Saharan Africa

Protocol number: HVTN 703/HPTN 081, The AMP Study

Site: [Insert site name]

Thank you for your interest in our research study. Please read this consent form or ask someone to read it to you. If you decide to join the study, we will ask you to sign or make your mark on this form. We will offer you a copy to keep. We will ask you questions to see if we have explained everything clearly. You can also ask us questions about the study.

Research is not the same as treatment or medical care. The purpose of a research study is to answer scientific questions.

#### About the study

The HIV Vaccine Trials Network (HVTN), the HIV Prevention Trials Network (HPTN), and [Insert site name] are doing a study to test the antibody called VRC01 against HIV. HIV is the virus that causes AIDS. Antibodies are one of the natural ways the body fights infection. Researchers can also make antibodies in laboratories and give them to people intravenously (with an IV). We will tell you more about this procedure below. This has been done successfully to prevent or treat some other health problems, such as a virus that causes respiratory infections in infants.

About 1900 people will take part in this study at multiple sites in Africa. The researcher in charge of this study at this clinic is [Insert name of site PI]. The US National Institutes of Health (NIH) is paying for the study.

In addition, a similar study will be done with 2700 men and transgender people who have sex with men and transgender people in the North America, South America, and Switzerland.

#### 1. We are doing this study to answer several questions.

- Is the antibody safe to give to people?
- Are people able to take the antibody without becoming too uncomfortable?
- Does the antibody lower people's chances of getting infected with HIV?
- If the antibody does lower people's chances of getting infected with HIV, how much of it is needed to provide protection from HIV?

#### 2. The antibody cannot give you HIV.

It is impossible for the antibody to give you HIV. Also, it cannot cause you to give HIV to someone else. However, we do not know if the antibody will decrease, increase, or not change your chance of becoming infected with HIV if you are exposed to the virus.

#### 3. The antibody is experimental.

The antibody being tested is called VRC-HIVMAB060-00-AB. It is an antibody against the HIV virus. From here on, we will call it VRC01 or the antibody. It is an experimental product. That means we do not know whether the antibody will be safe to use in people, or whether it will work to prevent HIV infection. This antibody is used only in research studies.

VRC01 was developed by the Vaccine Research Center at the US National Institutes of Health (NIH).

In laboratory and animal studies, VRC01 attached to and prevented infection by many strains of HIV viruses from around the world. We do not know if antibodies can prevent HIV infection when they are given to people. This study is designed to help answer that question. At this time there are no plans to make VRC01 for sale.

*Risks of VRC01 antibody:* 

As of April 2017, VRC01 has been given to people in 12 clinical studies in the United States, Peru, Brazil, Switzerland, and in sub-Saharan Africa. In these studies, more than 1800 adults and 33 infants have gotten VRC01 or a placebo (a liquid with no antibody in it).

Many of these studies are still going on and we don't know which people got VRC01 and which got a placebo. In early trials, more than 100 people got VRC01 and it did not make them too uncomfortable or cause serious health problems. After receiving the antibody, most people said that they had mild pain, itching, or redness where the antibody was given to them. Of these people, some said they felt like they had the flu after getting the antibody, but that this feeling lasted a few hours at most.

In a previous study, one person who got a VRC01 injection had a rash. One person had a brief fainting spell several hours after getting a VRC01 infusion. To be safe, no more injections or infusions were given to these people. Some participants had mild body discomfort, muscle pain, or joint pain after getting the VRC01 antibody.

VRC01 may have other side effects that we do not know about yet.

General risks of antibodies:

Antibodies that are different from VRC01 have been given to people for other illnesses. With those antibodies most side effects happen within the first 24 hours. Those antibodies have caused fever, chills, shaking, nausea, vomiting, pain, headache, dizziness, trouble breathing, high or low blood pressure, itchiness, rash, hives, lip or face swelling, diarrhea, racing heartbeat or chest pain.

Rarely, some antibodies have caused serious reactions. These reactions may be life-threatening. Please tell us if you have ever had any of the following reactions.

- One type of serious reaction, called anaphylaxis, may occur soon after getting an antibody. It includes difficulty breathing possibly leading to low blood oxygen, low blood pressure, hives or rash, and swelling in the mouth and face.
- A second type of serious reaction, called serum sickness, may occur several days to 3 weeks after getting an antibody. It includes hives or a rash, fever, big lymph nodes, muscle and joint pains, chest discomfort and shortness of breath.

Rarely, antibodies licensed for treatment of other diseases have been linked to a blood disorder that interferes with blood clotting, to cancer, to damage to the heart muscle, and to the body's immune system attacking healthy cells.

These rare side effects and reactions have not been seen in other studies with the VRC01 antibody.

When antibodies are given to a person by IV they do not last in the body more than a few months. Any antibody given to you in this study should be gone from your body several months after your last dose.

### Joining the study

#### 4. It is completely up to you whether or not to join the study.

Take your time in deciding. If it helps, talk to people you trust, such as your doctor, friends or family. If you decide not to join this study, or if you leave it after you have joined, your other care at this clinic and the benefits or rights you would normally have will not be affected.

If you join this study, you may not be allowed to join some other kinds of HIV prevention studies now or in the future. You cannot be in this study while you are in another study where you get a study product. Also during the study, you should not donate blood or tissue.

If you choose not to join this study, you may be able to join another study.

Site: Remove item 5 if you use a separate screening consent that covers these procedures.

#### 5. If you want to join the study, we will screen you to see if you are eligible.

Screening involves a physical exam, HIV test and health history. A physical exam may include, but is not limited to:

- Checking your weight, temperature and blood pressure
- Looking in your mouth and throat
- Listening to your heart and lungs
- Feeling your abdomen (stomach and liver)
- Checking your veins to see how easy it might be to start an IV

We will also do blood and urine tests. These tests tell us about some aspects of your health, such as how healthy your kidneys, liver, and immune system are. We will also ask you about medications you are taking. We will ask you about behaviors that might put you at risk for getting HIV. If you could become pregnant, we will test you for pregnancy. If you have had your uterus or ovaries removed (a hysterectomy or oophorectomy), verified by medical records, you are not required to have a pregnancy test.

We will review the screening results with you. The screening results may show you are not eligible to join the study, even if you want to.

(Sites: adapt the following section so it is applicable to the care available at your site)

6. If we find that you have a health problem during screening or during the study, we will tell you about the care that we can give here for free.

For the care that we cannot give, we will explain how we will help you get care elsewhere.

For health problems that are unrelated to the study, we will not pay for care.

7. If you could become pregnant, you must agree to use birth control to join this study.

Site: If you want to include Appendix B, Approved birth control methods (for sample informed consent form), in this consent form, paste it below and delete paragraph below.

You should not become pregnant during the study because we do not know how the antibody could affect the developing baby. You must agree to use effective birth control from 21 days before you first receive the antibody until your last scheduled clinic visit (about 13/4 years after your first IV). We will talk to you

about effective birth control methods. They are listed on a handout that we will give to you.

#### Being in the study

If you meet the study requirements and want to join, here is what will happen:

## 8. You will come to the clinic for scheduled visits about [#] times over about 2 years.

The study will require [#] visits. That is 1 visit every 4 weeks for about the first 1½ years and then about every 2 months after that. You may have to come for more visits if you have a lab or health issue.

Visits can last from about [#] minutes to [#] hours. The IV procedure can take about 15 minutes to an hour.

We may contact you after the main study ends (for example, to tell you about the study results).

# 9. We will give you [Site: Insert compensation] for each study visit you complete.

This amount is to cover the costs of [Site: Insert text]

Site: Insert any costs to participants (eg, birth control costs for participants who could become pregnant).

You do not have to pay anything to be in this study.

#### 10. We will give you either the antibody or a placebo.

Not everyone in this study will get the VRC01 antibody. Some people will get a placebo, a liquid that does not contain any antibody. We will compare the results from people who got the placebo with results from people who got the VRC01 antibody. In this study, the placebo is sterile salt water, which is found naturally in the body.

There are three groups in this study. One group will get a lower dose of the VRC01 antibody, one group will get a higher dose, and one group will get the placebo. The high and low doses of the antibody will be adjusted for your body weight. We will weigh you to determine the amount you will get.

Overall, if you join this study, you have a 2-in-3 chance of getting the study antibody.

Site: Modify the randomization metaphor in the next sentence as appropriate to your local culture.

Whether you get the low dose of the antibody, the high dose of the antibody, or the placebo is completely random, like flipping a coin.

We have no say in whether you get the antibody or the placebo. If you get the antibody, we have no say in which dose you get. We will not know what you are getting, and neither will you. Only the pharmacist at this clinic will have this information while the study is going on.

You will have to wait until everyone completes their final study visits to find out whether you got the antibody or the placebo. This could be up to about 5 years. But, if you have a serious medical problem and need to know what you got before the end of the study, we can tell you.

If it is found to be effective, there are no plans to give the antibody to participants after the study. Instead, we will use what is learned in this study to determine if the antibody would be useful to prevent HIV, how the antibody could be improved, and how to produce it for wide public use.

#### 11. We will give you the antibody or placebo on a schedule.

You will get the VRC01 antibody or the placebo during the study by IV, also known as a drip. To get an IV, a needle is used to place a small plastic tube into a vein in your arm. The tube is connected to a small bag of fluid that contains the antibody or placebo. An IV pump controls how fast the fluid drips from the bag, through the tube, and into your vein. There will be 10 IV procedures, one IV every 8 weeks. Other study visits will not include IVs.

| | Infusion schedule | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 6 month | ıs | | 1 yea | ar | | |
| | | | | | | Wee | ks after f | irst IV | | | <u> </u> |
| Group | Dose | First<br>IV | Wk<br>8 | Wk<br>16 | Wk<br>24 | Wk<br>32 | Wk<br>40 | Wk<br>48 | Wk<br>56 | Wk<br>64 | Wk<br>72 |
| Group<br>1 | Lower dose<br>VRC01 | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ |
| Group<br>2 | Higher dose<br>VRC01 | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ |
| Group<br>3 | Placebo | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ |

You will have to wait in the clinic for about 30 minutes after the first IV to see if there are any problems. You probably will not have to wait after the IVs at the rest of the IV visits. After each IV visit, for that night and for three more days, you will be asked to keep track of how you feel. To help you do this, we can give you tools and show you how to use them. We will ask you the ways we can contact you. We will contact you about 3 days after each IV visit to ask how you have been feeling. Contact the clinic staff if you have any concerns after getting an infusion. If you have a problem, we will continue to check on you until it goes away.

#### 12. In addition to giving you the antibody or placebo, we will:

- Do regular HIV testing, as well as counseling on your results and on how to avoid getting HIV;
- Do physical exams;
- Do pregnancy tests if you could become pregnant;
- Ask questions about your health, including medications you may be taking;
- Ask questions about any personal problems or benefits you may have from being in the study; and
- Take urine and blood samples.

When we take blood, the amount will depend on the lab tests we need to do. It will be some amount between 30 mL and 180 mL (6 teaspoons to <sup>3</sup>/<sub>4</sub> cup). Your body will make new blood to replace the blood we take out.

Site: You may want to add a sentence to the end of the previous paragraph contextualizing the blood volumes described (eg, "To compare, people who donate blood in the US can give a total of about 500 mL in an 8-week period."). Modify the example for cultural relevance and alter blood volumes as necessary.

Site: Insert the **first** table in Appendix D, Tables of procedures (for informed consent form) in this section or distribute it as a separate sheet if it is helpful to your study participants. You are not required to do either.

We will be looking for side effects.

About every six months we will do a blood test for syphilis and will test your urine or a cervical/vaginal swab for gonorrhea and chlamydia. At these times we will also test you for Trichomonas using a cervical/vaginal swab. We will explain what each of these infections is. If the tests show that you have an infection, we will provide counseling and will help you get treatment. This study cannot pay for that treatment. [Site: Revise preceding sentence if you provide or pay for STI treatment.]

We will review the results of the procedures and tests with you at your next visit, or sooner if necessary. If any of the results are important to your health, we will tell you.

#### 13. We will test your samples for this study.

We will send your samples (without your name) to labs approved by the HVTN and the HPTN for this study. These labs are located in the United States and South Africa. The samples will be tested to:

- measure how much antibody is in your blood,
- see how your immune system responds to the antibody, and
- see if there is antiretroviral medicine (also called ART/ARV) in your blood.

Researchers may also do genetic testing related to this study on your samples. Your genes are passed to you from your birth parents. They affect how you look and how your body works. The differences in people's genes can help explain why some people get a disease while others do not. These types of genetic tests involve only some of your genes, not all of your genes (your genome). The researchers will study the genes related to the immune system and HIV and those that affect how people get HIV.

If you become HIV infected, the researchers may look at all of the genes of the virus found in your samples. The researchers will use this information to learn more about HIV and the antibody.

In some cases, researchers may take cells from your samples and grow more of them over time, so that they can continue to contribute to this study.

Tests done on your samples are for research purposes only. The labs will not give the results to you or this clinic, and the results will not become part of your study record.

When your samples are no longer needed for this study, the HVTN will continue to store them.

Site: Delete next section if using separate consent for use of samples and information in other studies

14. When samples are no longer needed for this study, the study sponsors want to keep them for use in other studies by HVTN, HPTN, or other researchers. We will call these "extra samples."

This section gives you information so you can decide if you want your extra samples and information used in other studies. You will mark your decision at the end of the form. If you have any questions, please ask.

Do I have to agree? No. You are free to say yes or no, or to change your mind after you sign this form. At your request, we will destroy all extra samples that we have. Your decision will not affect your being in this study or have any negative consequences here.

Where are the samples stored? Extra samples are stored in a secure central place called a repository. Your samples will be stored in the HVTN repository in South Africa.

How long will the samples be stored? There is no limit on how long your extra samples will be stored. [Site: insert limits if your regulatory authority imposes them.]

Will I be paid for the use of my samples? No. Also, a researcher may make a new scientific discovery or product based on the use of your samples. If this happens, there is no plan to share any money with you. The researcher is not likely to ever know who you are.

Will I benefit from allowing my samples to be used in other studies? Probably not. Results from these other studies are not given to you, this clinic, or your doctor. They are not needed for your medical care. They are not part of your medical record. The studies are only being done for research purposes.

Will the HVTN or HPTN sell my samples and information? No, but the HVTN and HPTN may share your samples with other researchers. Once we share your samples and information, we will not be able to get them back.

How do other researchers get my samples and information? When a researcher wants to use your samples and/or information, their research plan must be approved by the HVTN and HPTN. Also, the researcher's institutional review board (IRB) or ethics committee (EC) will review their plan. [Site: If review by your institution's IRB/EC/RE is also required, insert a sentence stating this.] IRBs/ECs protect the rights and well-being of people in research. If the research plan is approved, the HVTN and HPTN will send your samples to the researcher's location.

What information is shared with other researchers? The samples and limited information will be labeled with a code number. Your name will not be part of the information. However, some information that we share may be personal, such as your race, ethnicity, gender, health information from the study, and HIV status. We may share information about the study product you received and how your body responded to the study product.

What kind of studies might be done with my extra samples and information? The studies will be related to HIV prevention or infection, the immune system, and other diseases.

Researchers may also do genetic testing on your samples.

If you become HIV infected, the researchers may look at all of the genes of the virus found in your samples. The researchers will use this information to learn more about HIV and the study product(s).

In some cases, researchers may take cells from your samples and grow more of them over time, so that they can continue to contribute to this study.

If you agree, your samples could also be used for genome wide studies. In these studies, researchers will look at all of your genes (your genome). The researchers compare the genomes of many people, looking for common patterns of genes that could help them understand diseases. The researchers may put the information from the genome-wide studies into a protected database so that other researchers can access it. Usually, no one would be able to look at your genome and link it to you as a person. However, if another database exists that also has information on your genome and your name, someone might be able to compare the databases and identify you. If others found out, it could lead to discrimination or other problems. The risk of this is very small.

Who will have access to my information in studies using my extra samples?

#### People who may see your information are:

- Researchers who use your stored samples and limited information for other research
- Government agencies that fund or monitor the research using your samples or information
- Any regulatory agency that reviews clinical trials
- The researcher's Institutional Review Board or Ethics Committee
- The people who work with the researcher

All of these people will do their best to protect your information. The results of any new studies that use your extra samples or information may be published. No publication will use your name or identify you personally.

#### 15. We will counsel you on reducing your risk for HIV infection.

We will ask you personal questions about your HIV risk factors such as sexual behavior and drug use. We will provide you with condoms and lubricant. We will talk with you about ways of lowering your risk of getting HIV. We will help you develop a risk reduction plan. Some topics we may discuss include:

- What you think causes risky behavior for you, and
- Ways to avoid getting HIV or giving it to someone else

[Site: Adjust the language in this paragraph about PrEP provision to meet local availability. The current text reflects the situation in the Republic of South Africa.] These methods may include not having sex, using condoms, or other behavior changes. We will talk about new methods of HIV prevention as they become available. These methods may include the use of anti-HIV drugs taken every day to prevent HIV. This is called pre-exposure prophylaxis or PrEP. In the

past few months a combination of two anti-HIV drugs (TDF/FTC) has been licensed in South Africa and Kenya for use to prevent HIV infection in people at high risk. Studies in women have shown this drug combination can reduce the risk of getting HIV when it is taken every day. The drug combination is not always effective and HIV infections may happen, especially if the medicine is not taken every day. This drug combination is available in the private health sector by prescription from a doctor. The Ministry of Health in South Africa is starting several programs called "demonstration projects" that provide this drug combination to people free of charge. We can refer you to the nearest of these programs if you are interested.

In this study, we will look at how many participants use PrEP. We will also try to find out if using PrEP has any effect on how VRC01 works.

[Site: If you prefer to use Appendix E, Sample consent form for participants with HIV infection at enrollment or during the study, include the following section and delete the two succeeding sections that are highlighted in green. If you prefer not to use Appendix E, delete the following section and INCLUDE the two sections highlighted in green.]

# 16. If you are HIV infected when you enroll or become infected during the study, we will help you get care and support.

We will test your blood for HIV before your first IV and during the study. Each time, it will take a few days to complete the tests. If you are infected with HIV, you cannot stay in the study for its whole length. If that happens, we will tell you as soon as possible. We will also ask you to come to the clinic for 2-5 more visits. We will tell you more about what will happen at these visits in another form.

## 17. If you are found to have been HIV-1 infected when you enrolled, or if you have HIV-2 infection:

If you are found to have been HIV infected when you enrolled, you were already infected with HIV before you got the antibody or placebo. It takes a few days to complete the tests to see if you have HIV, so your infection was not found until after you got your first IV.

#### HIV-2 is a rare kind of HIV, most often found in West Africa.

We will counsel you about your HIV infection, talk with you about ways to avoid transmission and about telling your partner(s).

We will ask you to come to the clinic for 2 more visits within about 6 months of your diagnosis. At these visits, we will:

- Ask questions about your health;
- Do physical exams based on your complaints or symptoms;

- Ask questions about your risk of infecting others with HIV, including sexual behavior and drug use;
- Counsel you on ways to avoid transmitting HIV to other people;
- Collect blood samples (between 30 and 45 mL, or about 2 to 3 tablespoons, at each visit); and
- Do pregnancy tests if you could become pregnant;
- Ask questions about any personal problems or benefits you may have from participating in the study.

[Site: Insert the **second** table in Appendix D, Tables of procedures (for informed consent form) in this section or distribute it as a separate sheet if it is helpful to your study participants. You are not required to do either.]

#### 18. If you got infected with HIV-1 during the study:

If you became infected with HIV-1, we will counsel you about your HIV infection, talk with you about ways to avoid transmission and about telling your partner(s). You will not get any more IVs. We will ask you to come in for 5 more visits within about 6 months of your diagnosis. At these visits, we will:

- Ask questions about your health;
- Do physical exams based on your complaints or symptoms;
- Ask questions about your risk of infecting others with HIV, including sexual behavior and drug use;
- Counsel you on ways to avoid transmitting HIV to other people;
- Collect blood samples (between 70 mL and 130 mL, about ½ to ½ cup, at each visit); and
- Ask questions about any personal problems or benefits you may have from participating in the study.

[Site: Insert the **third** table in Appendix D, Tables of procedures (for informed consent form) in this section or distribute it as a separate sheet if it is helpful to your study participants. You are not required to do either.]

19. If you stop getting IVs for reasons other than HIV infection, we may encourage you to stay in the study.

We will ask you to come in for study visits about every 3-4 months until 104 weeks (2 years) after your first infusion. That is how long you would be in the

study if you got all the infusions on schedule. Because you got some IVs, we want to keep track of your health. How many visits you will have will depend on when you stopped getting IVs. At these visits we will:

Ask questions about your health, including medications you may be taking;

- Do physical exams based on your complaints or side effects;
- Do regular HIV testing, as well as counseling on your results and on how to avoid getting HIV;
- Ask questions about any personal problems or benefits you may have from participating in the study;
- Do pregnancy tests if you could become pregnant;
- Collect urine samples; and
- Collect blood samples (between 70 mL and 120 mL, about ½ to ½ cup, at each visit).

[Site: Insert the **last** table in Appendix D, Tables of procedures (for informed consent form) in this section or distribute it as a separate sheet if it is helpful to your study participants. You are not required to do either.]

20. We may stop your IVs and take you out of the study at any time. We may do this even if you want to stay in the study and even if you were scheduled for more IVs.

This may happen if:

- we learn that you were enrolled in the study in error,
- you are unable to follow instructions,
- we think that staying in the study might harm you,
- you enroll in a different research study where you get another study product, or
- the study is stopped for any reason.

If we take you out of the study, we will ask you to come back to the clinic one last time for a physical exam, and we may ask to take some blood and urine samples. We will also ask about any personal problems or benefits you have experienced from being in the study.

#### 21. We will stop your IVs if you become pregnant during the study.

We will encourage you to stay in the study if you choose. We will discuss your study options with you. If you leave the study while you are still pregnant, we will contact you after your due date to ask some questions about your pregnancy and delivery.

#### 22. We will do our best to protect your private information.

Your study records and samples will be kept in a secure location. We will label all of your samples and most of your records with a code number, not your name or other personal information. However, it is possible to identify you, if necessary. We will not share your name with the lab that does the tests on your samples, or with anyone else who does not need to know your name.

Clinic staff will have access to your study records. Your records may also be reviewed by groups who watch over this study to see that we are protecting your rights, keeping you safe, and following the study plan. These groups include:

- The US National Institutes of Health, people who work for them, its study monitors, and its chosen South African representatives,
- The US Food and Drug Administration,
- Any regulatory agency that reviews clinical trials
- [Insert name of local IRB/EC],
- [Insert name of local and/or national regulatory authority as appropriate],
- The HVTN and HPTN and people who work for them,
- The US National Institutes for Allergy and Infectious Diseases Data and Safety Monitoring Board, and
- The US Office for Human Research Protections.

All reviewers will take steps to keep your records private.

We cannot guarantee absolute privacy. At this clinic, we have to report the following information:

Site: Include any public health or legal reporting requirements. Bulleted examples should include all appropriate cases (reportable communicable disease, risk of harm to self or others, etc.).

• [Item 1]

- [Item 2]
- [Item 3]

The results of this study may be published. No publication will use your name or identify you personally.

We may share information from the study with other researchers. We will not share your name or information that can identify you.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

#### Other Risks

#### 23. There are other risks to being in this study.

This section describes the other risks and restrictions we know about. There may also be unknown risks, even serious ones. We will tell you if we learn anything new that may affect your willingness to stay in the study.

Risks of taking blood:

Taking blood can cause bruising, pain, fainting, soreness, redness, swelling, itching, a sore, bleeding, and (rarely) muscle damage or infection where the needle was inserted. Taking blood can cause a low blood cell count (anemia), making you feel tired.

*Risks of the IV procedures:* 

Getting an IV may cause stinging, discomfort, pain, soreness, redness, bruising, itching, rash, and swelling where the needle goes into the skin. Rarely, needle sticks can result in infections.

*Personal problems/discrimination:* 

Some people who join HVTN or HPTN studies report personal problems or discrimination because of joining an HIV prevention study. Family or friends may worry, get upset or angry, or assume that you are infected with HIV or at high risk and treat you unfairly as a result. Rarely, a person has lost a job because the study took too much time away from work, or because their employer thought they had HIV.

HIV testing

HIV antibody tests are the usual way to test for HIV infections. Although 2 out of 3 people in this study will get an HIV antibody, we do not expect them to test positive on HIV antibody tests. We have used several common HIV antibody tests to test samples of blood containing the VRC01 antibody and none of them detected the antibody.

Although it has not been seen so far, getting VRC01 may cause common HIV antibody tests to show that someone is HIV-negative, even if they are actually infected.

To be absolutely safe we ask you to get HIV tests only at this clinic during the study. Our tests can always detect true HIV infection. They can also tell if someone is really not HIV infected. Since the antibodies do not last long in the body, we do not expect you to have any problems with HIV testing after the study ends.

#### Embarrassment/anxiety:

You may feel embarrassed when we ask about your HIV risks, such as having sex and using drugs. Also, waiting for your HIV test results or other health test results could make you feel anxious. You could feel worried if your test results show that you are infected with HIV. If you feel embarrassed or anxious, please tell us and we will try to help you.

#### Risks of disclosure of your personal information:

We will take several steps to protect your personal information. Although the risk is very low, it is possible that your personal information could be given to someone who should not have it. If that happened, you could face discrimination, stress, and embarrassment. We can tell you more about how we will protect your personal information if you would like it.

#### Risks of genetic testing:

The genetic testing could show you may be at risk for certain diseases. If others found out, it could lead to discrimination or other problems. However, it is almost impossible for you or others to know your test results from the genetic testing. The results are not part of your study records and are not given to you.

#### Unknown risks:

We do not know if the antibody will increase, decrease, or not change your risk of becoming infected with HIV if exposed.

If we find that you were already HIV infected when you got the antibody, we do not know how the antibody will affect your HIV disease. We also do not know how having gotten it will affect your HIV-related lab results.

If you get infected with HIV during the study, we do not know how the antibody might affect the course of your HIV disease.

If you become pregnant while you still have VRC01 in your body, we don't know if it could be passed to your baby. We do not know how the antibody will affect a pregnant participant or a developing baby.

#### **Benefits**

#### 24. The study may not benefit you.

Since we do not know if the antibody can prevent HIV infection in people, you should not expect any benefit from getting the antibody in this study. However, being in the study might still help you in some ways. The counseling that you get as part of the study may help you avoid getting HIV. The lab tests and physical exams that you get while in this study might detect health problems you don't yet know about.

This study may show us that the VRC01 antibody can prevent HIV and the study results may also help in the search for methods to prevent HIV. However, if the VRC01 antibody later becomes approved and sold or leads to an HIV prevention method, there are no plans to share any money with you.

#### Your rights and responsibilities

#### 25. If you join the study, you have rights and responsibilities.

You have many rights that we will respect. You also have responsibilities. We list these in the Participant's Bill of Rights and Responsibilities. We will give you a copy of it.

### Leaving the study

#### 26. Tell us if you decide to leave the study.

You are free to leave the study at any time and for any reason. Your care at this clinic and your legal rights will not be affected, but it is important for you to let us know.

If you decide to leave the study, we will ask you to come back to the clinic one last time for a physical exam, and we may ask to take some blood and urine samples. We will also ask about any personal problems or benefits you have experienced from being in the study. We believe these steps are important to protecting your health, but it is up to you whether to complete them.

#### **Injuries**

Sites: Do not make changes to the following section without obtaining approval from HVTN Regulatory Affairs at vtn.core.reg@hvtn.org.

#### 27. If you get sick or injured during the study, contact us immediately.

Your health is important to us. (Sites: adjust the following 2 sentences if applicable to the care available at your site) We will tell you about the care that we can give here. For the care that we cannot provide, we will explain how we will help you get care elsewhere.

If you become sick or injured in this study, there is a process to decide if it is related to the VRC01 antibody and/or study procedures. If it is, we call it a study-related injury.

Next paragraph for all sites except in Zimbabwe.

(Sites: adjust the language in this paragraph so it is applicable to your site. Note: Insurance is purchased for all African countries except Zimbabwe. The ABPI guidelines may only apply to South Africa and Mozambique.)

In this study, our clinic has insurance to cover your medical treatment in the case of a study-related injury. The insurance will follow the Association of the British Pharmaceutical Industry guidelines for payment of study-related injury. We can give you a copy of these guidelines. In rare cases, the insurance funds may not be enough. If needed, the HVTN and HPTN have limited funds to pay medical costs for study-related injuries that they determine are reasonable. (Sites: insert locale-appropriate medical insurance language in the following sentence) If the injury is not study related, then you and your health insurance will be responsible for treatment costs.

Some injuries are not physical. For example, you might be harmed emotionally by being in an HIV prevention study. Or you might lose wages because you cannot go to work. However, there are no funds to pay for these kinds of injuries, even if they are study related.

You may disagree with the decision about whether your injury is study related. If you wish, independent experts will be asked to review the decision. You always have the right to use the court system if you are not satisfied.

#### Questions

28. If you have questions or problems at any time during your participation in this study, use the following important contacts.

If you have questions about this study, contact [name and telephone number of the investigator or other study staff].

If you have any symptoms that you think may be related to this study, contact [name and telephone number of the investigator or other study staff].

If you have questions about your rights as a research participant, or problems or concerns about how you are being treated in this study, contact [name/title/phone of person on IRB or other appropriate organization].

If you want to leave this study, contact [name and telephone number of the investigator or other study staff].

#### South African sites: Include the following:

If you have questions about this trial you should first discuss them with your doctor or the ethics committee (contact details as provided on this form). After you have consulted your doctor or the ethics committee and if they have not provided you with answers to your satisfaction, you should write to the South African Medicines Control Council (MCC) at:

The Registrar of Medicines Medicines Control Council Department of Health Private Bag X828 PRETORIA 0001

Fax: (012) 395 9201

e-mail: gouwsj@health.gov.za

#### Your permissions and signature

Site: Delete this section if using a separate consent for use of samples and information in other studies.

29. In Section 14 of this form, we told you about possible other uses of your extra samples and limited information, outside this study. Please choose only one of the options below and write your initials or make your mark in the box next to it. Whatever you choose, the HVTN and HPTN keep track of your decision about how your samples and information can be used.

| other studie | extra samples combined with limite<br>s related to HIV prevention, the im-<br>nis may include genetic testing and | mune system, | and other |
|---|---|---|---|
| OR | | | |
| | e option above <i>and</i> also to allow mrmation to be used in genome wide | • | es combined with |
| OR | | | |
| | ow my extra samples to be used in a<br>g genetic testing, growing more of t | • | |
| | is study, you will need to sign or nor make your mark on this cons | • | |
| • You have read this | consent form, or someone has read | it to you. | |
| | nderstand what the study is about a<br>u understand what the possible risk | | |
| You have had your | questions answered and know that | you can ask n | nore. |
| <ul> <li>You agree to join the</li> </ul> | nis study. | | |
| | giving up any of your rights by sig | ning this cons | sent form. |
| Participant's name (print) | Participant's signature or mark | Date | Time |
| Clinic staff conducting consent discussion (print) | Clinic staff signature | Date | Time |
| For participants who ar signature block below: | re unable to read or write, a witness | should compl | ete the |
| Witness's name (print) | Witness's signature | Date | Time |

\*Witness is impartial and was present for the consent process.

# Appendix B Approved birth control methods (for sample informed consent form)

You should not become pregnant during the study because we do not know how the study antibody could affect the developing baby.

If you were born female and are sexually active in a way that could lead you to get pregnant, you must agree to use effective birth control from 21 days before your first IV until your last scheduled clinic visit (about 2 years after your first IV). You should not become pregnant during the study because we do not know how the antibody could affect the developing baby.

Effective birth control means using any of the following methods:

- Birth control drugs that prevent pregnancy—given by pills, patches, vaginal rings, injectables, or implant under the skin; or
- Intrauterine device (IUD).

You do not have to use birth control if:

- You have been diagnosed with early menopause, with no menstrual periods for one year;
- You have had a hysterectomy (your uterus removed);
- You have had your ovaries removed;
- You have a tubal ligation (your "tubes tied") or confirmed successful placement of a product that blocks the fallopian tubes.

Remember: If you are having sex, you need to use male or female condoms to protect yourself from HIV infection.

If you join the study, we will test you for pregnancy at some visits, including before each study IV.

# Appendix C Sample consent form for use of samples and information in other studies

Title: A phase 2b study to evaluate the safety and efficacy of VRC01 broadly neutralizing monoclonal antibody in reducing acquisition of HIV-1 infection in women in sub-Saharan Africa

HVTN protocol number: HVTN 703/HPTN 081, The AMP Study

Site: [Insert site name]

When samples are no longer needed for this study, the study sponsors want to keep them for use in other studies by HVTN, HPTN, or other researchers. We will call these "extra samples."

This form gives you information so you can decide if you want your extra samples and information used in other studies. You will mark your decision at the end of the form. If you have any questions, please ask.

#### 1. Do I have to agree?

No. You are free to say yes or no, or to change your mind after you sign this form. At your request, we will destroy all extra samples that we have. Your decision will not affect your being in this study or have any negative consequences here.

#### 2. Where are the samples stored?

Extra samples are stored in a secure central place called a repository. Your samples will be stored in the HVTN repository in South Africa.

#### 3. How long will the samples be stored?

There is no limit on how long your extra samples will be stored. [Site: insert limits if your regulatory authority imposes them.]

#### 4. Will I be paid for the use of my samples?

No. Also, a researcher may make a new scientific discovery or product based on the use of your samples. If this happens, there is no plan to share any money with you. The researcher is not likely to ever know who you are.

#### 5. Will I benefit from allowing my samples to be used in other studies?

Probably not. Results from these other studies are not given to you, this clinic, or your doctor. They are not needed for your medical care. They are not part of your medical record. The studies are only being done for research purposes.

#### 6. Will the HVTN or HPTN sell my samples and information?

No, but the HVTN and HPTN may share your samples with other researchers. Once we share your samples and information, we will not be able to get them back.

#### 7. How do other researchers get my samples and information?

When a researcher wants to use your samples and/or information, their research plan must be approved by the HVTN and HPTN. Also, the researcher's institutional review board (IRB) or ethics committee (EC) will review their plan. [Site: If review by your institution's IRB/EC/RE is also required, insert a sentence stating this.] IRBs/ECs protect the rights and well-being of people in research. If the research plan is approved, the HVTN and HPTN will send your samples to the researcher's location.

#### 8. What information is shared with other researchers?

The samples and limited information will be labeled with a code number. Your name will not be part of the information. However, some information that we share may be personal, such as your race, ethnicity, gender, health information from the study, and HIV status. We may share information about the study product you received and how your body responded to the study product.

#### 9. What kind of studies might be done with my extra samples and information?

The studies will be related to HIV prevention or infection, the immune system, and other diseases.

Researchers may also do genetic testing on your samples.

If you become HIV infected, the researchers may look at all of the genes of the virus found in your samples. The researchers will use this information to learn more about HIV and the study product(s).

In some cases, researchers may take cells from your samples and grow more of them over time, so that they can continue to contribute to this study.

If you agree, your samples could also be used for genome wide studies. In these studies, researchers will look at all of your genes (your genome). The researchers compare the genomes of many people, looking for common patterns of genes that could help them understand diseases. The researchers may put the information from the genome-wide studies into a protected database so that other researchers can access it. Usually, no one would be able to look at your genome and link it to you as a person. However, if another database exists that also has information on your genome and your name, someone might be able to compare the databases and identify you. If others found out, it could lead to discrimination or other problems. The risk of this is very small.

#### 10. What are the risks of genetic testing?

The genetic testing could show you may be at risk for certain diseases. If others found out, it could lead to discrimination or other problems. However, it is almost impossible for you or others to know your test results from the genetic testing. The results are not part of your study records and are not given to you.

#### 11. Who will have access to my information in studies using my extra samples?

People who may see your information are:

- Researchers who use your stored samples and limited information for other research
- Government agencies that fund or monitor the research using your samples or information
- Any regulatory agency that reviews clinical trials
- The researcher's Institutional Review Board or Ethics Committee
- The people who work with the researcher

All of these people will do their best to protect your information. The results of any new studies that use your extra samples or information may be published. No publication will use your name or identify you personally.

#### Questions

## 12. If you have questions or problems about allowing your samples and information to be used in other studies, use the following important contacts.

If you have questions about the use of your samples or information or if you want to change your mind about their use, contact [name and telephone number of the investigator or other study staff].

If you think you may have been harmed because of studies using your samples or information, contact [name and telephone number of the investigator or other study staff].

If you have questions about your rights as a research participant, contact [name/title/phone of person on IRB or other appropriate organization].

#### South African sites: Include the following:

If you have questions about this trial you should first discuss them with your doctor or the ethics committee (contact details as provided on this form). After you have consulted your doctor or the ethics committee and if they have not

provided you with answers to your satisfaction, you should write to the South African Medicines Control Council (MCC) at:

The Registrar of Medicines Medicines Control Council Department of Health Private Bag X828 PRETORIA 0001

Fax: (012) 395 9201

e-mail: mogobm@health.gov.za

13. Please choose only one of the options below and write your initials or make your mark in the box next to it. Whatever you choose, the HVTN and HPTN keep track of your decision about how your samples and information can be used.

| | studies related to HIV preven | nbined with limited information to be ution, the immune system, and other disceping my cells growing over time. | | ıay |
|---|---|---|---|---|
| OR | I agree to the option above an information to be used in gen | d also to allow my extra samples comome wide studies. | bined with lim | nited |
| OR | | | | |
| | | les to be used in any other studies. This wing more of my cells, or genome wide | | |
| ] | Participant's name (print) | Participant's signature or mark | Date | Time |
| Cli | nic staff conducting consent | Clinic staff signature | Date | Time |

For participants who are unable to read or write, a witness should complete the signature block below:

#### HVTN 703/HPTN 081 Version 4.0 / December 14, 2017

| Witness's name (print) | Witness's signature | Date | Time |
|---|---|---|---|
| *Witness is impartial and was | s present for the consent process. | | |

### **Appendix D** Tables of procedures (for sample informed consent form)

[Site: You may insert these tables of procedures into appropriate sections of your consent form(s) or give them to study volunteers/participants separately if you think they would be helpful. You are not required to do either.]

#### **HIV-uninfected participants**

| | | | | | | | | | 6 mc | onths | | | | | 1 | yea | r | | | | | 1½ y | ears | | 2 y | ears/ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | - | T | | · | | | т | | | | • | ····· | | | | I | , | | · | ······ | | | | | , | _ |
| Procedure | Screening<br>visit(s) | First IV<br>visit | 4 weeks | 8 weeks | 8 weeks +<br>5 days | 12 weeks | 16 weeks | 20 weeks | 24 weeks | 28 weeks | 32 weeks | 36 weeks | 40 weeks | 44 weeks | 48 weeks | 52 weeks | 56 weeks | 60 weeks | 64 weeks | 68 weeks | 72 weeks | 76 weeks | 80 weeks | 88 weeks | 96 weeks | 104 weeks |
| IV | • | ٧ | | ٧ | | | ٧ | | ٧ | | ٧ | | ٧ | | ٧ | | ٧ | | ٧ | | ٧ | | | | | |
| Medical history | ٧ | | • | | | | • | | | | | | | | | | • | - | | | • | | | | | |
| Complete physical exam | ٧ | | - | | | | | | | - | | | | | | | | - | | | | | - | | | ٧ |
| Brief physical exam | | ٧ | | ٧ | | | ٧ | | ٧ | | ٧ | | ٧ | | ٧ | | ٧ | | ٧ | | ٧ | | | | | |
| Urine test | ٧ | | | ٧ | | | | | | | | | | | - | | | | | | | | ٧ | | | |
| Blood drawn | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ |
| Pregnancy test* | ٧ | ٧ | - | ٧ | | | ٧ | | ٧ | | ٧ | | ٧ | | ٧ | | ٧ | | ٧ | | ٧ | | ٧ | | | |
| HIV test & pretest counseling | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ |
| Risk reduction counseling | ٧ | ٧ | | ٧ | | | ٧ | | ٧ | | ٧ | | ٧ | | ٧ | | ٧ | | ٧ | | ٧ | | | | | ٧ |
| Interview/Questionnaire | ٧ | ٧ | - | ٧ | | | ٧ | | ٧ | | ٧ | | ٧ | | ٧ | | ٧ | | ٧ | | ٧ | | | | | ٧ |
| STI testing (blood, urine, and/or swabs) † | | ٧ | | | | | | | ٧ | | | | | | ٧ | | | | | | ٧ | | | | | |

Not shown in this table is a time after all study participants have completed their last scheduled visit when you can find out whether you received the study antibody or the placebo.

<sup>\*</sup> Persons who have had their uterus or ovaries removed (a hysterectomy or oophorectomy), verified by medical records, are not required to have pregnancy tests.

<sup>†</sup> And if clinically indicated.

#### Participants discovered to have been HIV-1-infected at enrollment or who become HIV-2-infected

| | Weeks after 1 <sup>st</sup><br>positive HIV test | |
|---|---|---|
| Procedure | 4 | 24 |
| Medical history (as needed) | ٧ | ٧ |
| Brief physical (as needed) | ٧ | ٧ |
| Complete physical | | ٧ |
| Risk reduction counseling | ٧ | ٧ |
| Questions/questionnaire | ٧ | ٧ |
| Blood drawn | ٧ | ٧ |
| • | | ••••• |

Not shown in this table is a time after all study participants have completed their last scheduled visit when you can find out whether you received the study antibody or the placebo.

#### Participants who become HIV-1-infected

| | Weeks after 1 <sup>st</sup> positive<br>HIV test | | | | |
|---|---|---|---|---|---|
| Procedure | 4 | 6 | 8 | 12 | 24 |
| Medical history (as needed) | ٧ | ٧ | ٧ | ٧ | ٧ |
| Brief physical (as needed) | ٧ | ٧ | ٧ | ٧ | |
| Complete physical | | | | | ٧ |
| Risk reduction counseling | ٧ | ٧ | ٧ | ٧ | ٧ |
| Questions/questionnaire | ٧ | ٧ | ٧ | ٧ | ٧ |
| Blood drawn | ٧ | ٧ | ٧ | ٧ | ٧ |
| Pregnancy test* | | | | ٧ | |

Not shown in this table is a time after all study participants have completed their last scheduled visit when you can find out whether you received the study antibody or the placebo.

Participants who become HIV-1-infected may be invited to join a separate study for follow-up visits. That study will have a separate schedule of visits and procedures. It will also have a separate consent form, which will be reviewed with all participants who are invited to join that study.

<sup>\*</sup> Persons who have had their uterus or ovaries removed (a hysterectomy or oophorectomy), verified by medical records, are not required to have pregnancy tests.

#### Participants who discontinue infusions for reasons other than HIV infection

| | Weeks after enrollment | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Procedure | 8 | 20 | 32 | 44 | 56 | 72 | 88 | 104 |
| Brief physical (as needed) | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | |
| Complete physical | | | | | | | | ٧ |
| HIV testing & pretest counseling | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ |
| Risk reduction counseling | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ |
| Questions/questionnaire | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ |
| Urine test | ٧ | | | | | | ٧ | |
| Pregnancy test* | ٧ | | ٧ | | ٧ | | ٧ | |
| Blood drawn | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ | ٧ |

Study participants who discontinue infusions for reasons other than HIV infection will start this visit schedule at the first visit that occurs after their last infusion.

Not shown in this table is a time after all study participants have completed their last scheduled visit when you can find out whether you received the study antibody or the placebo.

<sup>\*</sup> Persons who have had their uterus or ovaries removed (a hysterectomy or oophorectomy), verified by medical records, are not required to have pregnancy tests.

# Appendix E Sample consent form for participants with HIV infection at enrollment or during the study

Title: A phase 2b study to evaluate the safety and efficacy of VRC01 broadly neutralizing monoclonal antibody in reducing acquisition of HIV-1 infection in women in sub-Saharan Africa

Protocol number: HVTN 703/HPTN 081, The AMP Study

Site: [Insert site name]

Please read this consent form or ask someone to read it to you. If you decide to, we will ask you to sign or make your mark on this form. We will offer you a copy to keep. We will ask you questions to see if we have explained everything clearly. You can also ask us questions about the study.

You are a participant in a study called HVTN 703/HPTN 081, The AMP Study. The rest of the information in the consent form that you signed earlier, about the study purpose, the risks and benefits of participation, your rights and responsibilities, and how your privacy is protected, continues to be important information for you and has not changed.

#### **About this form**

We tested your blood for HIV and you were found to be infected. We will help you get care and support.

You became infected either prior to enrollment or during your participation in the study. Because of this, you cannot stay in the study for its whole length. We would like you to come to the clinic for a different number of visits than what is explained in the main study consent form.

Depending on when you became infected, you will come to the clinic for 1-5 more visits, including today.

### 1. If you are found to have been HIV-1 infected when you enrolled, or if you have HIV-2 infection:

If you are found to have been HIV infected when you enrolled, you were already infected with HIV before you got the antibody or placebo. It takes a few days to complete the tests to see if you have HIV, so your infection was not found until after you got your first IV.

HIV-2 is a rare kind of HIV, most often found in West Africa.

We will counsel you about your HIV infection, talk with you about ways to avoid transmission and about telling your partner(s).

We are asking you to come to the clinic for 1-2 more visits (including today) within about 6 months of your diagnosis. At these visits, we will:

- Ask questions about your health;
- Do physical exams based on your complaints or symptoms;
- Ask questions about your risk of infecting others with HIV, including sexual behavior and drug use;
- Counsel you on ways to avoid transmitting HIV to other people;
- Collect blood samples (between 30 and 45 mL, or about 2 to 3 tablespoons, at each visit); and
- Ask questions about any personal problems or benefits you may have from participating in the study.

[Site: Insert the **second** table in Appendix D, Tables of procedures (for informed consent form) in this section or distribute it as a separate sheet if it is helpful to your study participants. You are not required to do either.]

#### 2. If you got infected with HIV-1 during the study:

If you became infected with HIV-1, we will counsel you about your HIV infection, talk with you about ways to avoid transmission and about telling your partner(s). You will not get any more IVs. We will ask you to come in for 4-5 more visits (including today) within about 6 months of your diagnosis. At these visits, we will:

- Ask questions about your health;
- Do physical exams based on your complaints or symptoms;
- Ask questions about your risk of infecting others with HIV, including sexual behavior and drug use;
- Counsel you on ways to avoid transmitting HIV to other people;
- Collect blood samples (between 70 mL and 130 mL, about ½ to ½ cup, at each visit); and
- Ask questions about any personal problems or benefits you may have from participating in the study.

[Site: Insert the **third** table in Appendix D, Tables of procedures (for informed consent form) in this section or distribute it as a separate sheet if it is helpful to your study participants. You are not required to do either.]

#### Leaving the study

**3.** Tell us if you decide to leave the study.

You are free to leave the study at any time and for any reason. Your care at this clinic and your legal rights will not be affected, but it is important for you to let us know.

We will ask you to come back to the clinic one last time for a physical exam, and we may ask to take some blood and urine samples. We will also ask about any personal problems or benefits you have experienced from being in the study. We believe these steps are important to protecting your health, but it is up to you whether to complete them.

#### Questions

If you have questions or problems at any time during your participation in this study, use the following important contacts.

If you have questions about this study, contact [name and telephone number of the investigator or other study staff].

If you have any symptoms that you think may be related to this study, contact [name and telephone number of the investigator or other study staff].

If you have questions about your rights as a research participant, or problems or concerns about how you are being treated in this study, contact [name/title/phone of person on IRB or other appropriate organization].

If you want to leave this study, contact [name and telephone number of the investigator or other study staff].

#### South African sites: Include the following:

If you have questions about this trial you should first discuss them with your doctor or the ethics committee (contact details as provided on this form). After you have consulted your doctor or the ethics committee and if they have not provided you with answers to your satisfaction, you should write to the South African Medicines Control Council (MCC) at:

The Registrar of Medicines Medicines Control Council Department of Health Private Bag X828 PRETORIA 0001

Fax: (012) 395 9201

e-mail: mogobm@health.gov.za

### Your permissions and signature

If you agree to continue in this study with this new visit schedule, you will need to sign or make your mark below. Before you sign or make your mark on this consent form, make sure of the following:

- You have read this consent form, or someone has read it to you.
- You feel that you understand the changes to the visit schedule and what will happen to you. You understand that the possible risks and benefits of participation have not changed.
- You have had your questions answered and know that you can ask more at any time.
- You agree to continue in this study.

You will not be giving up any of your rights by signing this consent form.

| Participant's name (print) | Participant's signature or mark | Date | Time |
|---|---|---|---|
| Study staff conducting consent discussion (print) | Study staff signature | Date | Time |
| For participants who as | re unable to read or write, also o | complete the signat | ure block |
| below: | | | |
| Witness's name (print)# | Witness's signature | Date | Time |

<sup>#</sup> Witness is impartial and was present for the consent process.
### Appendix F Schedule 1—Laboratory procedures for HIV-uninfected participants

| | | | | Visit: | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 | 23 | 24 | 25 | 26 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Day: | Screening | D0 | D28 | D56 | D61 | D84 | D112 | D140 | D168 | D196 | D224 | D252 | D280 | D308 | D336 | D364 | D392 | D420 | D448 | D476 | D504 | D532 | D560 | D616 | D672 | D728 | 1 |
| | | | | Week: | visit <sup>3</sup> | W0 | W4 | W8 | | W12 | W16 | W20 | W24 | W28 | W32 | W36 | W40 | W44 | W48 | W52 | W56 | W60 | W64 | W68 | W72 | W76 | W80 | W88 | W96 | W104 | 1 |
| | | | | | | Inf#1 | | Inf#2 | | | Inf#3 | | Inf#4 | | Inf#5 | | Inf#6 | | Inf#7 | | Inf#8 | | Inf#9 | | Inf#10 | | | | | | |
| | | | | Tube size | | 1111#1 | | IIII#2 | | | 1111#3 | | 1111#4 | | 1111#5 | | 1111#6 | | 1111#7 | | 1111#0 | | 1111#9 | | 1111#10 | | | | | | |
| | | | Tube | (vol. | | | | | | | | | | | | | | | | | | | | | | | | | | | Total |
| Procedure | Ship to <sup>1</sup> | Assay location <sup>1,2</sup> | Type⁴ | capacity)4 | | | | | | | | | | | | _ | | | | | | | | _ | | | | | | | |
| BLOOD COLLECTION | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Screening/Diagnostic | Local lab | Local lab | SST | 5mL | 5 | | | | | - | | | | | | ļ | - | - | | | | | | | | | | | | + | 5 |
| Screening HIV test HIV diagnostics <sup>7</sup> | HSML-NICD /<br>UW-VSL | HSML-NICD /<br>UW-VSL | EDTA | 10mL | _ | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 20 <sup>7</sup> | 260 |
| Safety labs | OW-VOL | OVV-VOL | | | L | - | - | - | - | - | L | | | | ł | | - | - | | | | | | | | | - | | | + | |
| CBC/ Differential | Local lab | Local lab | EDTA | 5mL | 5 | 5 | _ | 5 | _ | _ | 5 | _ | 5 | _ | 5 | - | 5 | _ | 5 | _ | 5 | _ | 5 | _ | 5 | _ | _ | _ | _ | _ | 55 |
| ALT, Creatinine | Local lab | Local lab | SST | 5mL | 5 | 5 | | 5 | <del> -</del> | += | 5 | = | 5 | | 5 | <del> =</del> | 5 | 1 = | 5 | | 5 | | 5 | <del> =</del> - | 5 | | | = | += | += | 55 |
| STI Serology | LOCALIAD | Local lab | 1 001 | JIIL | , , | | - | | _ | | | | 3 | | - 3 | - | | | , , | | J | | J | | | | - | | <del></del> | + | |
| Syphilis <sup>11</sup> | Local lab | Local lab | SST | 5mL | I – | 5 <sup>13</sup> | _ | - | | _ | | | 5 <sup>13</sup> | | | | <b>—</b> | - | 5 <sup>13</sup> | | | - | | | 5 <sup>13</sup> | | - | | | | 20 |
| Drug Levels/Detection | Local lab | Local lab | 1 001 | JIIL | l | 5 | ļ | | | <u> </u> | | | 3 | | | <del> </del> | | ļ <u></u> | 5 | | | | | ļ | 5 | | | | ļ | + | |
| VRC01 Ab levels | CSR | NVITAL | SST | 8.5mL | _ | v | V | V | v | v | v | v | v | v | v | v | v | v | v | v | v | v | v | v | v | V | v | v | v | v | 0 |
| ARV detection by serum or plasma <sup>10</sup> | CSR | JHU | SST | 8.5mL | | V | _ | v | - | ,<br>_ | v | , | V | | v | ,<br> _ | y<br>V | , , | V | _ | V | _ | V | <u>, , </u> | V | | V | ,<br>_ | v | , , | 0 |
| ARV detection by dried blood spots 16 | CSR | HVTN Labs | EDTA | 2mL | | <del>,</del> | 1 | <u></u> | l | i | L | L | L | L | · | L | )<br>Se | ee footnote | <u> </u> | l | | | | L | | L | <u> </u> | L | <u> </u> | اــــــا | 0 |
| Immunogenicity & Virologic Assays | | 111111111111111111111111111111111111111 | 1 2011 | | l | J | | | | | | | | | | | | | | | | | | | | | | | | | |
| Host genetics <sup>5</sup> | CSR | HVTN Labs | ACD | 8.5mL | _ | z | _ | _ | _ | _ | _ | _ | _ | | _ | <u> </u> | _ | _ | _ | _ | _ | - | _ | _ | _ | _ | _ | _ | - | _ | 0 |
| Anti-VRC01 Ab levels | CSR | VRC/NVITAL | SST | 8.5mL | _ | V | - | - | <del> </del> | <u> </u> | _ | _ | _ | | _ | V | <u> </u> | - | | | | <u> </u> | _ | - | _ | V | <u> </u> | _ | + | T - | 0 |
| Functional humoral assays <sup>8</sup> | CSR | HVTN Labs /<br>VRC / NVITAL | SST | 8.5mL | _ | у | у | у | у | у | у | у | у | у | у | у | у | у | у | у | у | у | у | у | у | у | у | у | у | у | 0 |
| Viral isolation/sequencing <sup>9</sup> | CSR | HVTN Labs | EDTA | 10mL | _ | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 250 |
| STORAGE | | | | | | - | 1 | - | - | - | | | | | - | - | - | | | | | | | | - | | 1 | | - | - | |
| Serum storage | CSR | _ | SST | 8.5mL | _ | 76.5 | 51 | 51 | 42.5 | 51 | 42.5 | 42.5 | 42.5 | 42.5 | 42.5 | 51 | 42.5 | 42.5 | 42.5 | 42.5 | 42.5 | 42.5 | 42.5 | 42.5 | 42.5 | 51 | 42.5 | 42.5 | 42.5 | 42.5 | 1139 |
| PBMC storage | CSR | _ | ACD | 8.5mL | _ | 51 | <u> </u> | - | - | T - | | _ | _ | | - | <u> </u> | 34 | <u> </u> | _ | _ | _ | _ | _ | - | 34 | _ | - | _ | _ | 34 | 153 |
| Visit total <sup>17</sup> | | | | | 15 | 165 | 73 | 83 | 65 | 73 | 75 | 65 | 80 | 65 | 75 | 73 | 109 | 65 | 80 | 65 | 75 | 65 | 75 | 65 | 114 | 73 | 65 | 65 | 65 | 109 | 1987 |
| 56-Day total 17 | | | | | 15 | 180 | 253 | 336 | 221 | 294 | 295 | 212 | 219 | 209 | 219 | 212 | 256 | 246 | 253 | 209 | 219 | 204 | 214 | 204 | 253 | 251 | 251 | 129 | 129 | 173 | 1 |
| URINE COLLECTION | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Urine dipstick <sup>15</sup> | Local lab | Local lab | | | Х | _ | _ | X | _ | T - | | _ | _ | _ | T | T | T - | T - | | | | _ | | Ι – | I – | _ | Х | | _ | _ | |
| Pregnancy Test <sup>6</sup> | Local lab | Local lab | | | X | Х | <u> </u> | X | <u> </u> | T — | X | _ | Х | _ | X | 1 | X | <u> </u> | X | | × | _ | X | <u> </u> | X | _ | Х | _ | T- | _ | 1 |
| CERVICAL/VAGINAL SWAB COLLECTION | ON . | | | | · | | | | | | | | | | | | 1 | | | | | | | | | | 1 | | | | |
| Trichomonas vaginalis | Local lab | Local lab | T | | _ | X <sup>14</sup> | _ | Ι – | <u> </u> | | _ | _ | X <sup>14</sup> | _ | T — | T - | 1 - | _ | X <sup>14</sup> | _ | _ | _ | _ | T - | X <sup>14</sup> | _ | <u> </u> | _ | T - | _ | i |
| EITHER URINE OR CERVICAL/VAGINAL | SWAB COLLECTIO | N | | | | | <b></b> | | <del>}</del> | | ····· | | | | | | | - | | <b>^</b> | · | | | | 4 | | <u> </u> | | | 1 | |
| Urine - Chlamydia/Gonorrhea <sup>12</sup> | Local lab | Local lab | | | _ | X <sup>13</sup> | _ | _ | - | _ | _ | _ | X <sup>13</sup> | _ | _ | _ | - | _ | X <sup>13</sup> | _ | _ | _ | _ | <u> </u> | X <sup>13</sup> | _ | _ | _ | <u> </u> | T – | |
| Cervical/Vaginal Swab -<br>Chlamydia/Gonorrhea <sup>12</sup> | Local lab | Local lab | | | _ | X <sup>13</sup> | - | - | - | - | - | - | X <sup>13</sup> | - | - | - | - | - | X <sup>13</sup> | - | - | - | - | - | X <sup>13</sup> | - | - | - | - | - | |

<sup>&</sup>lt;sup>1</sup> CSR = central specimen repository; HSML-NICD = HIV Sero-Molecular Laboratory, National Institute for Communicable Diseases (Johannesburg, South Africa); UW-VSL = University of Washington Virology Specialty Laboratory (Seattle, Washington, USA)

<sup>&</sup>lt;sup>2</sup> HVTN Laboratories include: Cape Town HVTN Immunology Laboratory (CHIL, Cape Town, South Africa); South Africa Immunology Laboratory-National Institute for Communicable Diseases (SAIL-NICD, Johannesburg, South Africa); Fred Hutchinson Cancer Research Center (Seattle, Washington, USA); Duke University Medical Center (Durham, North Carolina, USA); University of Cape Town (Cape Town, South Africa); University of Colorado Denver (Aurora, Colorado, USA).

Non-HVTN laboratories: NVITAL = NIAID Vaccine Immune T-Cell Antibody Laboratory (Gaithersburg, Maryland, USA); VRC = Vaccine Research Center (Bethesda, Maryland, USA); JHU = Johns Hopkins University, HPTN Laboratory Center (Baltimore, Maryland, USA).

<sup>&</sup>lt;sup>3</sup> Screening may occur over the course of several contacts/visits up to and including day 0 prior to infusion.

<sup>&</sup>lt;sup>4</sup>Local labs may assign appropriate alternative tube types for locally performed tests.

<sup>&</sup>lt;sup>5</sup> Genotyping may be performed on enrolled participants using cryopreserved PBMC collected at baseline.

- <sup>6</sup> Pregnancy test must be performed on urine or blood specimens on the day of infusion with negative results received prior to infusion.
- At an early termination visit for a withdrawn or terminated participant (see Section 7.12), blood should be drawn for HIV diagnostic testing, as shown for visit 26 above.
- <sup>8</sup> Functional humoral assays include nAb, ADCC, virion capture, and phagocytosis assays.
- <sup>9</sup> EDTA blood collected for plasma may also be used for ARV detection assay, if necessary.
- <sup>10</sup> Testing plan for ARV detection to be determined.
- <sup>11</sup> Syphilis testing will be done by serology.
- 12 Chlamydia/Gonorrhea testing will be done with EITHER urine OR cervical/vaginal swab. Either specimen is acceptable, and clinics will determine which specimen will be collected and tested.
- 13 Syphilis testing, and chlamydia/gonorrhea testing by either urine or cervical/vaginal swab, will be performed at visits 2, 9, 15, and 21; in addition, testing may occur at any visit if clinically indicated.
- <sup>14</sup> Cervical/vaginal swab will be collected for Trichomonas testing at visits 2, 9, 15, and 21; in addition, testing may occur at any visit if clinically indicated.
- <sup>15</sup> And microscopy if needed.
- <sup>16</sup> EDTA blood for dried blood spots will be collected on regularly scheduled calendar days throughout the study. Refer to the Specimen Collection SSP for more information.
- <sup>17</sup> The total 56-day blood collection includes 2mL EDTA blood collection for dried blood spots. It is highly improbable that the 2mL EDTA blood collection will occur at every possible timepoint, but it is reflected in the blood draw totals for every visit to account for this extreme possibility.
- y = SST blood collected for serum storage will also cover specimen needs for the VRC01 drug level, ARV detection, and functional humoral assays; no separate blood draw is needed.
- z = ACD blood collected for PBMC storage will also cover specimen needs for host genetics assay; no separate blood draw is needed.

## **Appendix G** Schedule 2—Laboratory procedures for HIV-1–infected participants

| | | | | Visit: | #.X <sup>5</sup> | Visit: | 31 | 32 | 33 | 34 | 35 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | Days: | D28 | D42 | D56 | D84 | D168 | |
| | | | | | | Weeks after<br>diagnosis <sup>7</sup> : | W4 | W6 | W8 | W12 | W24 | |
| Procedure | Ship to <sup>1</sup> | Assay location <sup>1,2</sup> | Tube<br>Type <sup>3</sup> | Tube size<br>(vol. capacity) <sup>3</sup> | | | | | | | | Total |
| BLOOD COLLECTION | | | | | | | | | | | | |
| Screening or diagnostic assays | | | | | | | | | | | | |
| HIV diagnostics | HSML-NICD /<br>UW-VSL | HSML-NICD /<br>UW-VSL | EDTA | 10mL | 20 | | _ | _ | _ | _ | _ | 20 |
| HIV PCR viral load | HSML-NICD | HSML-NICD | EDTA | 10mL | _ | *************************************** | 10 | 10 | 10 | 10 | 10 | 50 |
| CD4+T cell count | Local Lab | Local Lab | EDTA | 5mL | 5 | | 5 | 5 | 5 | 5 | 5 | 30 |
| Safety lab | | | | | *************************************** | | | | | | | |
| Hemoglobin | Local Lab | Local Lab | EDTA | 5mL | _ | | _ | _ | 5 | 5 | | 10 |
| Drug levels | | | | | × | , | | - | V | | | |
| VRC01 Ab levels | CSR | NVITAL | SST | 8.5mL | 8.5 | D | 8.5 | 8.5 | 8.5 | 8.5 | 8.5 | 51 |
| Immunogenicity & Virologic Assays | | | | | | | | | å | *************************************** | · | |
| Functional humoral assays <sup>6</sup> | CSR | HVTN Labs /<br>VRC / NVITAL | SST | 8.5mL | 17 | | 17 | 17 | 17 | 17 | 17 | 102 |
| Viral isolation/sequencing | CSR | HVTN Labs | EDTA | 10mL | 10 | | 10 | 10 | 10 | 10 | 10 | 60 |
| Storage | | | | | | | | | | | | |
| Serum | CSR | | SST | 8.5mL | 25.5 | | 17 | 17 | 17 | 17 | 17 | 110.5 |
| Plasma | CSR | | EDTA | 5mL | 5 | | 5 | 5 | 5 | 5 | 5 | 30 |
| PBMC | CSR | | ACD | 8.5mL | 34 | | _ | _ | _ | 34 | 34 | 102 |
| Visit total | | , | | | 125 | | 72.5 | 72.5 | 77.5 | 111.5 | 106.5 | 566 |
| 56-Day total | | | | | 125 | | 198 | 270 | 348 | 334 | 106.5 | |
| URINE COLLECTION | | | | | | , | | | | | | |
| Pregnancy Test <sup>4</sup> | Local Lab | Local Lab | | | Х | | _ | _ | _ | Х | _ | |

<sup>&</sup>lt;sup>1</sup> CSR = central specimen repository; HSML-NICD = HIV Sero-Molecular Laboratory-National Institute for Communicable Diseases (Johannesburg, South Africa); UW-VSL = University of Washington Virology Specialty Laboratory (Seattle, Washington, USA)

<sup>&</sup>lt;sup>2</sup> HVTN Laboratories include: South African Immunology Laboratory-National Institute for Communicable Diseases (SAIL-NICD, Johannesburg, South Africa); Duke University Medical Center (Durham, North Carolina, USA); University of Cape Town (Cape Town, South Africa)

Non-HVTN laboratories: NVITAL = NIAID Vaccine Immune T-Cell Antibody Laboratory (Gaithersburg, Maryland, USA); VRC = Vaccine Research Center (Bethesda, Maryland, USA)

<sup>&</sup>lt;sup>3</sup> Local labs may assign appropriate alternative tube types for locally performed tests.

<sup>&</sup>lt;sup>4</sup> Pregnancy test may be performed on blood specimens.

<sup>&</sup>lt;sup>5</sup> Visit #.X indicates a Redraw visit where # is a Schedule 1 visit number. Confirmatory draw for HIV diagnostics will be collected at the Redraw visit, in addition to the other indicated specimens. The Redraw visit should occur as soon as possible after the clinic receives a Redraw Request from the HIV diagnostics laboratory. Multiple subsequent Redraw visits may be necessary; only the EDTA blood specimens for HIV diagnostics, viral isolation/sequencing, and plasma storage will be collected at the subsequent Redraw visits. Refer to the HIV Testing SSP for more information.

<sup>&</sup>lt;sup>6</sup> Functional humoral assays include nAb, ADCC, virion capture, and phagocytosis assays.

<sup>&</sup>lt;sup>7</sup> Date of diagnosis = date of the initial specimen draw that led to the first Redraw Request.

# Appendix H Schedule 3—Laboratory procedures for participants discovered to have been HIV-1-infected at enrollment or who become HIV-2-infected

| | | | | | 5 | | | l | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | Visit: | #.X <sup>5</sup> | Visit: | 47 | 48 | |
| | | | | | | Days: | D28 | D168 | |
| | | | | | | Weeks after diagnosis 7: | W4 | W24 | |
| | | | Tube | Tube size | | | | | |
| Procedure | Ship to <sup>1</sup> | Assay location <sup>1,2</sup> | Type <sup>3</sup> | (vol. capacity) <sup>3</sup> | | | | | Total |
| BLOOD COLLECTION | | | | | | | | | |
| Screening or diagnostic assays | | | | | | | | | |
| HIV diagnostics | HSML-NICD /<br>UW-VSL | HSML-NICD /<br>UW-VSL | EDTA | 10mL | 20 | | | _ | 20 |
| HIV PCR viral load | HSML-NICD | HSML-NICD | EDTA | 10mL | _ | | 10 | 10 | 20 |
| CD4+T cell count | Local Lab | Local Lab | EDTA | 5mL | 5 | | 5 | 5 | 15 |
| Drug levels | | | | | | | | | |
| VRC01 Ab levels | CSR | NVITAL | SST | 8.5mL | 8.5 | | _ | _ | 8.5 |
| Immunogenicity & Virologic Assays | | | | | | | | | |
| Functional humoral assays <sup>6</sup> | CSR | HVTN Labs /<br>VRC / NVITAL | SST | 8.5mL | 17 | | | _ | 17 |
| Viral isolation/sequencing | CSR | HVTN Labs | EDTA | 10mL | 10 | | _ | _ | 10 |
| Storage | | | | | | | | | |
| Serum | CSR | | SST | 8.5mL | 25.5 | | 17 | 17 | 59.5 |
| Plasma | CSR | | EDTA | 5mL | 5 | | _ | | 5 |
| PBMC | CSR | | ACD | 8.5mL | 34 | | _ | _ | 34 |
| Visit total | | | | | 125 | | 32 | 32 | 189 |
| 56-Day total | | | | | 125 | | 157 | 32 | |
| URINE COLLECTION | | | | | | , | | | |
| Pregnancy Test <sup>4</sup> | Local Lab | Local Lab | - | | Х | | _ | _ | |

<sup>&</sup>lt;sup>1</sup> CSR = central specimen repository; HSML-NICD = HIV Sero-Molecular Laboratory-National Institute for Communicable Diseases (Johannesburg, South Africa); UW-VSL = University of Washington Virology Specialty Laboratory (Seattle, Washington, USA).

<sup>&</sup>lt;sup>2</sup> HVTN Laboratories include: South African Immunology Laboratory–National Institute for Communicable Diseases (SAIL-NICD, Johannesburg, South Africa); Duke University Medical Center (Durham, North Carolina, USA); University of Cape Town (Cape Town, South Africa).

Non-HVTN laboratories: NVITAL = NIAID Vaccine Immune T-Cell Antibody Laboratory (Gaithersburg, Maryland, USA); VRC = Vaccine Research Center (Bethesda, Maryland, USA).

<sup>&</sup>lt;sup>3</sup> Local labs may assign appropriate alternative tube types for locally performed tests.

<sup>&</sup>lt;sup>4</sup> Pregnancy test may be performed on blood specimens.

<sup>&</sup>lt;sup>5</sup> Visit #.X indicates a Redraw visit where # is a Schedule 1 visit number. Confirmatory draw for HIV diagnostics will be collected at the Redraw visit, in addition to the other indicated specimens. The Redraw visit should occur as soon as possible after the clinic receives a Redraw Request from the HIV diagnostics laboratory. Multiple subsequent Redraw visits may be necessary; only the EDTA blood specimens for HIV diagnostics, viral isolation/sequencing, and plasma storage will be collected at the subsequent Redraw visits. Refer to the HIV Testing SSP for more information.

<sup>&</sup>lt;sup>6</sup> Functional humoral assays include nAb, ADCC, virion capture, and phagocytosis assays.

<sup>&</sup>lt;sup>7</sup> Date of diagnosis = date of the initial specimen draw that led to the first Redraw Request.

## Appendix I Schedule 4—Laboratory procedures for participants who discontinue infusions for reasons other than HIV infection

| | | | | Visit: | 71 | 72 | 73 | 74 | 75 | 76 | 77 | 78 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Days after enrollment: | D56 | D140 | D224 | D308 | D392 | D504 | D616 | D728 | |
| | | | | Weeks after enrollment: | W8 | W20 | W32 | W44 | W56 | W72 | W88 | W104 | |
| Procedure | Ship to <sup>1</sup> | Assay location <sup>1,2</sup> | Tube Type <sup>3</sup> | Tube size<br>(vol. capacity)³ | | | | | | | | | Total |
| BLOOD COLLECTION | | | ~~~~ | | | | | | | | | | |
| Screening or diagnostic assays | | | | | | | | | | | | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | |
| HIV diagnostics <sup>5</sup> | HSML-NICD /<br>UW-VSL | HSML-NICD /<br>UW-VSL | EDTA | 10mL | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 20 <sup>5</sup> | 90 |
| Safety labs | | | | | | | | | | | | | |
| CBC/ Differential | Local lab | Local lab | EDTA | 5mL | 5 | <del>-</del> | 5 | _ | 5 | _ | _ | <u> </u> | 15 |
| ALT, Creatinine | Local lab | Local lab | SST | 5mL | 5 | <u> </u> | 5 | <u> </u> | 5 | _ | _ | <u> </u> | 15 |
| Drug Levels | | | | | | | | | | | | | |
| VRC01 Ab levels | CSR | NVITAL | SST | 8.5mL | у | у | у | у | у | у | у | у | 0 |
| Immunogenicity & Virologic Assay | ys | | | | | | | | | | | | |
| Functional humoral assays <sup>6</sup> | CSR | HVTN Labs /<br>VRC / NVITAL | SST | 8.5mL | у | у | у | у | у | у | у | у | 0 |
| Viral isolation/sequencing | CSR | HVTN Labs | EDTA | 10mL | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 80 |
| STORAGE | | | | | | | | | | | | | |
| Serum storage | CSR | _ | SST | 8.5mL | 51 | 42.5 | 42.5 | 42.5 | 42.5 | 42.5 | 42.5 | 42.5 | 349 |
| PBMC storage | CSR | _ | ACD | 8.5mL | _ | _ | <u> </u> | _ | _ | _ | _ | 34 | 34 |
| Visit total | | | | | 81 | 63 | 73 | 63 | 73 | 63 | 63 | 107 | 583 |
| 56-Day total | | | | | 81 | 63 | 73 | 63 | 73 | 63 | 63 | 107 | |
| URINE COLLECTION | | | | | | | | | | | | | |
| Urine dipstick <sup>7</sup> | Local lab | Local lab | | | X | <u> </u> | <u> </u> | _ | | _ | Х | _ | |
| Pregnancy Test <sup>4</sup> | Local lab | Local lab | | | Х | <u> </u> | Х | _ | Х | _ | Х | <u> </u> | |

<sup>&</sup>lt;sup>1</sup> CSR = central specimen repository; HSML-NICD = HIV Sero-Molecular Laboratory-National Institute for Communicable Diseases (Johannesburg, South Africa); UW-VSL = University of Washington Virology Specialty Laboratory (Seattle, Washington, USA)

Non-HVTN laboratory: NVITAL = NIAID Vaccine Immune T-Cell Antibody Laboratory (Gaithersburg, Maryland, USA); VRC = Vaccine Research Center (Bethesda, Maryland, USA).

<sup>&</sup>lt;sup>2</sup> HVTN Laboratories include: South African Immunology, Laboratory-National Institute for Communicable Diseases (SAIL-NICD Johannesburg, South Africa); Duke = Duke University Medical Center (Durham, North Carolina, USA); University of Cape Town, South Africa)

<sup>&</sup>lt;sup>3</sup> Local labs may assign appropriate alternative tube types for locally performed tests.

<sup>&</sup>lt;sup>4</sup> Pregnancy test may be performed on blood specimens.

<sup>&</sup>lt;sup>5</sup> At an early termination visit for a withdrawn or terminated participant (see Section 7.12), blood should be drawn for HIV diagnostic testing, as shown for visit 78 above.

<sup>&</sup>lt;sup>6</sup> Functional humoral assays include nAb, ADCC, virion capture, and phagocytosis assays.

<sup>&</sup>lt;sup>7</sup> And microscopy if needed.

y = SST blood collected for serum storage will also cover specimen needs for the VRC01 drug level and functional humoral assays; no separate blood draw is needed.

## Appendix J Schedule 1—Procedures at CRS for HIV-uninfected participants

| Visit: | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 | 23 | 24 | 25 | 26 | Post |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day: | Screening | D0 | D28 | D56 | D61 | D84 | D112 | D140 | D168 | D196 | D224 | D252 | D280 | D308 | D336 | D364 | D392 | D420 | D448 | D476 | D504 | D532 | D560 | D616 | D672 | D728 | |
| Week: | visit <sup>1</sup> | W0 | W4 | W8 | | W12 | W16 | W20 | W24 | W28 | W32 | W36 | W40 | W44 | W48 | W52 | W56 | W60 | W64 | W68 | W72 | W76 | W80 | W88 | W96 | W104 | |
| Procedure | Scr. | Inf#1 | | Inf#2 | | | Inf#3 | | Inf#4 | | Inf#5 | | Inf#6 | | Inf#7 | | Inf#8 | | Inf#9 | | Inf#10 | | | | | | |
| tudy procedures <sup>2</sup> | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Signed screening consent (if used) | Х | - | _ | _ | - | - | _ | _ | _ | _ | _ | - | _ | _ | - | _ | _ | - | _ | _ | _ | - | _ | _ | _ | _ | - |
| Assessment of understanding | Х | - | _ | _ | - | _ | _ | _ | - | _ | - | - | _ | _ | - | _ | - | - | _ | _ | _ | - | _ | _ | _ | _ | - |
| Signed protocol consent | Х | - | _ | _ | - | _ | _ | _ | _ | _ | _ | - | _ | _ | _ | _ | _ | - | _ | _ | _ | _ | _ | _ | _ | _ | - |
| Medical history | Х | - | _ | - | - | - | _ | _ | - | _ | - | - 1 | _ | _ | - | _ | - | - | _ | _ | _ | - | - | _ | - | - | - |
| Complete physical exam | Х | - | _ | - | - | - | _ | — | - | _ | - | - 1 | _ | _ | - | _ | - | - | _ | _ | _ | - | l – | _ | - | Х | T - |
| Abbreviated physical exam | _ | Х | _ | Х | <u> </u> | - | Х | <u> </u> | Х | _ | Х | - | Х | _ | Х | _ | Х | - | Х | _ | Х | - | _ | - | _ | _ | - |
| Risk reduction counseling | Х | Х | _ | Х | - | | Х | _ | Х | _ | Х | - | Х | _ | Х | _ | Х | - 1 | Х | _ | Х | _ | <u> </u> | - | - | Х | T - |
| Pregnancy prevention assessment <sup>3</sup> | X | Х | _ | Х | _ | - | Х | _ | Х | _ | Х | - | Х | _ | Х | _ | Х | - | Х | _ | Х | - | _ | - | _ | Х | - |
| Confirm eligibility, obtain demographics, randomize | X | | _ | - | _ | <b>—</b> | _ | _ | | _ | _ | - | _ | _ | - | _ | - | - 1 | _ | _ | - | | _ | _ | - | _ | T - |
| Social impact assessment | _ | Х | _ | Х | | <b>—</b> | Х | <u> </u> | Х | _ | Х | - | Х | _ | Х | _ | Х | - | Х | _ | Х | - | _ | _ | <b>—</b> | Х | |
| Participant Questionnaire | _ | Х | _ | Х | | - | Х | _ | Х | - | Х | - | Х | _ | Х | _ | Х | - | Х | - | Χ | | _ | - | _ | Х | <u> </u> |
| Concomitant medications | X | Х | _ | Х | T — | _ | Х | _ | Х | - | Х | - | Х | _ | Х | _ | Х | - | Х | - | Х | _ | _ | - | - | Х | <b>-</b> |
| Intercurrent illness/adverse experience | _ | Х | _ | Х | _ | _ | Х | <u> </u> | Х | _ | Х | - | Х | _ | Х | _ | Х | - | Х | _ | Х | - | _ | _ | _ | Х | _ |
| HIV infection assessment <sup>4</sup> | X | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | - |
| Confirm HIV test results provided to participant 13 | _ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| ocal lab assessment | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Screening HIV test | Х | - | _ | _ | - | _ | _ | _ | _ | _ | _ | - | _ | _ | - | _ | - | - | _ | _ | _ | - | _ | _ | _ | _ | - |
| Urine dipstick <sup>12</sup> | Х | | _ | Х | — | - | _ | _ | — | _ | _ | - 1 | _ | _ | - | _ | _ | - | _ | _ | _ | - | Х | _ | - | _ | - |
| Pregnancy (urine or serum HCG) <sup>5</sup> | X | Х | _ | Х | - | - | Х | _ | Х | _ | Х | - | Х | _ | Х | _ | Х | - | Х | _ | Х | - | Х | _ | - | _ | _ |
| CBC, differential | Х | Х | _ | Х | - | - | Х | _ | Х | _ | Х | - | Х | _ | Х | _ | Х | - | Х | _ | Х | - | _ | _ | - | _ | - |
| ALT, Creatinine | X | Х | _ | Х | - | - | Х | <u> </u> | Х | _ | Х | - | Х | _ | Х | _ | Х | - | Х | _ | Х | - | _ | _ | _ | - | – |
| Syphilis <sup>6</sup> | _ | X <sup>7</sup> | _ | _ | | — | _ | | X <sup>7</sup> | _ | _ | - | _ | _ | X <sup>7</sup> | _ | - | - 1 | _ | _ | X <sup>7</sup> | | | | _ | _ | - |
| Chlamydia, Gonorrhea <sup>8</sup> | _ | X <sup>7</sup> | _ | _ | _ | _ | _ | <u> </u> | X <sup>7</sup> | _ | _ | - | _ | _ | X <sup>7</sup> | _ | - | - | _ | _ | X <sup>7</sup> | _ | _ | _ | _ | _ | <b>-</b> |
| Trichomonas vaginalis (cervical/vaginal swab) | _ | X <sup>9</sup> | _ | - | | - | _ | _ | X <sup>9</sup> | _ | _ | - | _ | _ | X <sup>9</sup> | _ | _ | - 1 | _ | _ | X <sup>9</sup> | - | _ | - | _ | _ | T - |
| tudy product administration procedures | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| IV infusion <sup>10</sup> | _ | Х | _ | Х | _ | <u> </u> | Χ | | Х | _ | Х | - | Х | _ | Х | _ | Х | - | Х | _ | Х | | _ | _ | _ | _ | _ |
| Reactogenicity assessment <sup>11</sup> | _ | Х | _ | Х | _ | T - | Х | _ | Х | _ | Х | _ | Х | _ | Х | _ | Х | _ | Х | _ | Х | <u> </u> | _ | _ | <u> </u> | _ | <u> </u> |
| | | | | 1 | | | | | | | | | | | | | | | | | | | | | | | |
| Poststudy | | | | | | | | | | | | 90 | | | | | | | | | | | | | | | |

Screening may occur over the course of several contacts/visits up to and including day 0 prior to infusion.

<sup>&</sup>lt;sup>2</sup> For specimen collection requirements, see Appendix F.

<sup>&</sup>lt;sup>3</sup> Pregnancy prevention assessments are required only for participants who are capable of becoming pregnant.

<sup>&</sup>lt;sup>4</sup> Includes pre-test counseling and HIV testing. A subsequent follow-up contact is conducted to provide post-test counseling and to report results to participant.

- <sup>5</sup> Pregnancy test must be performed on the day of infusion with negative results received prior to infusion. Pregnancy test to determine eligibility may be performed at screening, but must also be done on Day 0 prior to infusion. Persons who are NOT capable of becoming pregnant due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing. Serum pregnancy tests may be used to confirm the results of, or substitute for, a urine pregnancy test.
- <sup>6</sup> Syphilis testing will be done by serology.
- <sup>7</sup> Syphilis and Chlamydia/Gonorrhea testing may be performed at additional timepoints if clinically indicated.
- <sup>8</sup> Chlamydia/Gonorrhea testing will be done by urine or cervical/vaginal swab.
- <sup>9</sup> Cervical/vaginal swab may be collected for Trichomonas testing at additional timepoints if clinically indicated.
- <sup>10</sup> Blood draws required at infusion visits must be performed prior to administration of study product; however, it is not necessary to have results prior to administration, except for results of a serum pregnancy test, if indicated. Lab tests must be drawn within the 3 days prior to infusion.
- <sup>11</sup> Reactogenicity assessments performed for 3 days postinfusion (see Section 7.10).
- <sup>12</sup> And microscopy if needed.
- 13 If HIV test results are not available at the visit indicated, provide test results at the next available opportunity.

## Appendix K Schedule 2—Procedures at CRS for HIV-1-infected participants

| Visit Number: | #.X <sup>1</sup> | | 31 | 32 | 33 | 34 | 35 |
|---|---|---|---|---|---|---|---|
| | | Days after diagnosis <sup>2</sup> | D28 | D42 | D56 | D84 | D168 |
| | | Weeks<br>after<br>diagnosis | 4 | 6 | 8 | 12 | 24 |
| Study procedures <sup>3</sup> | | | | | | | |
| Counseling on HIV-1 testing/diagnosis | Х | | Х | _ | _ | _ | _ |
| Abbreviated physical exam <sup>4</sup> | Х | | Х | Х | Х | Х | _ |
| Complete physical exam <sup>4</sup> | _ | | _ | _ | _ | _ | х |
| ART assessment | Х | | х | Χ | Х | Х | Х |
| Concomitant medications | _ | | Х | Х | х | Х | х |
| Intercurrent illness/adverse experience | _ | | Х | Х | Х | Х | Х |
| Transmission risk reduction counseling | Х | | Х | Х | Х | Х | Х |
| Behavioral risk assessment questionnaire | _ | | - | _ | _ | _ | х |
| Social impact assessment | Х | | Х | Х | х | Х | х |
| Local lab assessment | | | | | | | |
| Pregnancy test <sup>5</sup> | Х | | _ | _ | _ | Х | _ |
| CD4+ T cell count | Х | | Х | Χ | Х | Х | х |
| Hemoglobin | | | | | Х | х | |

<sup>&</sup>lt;sup>1</sup> Visit #.X indicates a Redraw visit where # is a Schedule 1 visit number. Confirmatory draw for HIV diagnostics will be collected at the Redraw visit. The Redraw visit should occur as soon as possible after the clinic receives a Redraw Request from the HIV diagnostics laboratory. Multiple Redraw visits may be necessary; only the blood specimen indicated in Appendix G will be collected at the subsequent Redraw visits.

<sup>&</sup>lt;sup>2</sup> Date of diagnosis = date of the initial specimen draw that led to the first Redraw Request

<sup>&</sup>lt;sup>3</sup> For specimen collection requirements, see Appendix G.

<sup>&</sup>lt;sup>4</sup> Includes assessment of HIV/AIDS-related conditions.

<sup>&</sup>lt;sup>5</sup> For participants capable of becoming pregnant, pregnancy test may be performed on urine or blood specimens.

# Appendix L Schedule 3—Procedures at CRS for participants discovered to have been HIV-1-infected at enrollment or who become HIV-2-infected

| Visit Number | #.X <sup>1</sup> | | 47 | 48 |
|---|---|---|---|---|
| | | Days after diagnosis <sup>2</sup> | D28 | D168 |
| | | Weeks after diagnosis | 4 | 24 |
| Study procedures <sup>3</sup> | | | | |
| Counseling on HIV-1 testing/diagnosis | Х | | Χ | _ |
| Abbreviated physical exam <sup>4</sup> | Х | | Χ | _ |
| Complete physical exam <sup>4</sup> | _ | | _ | х |
| ART assessment | Х | | Х | Х |
| Concomitant medications | _ | | Х | Х |
| Intercurrent illness/adverse experience | _ | | Χ | Х |
| Transmission risk reduction counseling | Х | | Χ | Х |
| Behavioral risk assessment questionnaire | _ | | _ | Х |
| Social impact assessment | Х | | Χ | Х |
| Local lab assessment | | | | |
| Pregnancy test <sup>5</sup> | Х | | _ | _ |
| CD4+ T cell count | Х | | Χ | Х |

<sup>&</sup>lt;sup>1</sup> Visit #.X indicates a Redraw visit where # is a Schedule 1 visit number. Confirmatory draw for HIV diagnostics will be collected at the Redraw visit. The Redraw visit should occur as soon as possible after the clinic receives a Redraw Request from the HIV diagnostics laboratory. Multiple Redraw visits may be necessary; only the blood specimens indicated in Appendix H will be collected at the subsequent Redraw visits.

<sup>&</sup>lt;sup>2</sup> Date of diagnosis = date of the initial specimen draw that led to the first Redraw Request

<sup>&</sup>lt;sup>3</sup> For specimen collection requirements, see Appendix H.

<sup>&</sup>lt;sup>4</sup> Includes assessment of HIV/AIDS-related conditions.

<sup>&</sup>lt;sup>5</sup> For participants capable of becoming pregnant, pregnancy test may be performed on urine or blood specimens.

# Appendix M Schedule 4—Procedures at CRS for participants who discontinue infusions for reasons other than HIV infection

| Visit Number: | 71 | 72 | 73 | 74 | 75 | 76 | 77 | 78 | Post |
|---|---|---|---|---|---|---|---|---|---|
| Days after enrollment: | 56 | 140 | 224 | 308 | 392 | 504 | 616 | 728 | |
| Weeks after enrollment: | 8 | 20 | 32 | 44 | 56 | 72 | 88 | 104 | |
| Study procedures <sup>1</sup> | | | | | | | | | |
| Abbreviated physical exam | Х | Х | Х | Х | Х | Х | Х | _ | _ |
| Complete physical exam | - | _ | _ | _ | _ | _ | _ | Х | _ |
| Risk reduction counseling | Х | Х | Х | Х | Х | Х | Х | Х | _ |
| Concomitant medications | Х | Х | Х | Х | Х | Х | Х | Х | _ |
| Intercurrent illness/adverse experience | Х | Х | Х | Х | Х | Х | Х | Х | _ |
| HIV infection assessment <sup>2</sup> | Х | Х | Х | Х | Х | Х | Х | Х | _ |
| Confirm HIV test results provided to participant <sup>3</sup> | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Behavioral risk assessment questionnaire | - | Х | _ | Х | _ | Х | _ | Х | _ |
| Social impact assessment | Х | Х | Х | Х | Х | Х | Х | Х | _ |
| Local lab assessment | | | | | | | | | |
| Urine dipstick <sup>4</sup> | Х | _ | _ | _ | _ | _ | Х | _ | _ |
| Pregnancy test <sup>5</sup> | Х | _ | Х | _ | Х | _ | Х | _ | _ |
| Poststudy | | | | | | | | | |
| Unblind participant | _ | _ | _ | _ | _ | _ | _ | _ | Х |

<sup>&</sup>lt;sup>1</sup> For specimen collection requirements, see Appendix I..

<sup>&</sup>lt;sup>2</sup> Includes pre-test counseling and HIV testing. A subsequent follow-up contact is conducted to provide post-test counseling and to report results to participant.

<sup>&</sup>lt;sup>3</sup> If HIV test results are not available at the visit indicated, provide test results at next available opportunity.

<sup>&</sup>lt;sup>4</sup> And microscopy if needed.

<sup>&</sup>lt;sup>5</sup> For participants capable of becoming pregnant, pregnancy test may be performed on urine or blood specimens.

### **Appendix N** Protocol Signature Page

A phase 2b study to evaluate the safety and efficacy of VRC01 broadly neutralizing monoclonal antibody in reducing acquisition of HIV-1 infection in women in sub-Saharan Africa

I will conduct the study in accordance with the provisions of this protocol and all applicable protocol-related documents. I agree to conduct this study in compliance with United States (US) Health and Human Service regulations (45 CFR 46); applicable U.S. Food and Drug Administration regulations; standards of the International Conference on Harmonization Guideline for Good Clinical Practice (E6); Institutional Review Board/Ethics Committee determinations; all applicable in-country, state, and local laws and regulations; and other applicable requirements (e.g., US National Institutes of Health, Division of AIDS) and institutional policies

Investigator of Record Name (print)

Investigator of Record Signature

Date

DAIDS Protocol Number: HVTN 703/HPTN 081

DAIDS Protocol Version: Version 4.0

Protocol Date: December 14, 2017